### Janssen Research & Development

### **Statistical Analysis Plan**

A Pilot Phase 2a, Randomized, Double-blind, Placebo-controlled Study to Explore the Antiviral Activity, Clinical Outcomes, Safety, Tolerability, and Pharmacokinetics of JNJ-53718678 at Two Dose Levels in Non-Hospitalized Adult Subjects Infected With Respiratory Syncytial Virus

## Protocol 53718678RSV2004; Phase 2a AMENDMENT 1

JNJ-53718678

**Status:** Approved

Date: 27 September 2019

Prepared by: Janssen Research & Development, LLC; Janssen Research & Development, a

division of Janssen Pharmaceutica NV

**Document No.:** EDMS-ERI-171344037; 2.0

**Compliance:** The study described in this report was performed according to the principles of Good Clinical Practice (GCP).

#### **Confidentiality Statement**

The information in this document contains trade secrets and commercial information that are privileged or confidential and may not be disclosed unless such disclosure is required by applicable law or regulations. In any event, persons to whom the information is disclosed must be informed that the information is privileged or confidential and may not be further disclosed by them. These restrictions on disclosure will apply equally to all future information supplied to you that is indicated as privileged or confidential.

# **TABLE OF CONTENTS**

| TABLE | OF CONTENTS | <mark>2</mark> |
|---|---|---|
| LIST C | OF IN-TEXT TABLES AND FIGURES | 4 |
| AMEN | DMENT HISTORY | 5 |
| ABBRI | EVIATIONS | 13 |
| 1. II | NTRODUCTION | 14 |
| 1.1. | Trial Objectives | 14 |
| 1.2. | Trial Design | 15 |
| 1.3. | Statistical Hypotheses for Trial Objectives | 16 |
| 1.4. | Sample Size Justification | 16 |
| 1.5. | Randomization and Blinding | 17 |
| | GENERAL ANALYSIS DEFINITIONS | 17 |
| 2.1. | Phase Definitions, Visit Windows and Baseline | 17 |
| 2.1.1. | Phase Definitions | 18 |
| 2.1.2. | Analysis Windows for Analysis Visits and Timepoints | 19 |
| 2.1.3. | Study Day and Relative Day | |
| 2.1.4. | Baseline | 23 |
| 2.2. | Pooling Algorithm for Analysis Centers | <mark>23</mark> |
| 2.3. | Analysis Sets | 24 |
| 2.3.1. | All Randomized Analysis Sets | 24 |
| 2.3.1.1 | . All Randomized Analysis (RAND) Set | 24 |
| 2.3.2. | Efficacy Analysis Set(s) | |
| 2.3.2.1 | | |
| 2.3.2.2 | | |
| 2.3.2.3 | | |
| 2.3.3. | Safety Analysis Set | |
| 2.3.3.1 | | |
| 2.4. | Definition of Subgroups | |
| 2.5. | Imputation Rules for Missing AE Date/Time of Onset/Resolution | 26 |
| | NTERIM ANALYSIS AND DATA REVIEW COMMITTEE | |
| 3.1. | Interim Analysis | |
| 3.2. | Data Review Committee | 27 |
| | SUBJECT INFORMATION | |
| 4.1. | Demographics and Baseline Characteristics | |
| 4.2. | Disposition Information | |
| 4.3. | Treatment Compliance | |
| 4.4. | Extent of Exposure | |
| 4.5. | Protocol Deviations | |
| 4.6. | Medical History | |
| 4.7. | Prior and Concomitant Medications | |
| 4.8. | Co-Infections | 31 |
| | FFICACY | |
| 5.1. | Analysis Specifications | |
| 5.1.1. | Level of Significance | |
| 5.1.2. | Data Handling Rules | |
| 5.2. | Primary Efficacy Endpoints – Viral Load | |
| 5.2.1. | Definition | |
| 5.2.2. | Analysis Methods | |
| 5.3. | Secondary Endpoints - Clinical Course | 39 |

| 5.3.1. Definition | |
|---|---|
| 5.3.1.1. ePROs | |
| 5.3.1.2. Clinical Course Endpoints related to Respiratory, Heart Rate and Body Temperature | 49 |
| 5.3.1.2.1. Respiratory Rate, Heart Rate, Oxygen Saturation and Body Temperature | 49 |
| 5.3.1.2.2. Other Clinical Course Parameters | |
| 5.3.2. Analysis Methods | |
| 5.3.2.1. Endpoint-specific analysis methods | 52 |
| 5.4. Sensitivity Analyses | 54 |
| 5.5. Other Efficacy Variable(s) | |
| 5.5.1. Definition | |
| 5.5.2. Analysis Methods | 55 |
| 5.6. Exploratory Analyses | 55 |
| 6. SAFETY | <b>56</b> |
| 6.1. Adverse Events | |
| 6.1.1. Definitions | 56 |
| 6.1.2. Analysis Methods | 56 |
| 6.2. Clinical Laboratory Tests | |
| 6.2.1. Definitions | |
| 6.2.2. Analysis Methods | |
| 6.3. Vital Signs and Physical Examination Findings | |
| 6.3.1. Definitions | |
| 6.3.2. Analysis Methods | |
| 6.4. Electrocardiogram | |
| 6.4.1. Definitions | |
| 6.4.2. Analysis Methods | |
| 7. HEALTH ECONOMICS | 62 |
| 7.1 Definitions | |
| 7.2. Analysis Methods | 62 |
| 8. VIROLOGY | <mark>63</mark> |
| 8.1. Definitions | 63 |
| 8.2. Analysis Methods | 64 |
| 8.2.1. Viral Strain Typing | 64 |
| 8.2.2. Viral Sequencing | |
| REFERENCES | 88 |
| ATTACHMENTS | <mark>67</mark> |
| Attachment [1]: Division of Microbiology and Infectious Diseases (DMID) Adult Toxicity Table | 67 |
| November 2007 Attachment [2]: Inclusion/exclusion criteria | |
| The state of the s | /5 |
| Attachment [3]: 79 | 70 |
| Respiratory infection-patient reported outcomes (ri-pro © ) symptom questionnaire | |
| Adult RSV additional questions | |
| Respiratory Infection Intensity and Impact Questionnaire (RiiQ™) | |
| Attachment [4]: EQ-5D-5L | |
| EQ-5D-5L Dimensions | 84 |
| EQ-5D-5L VAS 85 | |
| Valuation Index 86 | |

# **LIST OF IN-TEXT TABLES AND FIGURES**

# **TABLES**

| Table 1: | Definition of Analysis Phases | 18 |
|-----------|---------------------------------------------------|----|
| Table 2: | Visit Windows | |
| Table 3: | Visit Windows for ePRO | |
| Table 4: | Worst per Day | |
| Table 5: | ePRO Time Slot in a Day | |
| Table 6: | Subgroups | 25 |
| Table 7: | Demographic Variables | |
| Table 8: | Time Šlot in a Day | |
| Table 9: | Correction Factor for Time Slot in a Day | 29 |
| Table 10: | Baseline Characteristics | 29 |
| Table 11: | AUC viral load | 34 |
| Table 12: | Clinically Important Abnormalities in Vital Signs | 60 |
| Table 13: | ECG Abnormalities | 61 |
| FIGURES | S | |
| Figure 1: | Schematic Overview of the Study | 18 |

## **AMENDMENT HISTORY**

| Version | <b>Effective Date</b> | Description of Changes |
|---|---|---|
| 1.0 | 18DEC2018 | This is the original SAP. |
| 2.0 | 27AUG2019 | All changes and clarifications of planned analyses in the SAP Version 2.0 compared with the SAP Version 1.0 are listed below. |

| Topic or Section | Description of Changes and Clarifications of Planned Analyses |
|---|---|
| 1. Introduction | This SAP (Version 2.0) is based on the Clinical Protocol finalized on 26 September 2018 and the Clinical Protocol Amendment INT-1 finalized on 12 April 2019. Any changes of the text in the original SAP (Version 1.0) are explicitly stated in this updated SAP. |
| The statement on the RSV viral load mean change from to Day 8 associated with the sample size calculation without affecting the sample size itself. Using assumptions on the mean change and its SD, the precision was updated to be the half width of confidence interval for the between-group different viral load change from baseline, instead of the single arm 90% CI. | |
| | The following text: With an assumed SD of 1.85 log <sub>10</sub> copies/mL, 20 subjects per treatment group will lead to a precision (90% confidence interval [CI] half width) of 0.715 and 24 subjects per treatment group to a precision of 0.647 log <sub>10</sub> copies/mL for the estimate of the mean change from baseline per treatment group. was replaced by: |
| | With an assumed SD of 1.85 log <sub>10</sub> copies/mL, 20 subjects per treatment group will lead to a precision (90% confidence interval [CI] half width) of 0.986 and 24 subjects per treatment group to a precision of 0.896 log <sub>10</sub> copies/mL for the estimate of the difference between treatment groups in the mean change from baseline to Day 8. |

| 2.1.2 Analysis Windows for Analysis Visits and | 1. In Table 3, the following typos were corrected for Days 10.5 and 11: |
|---|---|
| Timepoints | Day 10.5: 231h 59 min was replaced by 233h 59 min |
| | Day 11: 232h was replaced by 234h |
| | 2. The following text was added to clarify Table 4: |
| | The secondary selection approach will only be considered in the analysis if no record is assigned to Day 3, Day 5, Day 8 and Day 14 according to the rules in the primary selection column. If 'worst per day' as per primary selection is available, same value will be assigned for the secondary selection of 'worst per day'. Otherwise, 'worst per day' as per secondary selection will be derived considering all possible values within the relative day window. The worst possible results will be selected regardless of being the closest one to target day. |
| 2.3.2 Efficacy Analysis Set(s) | 1. The following text was moved to section 5. Efficacy and further clarified: |
| | Efficacy will be analyzed on the ITT infected (ITT-i) set. The primary endpoint will also be analyzed on the Per Protocol (PP) set. |
| | 2. The following sub-section was added to ensure a minimal level of viral load at the start of treatment, allowing the antiviral effect of JNJ8678 to be evaluated: |
| | 2.3.2.2 Modified Intent-To-Treat infected (mITT-i) Set |
| | All subjects in the ITT-i analysis set with RSV viral load >= 1 log <sub>10</sub> copies/mL above the Lower Limit of Quantification (LLOQ) at baseline. |
| 3.1 Interim Analysis | As a clarification for completeness, the following text |
| | An interim analysis, encompassing efficacy, safety, and pharmacokinetics is planned after at least 36 subjects have been dosed and have completed the assessments of Day 8. |
| | was replaced by: |
| | An interim analysis, encompassing efficacy, safety, and pharmacokinetics is planned after at least 36 subjects have been dosed and have completed the assessments of Day 8, or |

| | discontinued earlier. |
|---|---|
| 4.1 Demographics and Baseline Characteristics | <ul> <li>The following baseline characteristics were added to Table 10:</li> <li>Baseline RSV Viral Load (log<sub>10</sub> copies/ml) by RSV Subtype</li> <li>Baseline RSV Viral Load (log<sub>10</sub> copies/ml) by symptom onset day</li> </ul> |
| 5. Efficacy | The following text was added: |
| | The primary endpoint will also be analyzed on mITT-i set and PP set. |
| 5.1 Analysis Specifications | 1. The following text was added: |
| | In addition, descriptive summaries will be presented by the randomization stratification factor, time of symptom onset ( $\leq$ 3 days vs >3 days before randomization). |
| | 2. The following clarification was added: |
| | For all the stratified statistical analyses, the derived randomization stratification factor will be used instead of the randomization stratification factor as collected in the IWRS. |
| 5.2.1 Definitions | 1. As the protocol was updated (Protocol-Amendment 1 dated on 12 April 2019) to include Day 5 as an additional timepoint for the assessment of the area under the RSV viral load-time curve (AUC), the following text was removed: |
| | Change from planned analyses; For viral load the AUC for Day 5 has been included. |
| | 2. The following text was added as a clarification on the calculation of the viral load of AUC with missing data: |
| | Carrying forward should only be performed if the time between<br>the available observation and the value at xxh is at most 24<br>hours. |
| | In case the last observation is before xxh, and the value at xxh cannot be determined, the AUCs through xxh and through any later timepoint will not be derived. |
| 5.2.2 Analysis Methods | 1. A clarification about the subgroup analyses for AUC viral load was added: |
| | The homogeneity of treatment effect on the occurrence of AUC viral load from baseline to Days 3, 5, and 8 across subgroups |

will be examined using the same MMRM model approach for the primary analysis, but also includes the subgroup-bytreatment and subgroup-by-visit interaction terms in the model. A forest plot will present the Least Square means and 95% CI for all subgroups of interest.

2.A clarification about the stratified Cox proportional hazard model as well as the calculation of the 90% confidence intervals based on the Kaplan-Meier method was added:

Time-to event variable will be analyzed and plotted using Kaplan-Meier estimates analysis. The estimate of the hazard ratio (HR) and the 90% confidence intervals for the treatment effect will be provided based on a stratified Cox proportional hazard model (derived randomization stratification factor: ≤3 days, >3 days) and including treatment group as a covariate.

A summary table including number of subjects included in the analysis, number of subjects censored, 25<sup>th</sup> and 75<sup>th</sup> percentiles and median time-to event, with 90% confidence intervals based on the Kaplan-Meier method, will be presented by treatment group.

3.A clarification about the subgroup analyses for the time to virus undetectable was added:

The potential impact of selected variables that identify the subgroups of interest on the time to virus undetectable will be assessed by the stratified Cox proportional hazard model. The model will be stratified by the randomization stratification factors and include treatment group and subgroup variable as covariates, and the subgroup-by-treatment interaction term. A forest plot will present the HRs and 90% CI for all subgroups of interest.

4. A clarification about the calculation of the difference in proportion of subjects with undetectable RSV viral load was added. The subjects with detectable or quantifiable RSV viral load are grouped into one category, so the subjects can be classified as either with RSV viral load 'undetectable' or 'detectable or quantifiable':

The difference in proportions for undetectable versus detectable/quantifiable between each active group and placebo, will be tabulated descriptively (n and % per treatment group), for

| each post baseline timepoint. | |
|---|---|
| 5.3. Secondary Endpoints - Clinical Course | According to Protocol-Amendment 1, the RI-PRO (for newly recruited subjects) was replaced by RiiQ (RI-PRO still being collected at certain timepoints). Therefore, endpoints derived from RiiQ were added: |
| | • Duration and severity of signs and symptoms of RSV infection assessed through either the Respiratory Infection Patient Reported Outcome (RI-PRO) or the Respiratory Infection Intensity and Impact Questionnaire [RiiQ] questionnaire, and Additional Questions about Health and Functioning. |
| | Time to resolution of selected RSV symptoms as reported by the subject through either the RI-PRO or RiiQ. |
| 5.3.1.1 ePROs | According to Protocol-Amendment 1, the RI-PRO (for newly recruited subjects) was replaced by RiiQ (RI-PRO still being collected at certain timepoints). Therefore, information regarding the RiiQ, calculation and analyses of the RiiQ (symptom or impact) domain scores, RiiQ key symptom score, and related time to (complete) resolution were added to this section. |
| | in addition, details about the RI-PRO key RSV symptom score and related time to (complete) resolution analyses were added. |
| | Time to (complete) resolution analyses based on the common key symptoms from either RI-PRO or RiiQ were also added to this section. |
| 5.3.2.1 Endpoint-specific analysis methods | 1. According to Protocol-Amendment 1, the RI-PRO (for newly recruited subjects) was replaced by RiiQ (RI-PRO still being collected at certain timepoints). Therefore, the following text was added: |
| | Changes from baseline on each of the RI-PRO and RiiQ domains will be analyzed using a restricted maximum likelihood based repeated measures approach as per Section 5.2.2. An unstructured covariance structure will be selected. |
| | 2. The typo regarding the confidence level for the confidence interval based on Wilson score test was corrected: '95% confidence interval' was replaced by '90% confidence interval': |
| | The difference in proportions between each active group and |

placebo will be tabulated, and summaries will include 2-sided 90% confidence intervals based on the Wilson score test.

3. The following text was added under 'Time to resolution of symptoms, Time to return to usual health and Time to return to usual activity':

The estimate of the hazard ratio (HR) and the 90% confidence intervals for the treatment effect will be provided based on a stratified Cox proportional hazard model (derived randomization stratification factor:  $\leq 3$  days, > 3 days) and including treatment group as a covariate.

4. A clarification about the calculation of the 90% confidence intervals was added under 'Time to resolution of symptoms, Time to return to usual health and Time to return to usual activity':

A summary table including number of subjects included in the analysis, number of subjects censored, 25<sup>th</sup> and 75<sup>th</sup> percentiles and median time-to event, with 90% confidence intervals based on the Kaplan-Meier method, will be presented by treatment group.

5. A clarification on the subgroup analyses for the time to resolution of symptoms was added:

The potential impact of selected variables that identify the subgroups of interest on the time to resolution of symptoms will be assessed by the stratified Cox proportional hazard model. The model will be stratified by the randomization stratification factors and include treatment group and subgroup variable as covariates, and the subgroup by treatment interaction term. A forest plot will present the HRs and 90% CI for all subgroups of interest.

### 5.4. Sensitivity Analyses

The following sensitivity analyses were added:

Sensitivity analyses to assess the robustness of the primary efficacy analysis of viral load AUC will be performed by including the stratification factor, RSV symptom onset ( $\leq$ 3 days or > 3 days) as collected in the IWRS, in the mixed-effects model. Additionally, the primary efficacy analysis will be repeated on the mITT-I set.

For the time to resolution of selected RSV symptoms, sensitivity

| | <ul> <li>analyses will be performed considering 4 different imputation methods:</li> <li>Method 1: from first resolution (score 0 or 1) after last unresolved value onwards, impute missing data as resolution.</li> <li>Method 2: impute all missing values as unresolved (score &gt;1).</li> <li>Method 3: impute all missing values in-between resolved observations (score 0 or 1) as resolved.</li> <li>Method 4: impute all missing values as unresolved (score &gt;1), except when in-between resolved values where resolved is imputed.</li> </ul> |
|---|---|
| 5.6 Exploratory Analyses | According to Protocol-Amendment 1, the RI-PRO (for newly recruited subjects) was replaced by RiiQ (RI-PRO still being collected at certain timepoints). Therefore, information regarding the RiiQ analyses was added under the 'Clinical course endpoints'. |
| 7.2. Analysis Methods | A clarification about the method used in calculating the 90% confidence interval for a binomial proportion was added as follows: The proportion of subjects requiring any medical encounter will be shown in a frequency tabulation by treatment group with the corresponding 90% confidence interval (exact Clopper-Pearson method). |
| 8.1 Definitions | 1. Position 127 was added to the following text: Long list of 20 F-gene positions of interest for the class of RSV fusion inhibitors, based on in vitro selection experiments, clinical observations, and/or in vitro reduced susceptibility to RSV fusion inhibitors: positions 127, 138, 140, 141, 143, 144, 323, 338, 392, 394, 398, 399, 400, 401, 474, 486, 487, 488, 489, and 517. |
| | <ul> <li>2. The following clarification was added for the 'Last Evaluable On-Treatment Time Point', under 'Analysis Time Points':</li> <li>In case no On-Treatment assessment is available, the first assessment during Follow-Up is selected instead.</li> <li>3. 'During the follow-up phase' was added as a clarification to the definition of the 'Time Point of Sequence during the Follow-Up phase', under 'Analysis Time Points'.</li> </ul> |

### **ABBREVIATIONS**

ΑE adverse event

Accelerated Failure Time **AFT** ALT/SGPT alanine aminotransferase AST/SGOT aspartate aminotransferase ATC anatomic and therapeutic Class

**AUC** area under the curve body mass index BMI CI confidence interval

COPD chronic obstructive pulmonary disease **CPAP** Clinical Pharmacology Analysis Plan

CRF case report form Clinical Study Report **CSR** coefficient of variation CV

Division of Microbiology and Infectious Diseases **DMID** 

Data Review Committee DRC

DPS Data Presentation Specifications

**ECG** Electrocardiogram

eCRF electronic case report form FDA Food and Drug Administration

**HCP** Health Care Provider

**HRQOL** Health-Related Quality of Life

Interim Analysis IΑ **ICF** Informed Consent Form

International Conference on Harmonization ICH

Interquartile IQ

ITT-i Intent-to-Treat infected **IRBs Institutional Review Boards** interactive web response system **IWRS** Lower limit of quantification LLOO **LOCF** last observation carried forward

LOD Limit of detection Least Squares LS

MedDRA Medical Dictionary for Regulatory Activities

Modified Intent-to-Treat infected mITT-i

PD Pharmacodynamic PΙ principal investigator PΚ pharmacokinetic(s) per protocol

PP

Patient Reported Outcome PRO

quantitative reverse transcription polymerase chain reaction qRT-PCR RI-PRO Respiratory Infection-Patient Reported Outcomes questionnaire Respiratory Infection Intensity and Impact Questionnaire RiiQ

serious adverse event SAE SAF Safety Analysis Set Statistical Analysis Plan SAP standard deviation SD

**SDTM** Study Data Tabulation Model

SE Standard Error

peripheral capillary oxygen saturation  $SpO_2$ 

TD Target Detected TND Target Not Detected

treatment-emergent adverse event **TEAE** 

#### 1. INTRODUCTION

This Statistical Analysis Plan (SAP) contains definitions of analysis sets, derived variables and statistical methods for the efficacy and safety analyses of the study JNJ-57318678RSV2004. The SAP is to be interpreted in conjunction with the protocol.

This SAP (Version 2.0) is based on the Clinical Protocol finalized on 26 September 2018 and the Clinical Protocol Amendment INT-1 finalized on 12 April 2019. Any changes from the text in the original SAP (Version 1.0) are explicitly stated in this updated SAP.

A detailed analysis plan for the pharmacokinetic and pharmacokinetic/pharmacodynamics data will be described in a Clinical Pharmacology Analysis Plan (CPAP).

JNJ-53718678 is an investigational RSV specific fusion inhibitor belonging to the indole chemical class and is under development for the treatment of RSV infection. The study drug shows in vitro activity against a panel of viruses belonging to both the RSV subfamilies A or B. In addition, antiviral activity of JNJ-53718678 was demonstrated during clinical studies in healthy adults inoculated with RSV (study 53718678RSV2001) and in pediatric subjects hospitalized due to RSV-infection (study 53718678RSV1005).

## 1.1. Trial Objectives

### Primary Objective

The primary objective of the study is to explore the antiviral effect of JNJ-53718678 at 2 dose levels (80 mg and 500 mg) once daily for 7 days in adults with RSV infection, as measured by RSV viral load in nasal secretions by quantitative reverse transcription polymerase chain reaction (qRT-PCR) assay.

### Secondary Objectives

The secondary objectives are to explore in adults with RSV infection, after repeated oral dosing with JNJ-53718678:

- The safety and tolerability of JNJ-53718678
- The impact of JNJ-53718678 on the clinical course of RSV infection
- The pharmacokinetics of JNJ-53718678.

### **Exploratory Objectives**

The exploratory objectives are to explore in adults with RSV infection after repeated oral dosing with JNJ-53718678:

- The relationship between antiviral activity and clinical course
- The relationship between pharmacokinetics and pharmacodynamics (selected antiviral activity
- parameters, clinical outcomes, and safety parameters)

- Potential differences in antiviral activity and clinical course between:
  - o otherwise healthy and comorbid subjects;
  - o subjects with symptom onset  $\leq 3$  days before randomization and subjects with symptom onset  $\geq 3$  days before randomization.
- The occurrence of complications associated with RSV per investigator assessment after initiation of treatment
- Medical resource utilization, including hospitalization, for clinical management of subjects during treatment and posttreatment follow-up
- The impact of the baseline RSV viral subtype and genotype on the antiviral activity and clinical course
- The emergence of mutations in the viral genome potentially associated with resistance to JNJ-53718678
- The RSV infectious virus titers as assessed by quantitative culture of RSV (plaque assay) on selected nasal swab samples (optional objective, pending feasibility of performing such an assay)
- Impact of RSV and its treatment on health-related quality of life (HRQOL).

## 1.2. Trial Design

This is a Phase 2a, randomized, double-blind, placebo-controlled study to explore the antiviral activity, clinical outcomes, safety, tolerability, and pharmacokinetics of JNJ-53718678 at 2 dose levels (80 mg and 500 mg) once daily for 7 days in adult subjects with respiratory illness due to RSV infection. Subjects may be otherwise healthy or comorbid and should not be in need of hospitalization.

A population of 75 subjects is targeted. However, given the recruitment challenges associated with the seasonality of RSV, a minimum of 63 subjects may be considered sufficient to complete the study.

The study includes a Screening Period (Day -1 to Day 1), a Treatment Period (Day 1 to Day 8), and a Follow-up Period (Day 9 to Day 28[±3]). The total study duration for each subject is 29 days (screening included).

After screening, eligible subjects are randomized on Day 1 (1:1:1) to receive 1 of 3 treatments:

- Treatment A: 500 mg JNJ-53718678 once daily for 7 days (n = 25 [target]);
- Treatment B: 80 mg JNJ-53718678 once daily for 7 days (n = 25 [target]);
- Treatment C: placebo once daily for 7 days (n = 25 [target]).

Randomization is stratified by time of symptom onset ( $\leq 3$  days vs > 3 days before randomization). Subjects with symptom onset > 3 days before randomization may account for maximum of 50% of all enrolled subjects.

An interim analysis is planned after at least 36 subjects have been dosed and have completed the assessments of Day 8.

A Data Review Committee (DRC) is in place for this study. The DRC monitors safety data during study conduct on a regular basis and/or ad hoc in case of emergent safety signals identified through medical monitoring.

## 1.3. Statistical Hypotheses for Trial Objectives

The primary objective of the study is to explore the antiviral effect of JNJ-53718678 at 2 dose levels (80 mg and 500 mg) once daily for 7 days in adults with RSV infection, as measured by RSV viral load in nasal secretions by quantitative reverse transcription polymerase chain reaction (qRT-PCR) assay.

No statistical hypotheses are to be tested.

## 1.4. Sample Size Justification

The interim results (estimates of mean AUC and change from baseline of RSV viral load  $\pm$ SD) of study 53718678RSV1005 were the basis of the sample size calculation. In that study, median (range) time to onset of symptoms was 5 (2-12) days and baseline viral load was 5.3 (2.1-8.3) log10 copies/mL.

For the AUC viral load from Day 1 to Day 7, a (placebo) point estimate of 490 and an SD of 135 log10 copies x hr/mL was observed for the AUC viral load from Day 1 to Day 7. The sample size was determined in order to obtain estimates of the mean AUC viral load with a precision of approximately 50 log10 copies x hr/mL of the true value with 90% confidence; with 20 subjects per treatment group the half-width of the 90% confidence would be approximately 52 and with 24 subjects per treatment group the precision would be approximately 47 log10 copies x hr/mL.

For the change from baseline (on Day 2 or Day 3), (placebo) point estimates of -0.11 and -0.33 and SDs of 1.85 and 1.56 log10 copies/mL, respectively, were observed. The observed difference (active versus placebo) was -1 to -2 log10 copies/mL. With an assumed SD of 1.85 log10 copies/mL, 20 subjects per treatment group will lead to a precision (90% confidence interval [CI] half width) of 0.986 and 24 subjects per treatment group to a precision of 0.896 log10 copies/mL for the estimate of the difference between treatment groups in the mean change from baseline.

As further guidance for the design, the power to detect a dose-response was calculated. To evaluate a potential dose-response, 3 contrasts will be tested: a contrast with no difference between the 2 active doses tested against placebo; a contrast with no difference between low dose and placebo tested against high dose; and a contrast with a linear dose-response relationship with respect to the active doses. No correction for multiplicity is considered in view of the exploratory nature of the study. Based on 10,000 simulations, and assuming a reduction in AUC viral load of 20% of high dose versus placebo, the power to detect a positive dose-response relationship will be between 79% and 86% (depending on the effect of the low dose) with a total sample size of 60, and between 83% and 89% with a total sample size of 72.

16

To account for potential false-positive RSV screening testing (ie, diagnosed with RSV infection using a rapid PCR-based or rapid antigen-detection test, but negative at the central lab using a qRT-PCR assay, and therefore not included in the primary analysis population of ITT-i) and withdrawals from treatment for abnormal screening laboratory results, an overage of approximately 5% will be enrolled, ie, 75 subjects are targeted.

In view of the seasonality of the disease, recruitment will be halted if at the end of a hemispheric RSV season 63 or more subjects have been enrolled and dosed. If at the end of a hemispheric RSV season the minimum of 63 dosed subjects is not reached, recruitment will continue in a next RSV season until this minimum has been reached, up to a maximum of 75 subjects to be enrolled overall.

## 1.5. Randomization and Blinding

Central randomization is implemented in this study. The codes will be maintained within the IWRS, which has the functionality to allow the investigator to break the blind for an individual subject. Subjects are randomly assigned to 1 of the 3 treatments to receive either a high (500 mg/day) or a low (80mg/day) dose of JNJ53718678 or placebo in 1:1:1 ratio. The randomization is balanced by using randomly permuted blocks and stratified by time since symptom onsent at randomization ( $\leq$ 3 days vs  $\geq$ 3 days). Subjects with symptom onset  $\geq$ 3 days before randomization may account for maximum of 50% of all enrolled subjects.

In order to maintain study blind, all subjects receive once daily the same total volume of study drug solution divided over 2 separate but sequential intakes at the same time of day.

#### 2. GENERAL ANALYSIS DEFINITIONS

All analysis dataset preparations and statistical analyses will be performed using SAS® version 9.2 (or higher).

### 2.1. Phase Definitions, Visit Windows and Baseline

A diagram of the study design is provided in Figure 1.

Figure 1: Schematic Overview of the Study



#### 2.1.1. Phase Definitions

Phases will be defined as in Table 1.

Table 1: Definition of Analysis Phases

| Analysis | Start Date/Time | End Date/Time |
|---|---|---|
| Phase | | |
| [Phase No.] | | |
| Screening | 00:00 of the date of signing the | 1 minute before the first study drug |
| [1] | informed consent form | administration in the trial |
| Treatment | Date and time of first study drug | 23:59 of the last day of treatment +3 |
| [2] | administration in the trial (Study Day | days (or date of last contact if still on |
| | 1) | treatment) |
| | • | or |
| | | 23:59 of the cut-off date for the IA, |
| | | whichever occurs first |
| Follow-up | 1 minute after End of Treatment Phase | 23:59 of the day of trial termination (date |
| [3] | | of last contact) or |
| | | 23:59 of the cut-off date for the IA, |
| | | whichever comes first |

Assessments will be assigned to phases based on their datetime, but seconds will be ignored overall. If the day part of the start date of the assessment is present but the time part is missing, the assessment will be treated as if it started at 00:00 on the day of the event (unless for Adverse Events see details in Section 2.5). If the day part of the end date of the assessment is present but the time part is missing, the assessment will be treated as if it happened at 23:59 on the day of the assessment. No formal imputation will be done, these rules will only be applied to allocate assessments to phases.

### 2.1.2. Analysis Windows for Analysis Visits and Timepoints

As subjects do not always adhere to the protocol visit schedule, the following rules are applied to assign actual visits to analysis visits. All assignments will be made in chronological order. Once a visit date is assigned to a visit window, it will no longer be used for a later time point except for the endpoint. Listed below (please see Table 2, Table 3 and Table 4) are the visit windows and the target days for each visit defined in the protocol.

For the analyses of measurements scheduled once daily the following rules will be applied to have only one evaluation per subject per analysis visit:

- If two assessments fall within the same visit window, the measurement closest to the target day will be used.
- If the assessments are equidistant, the last measurement within the interval will be used.
- If there are two measurements on the same date and time, then the measurement with the highest sequence number will be used.

Once baseline is assigned, any assessment performed prior to the defined baseline, will be assigned to Screening. Screening visits will not be used in summary tables but only in listings.

Any assessment performed within Day 1 but after first drug intake, will be assigned to Day 1 post-dose.

Exceptions to the general rule:

#### Viral Load

For the analyses of viral load (scheduled once daily), if multiple nasal swabs were taken on a single day, the above rules will only be applied after having determined per day the maximum viral load. The maximum viral load on a day will be used for windowing. Please notice that baseline viral load follows the rules described in Section 2.1.4.

### • *Electrocardiogram*

In case there is more than one assessment per analysis visit window, the following rule will be used to have only one evaluation per analysis timepoint:

- The average of the last available complete ECG triplicate should be considered in first instance.
- In absence of complete triplicate ECGs, the average of the last available ECG duplicate should be considered.
- In absence of complete or partial triplicates, the last available single ECG can be used.

If an assessment is performed but not planned per protocol, it may be assigned to a visit window for consistency, based on the relative day. However, it will not be shown in the summary tables and figures as only scheduled visits per protocol are used.

Screening visits will not be used in summary tables but only in listings. All information will be listed.

Table 2: Visit Windows

| Table 2. Visi | it Williams | | | | | | |
|---|---|---|---|---|---|---|---|
| Analysis Visit<br>[scheduled<br>Analysis Visit | TIME INTERVAL (Day)*<br>[TARGET TIMEPOINT (Day)] | | | | | | |
| No.] | EQ-5D-5L <sup>§</sup> | Clinical | Body Temp. | Viral Load | Vital Signs | ECG | Clinical |
| | | Parameters | | | Ü | / | Laboratory |
| | | (excluding | | | | PK | |
| | | Body | | | | | |
| | | Temp.) | | | | | |
| Screening<br>[-1] | <1<br>[-1 to 1] | <1<br>[-1 to 1] | <1<br>[-1 to 1] | <1<br>[-1 to 1] | <1<br>[-1 to 1] | <1<br>[-1 to 1] | <1<br>[-1 to 1] |
| Baseline+ | <=1 | <=1 | <=1 | <=1 | <=1 | <=1 | <=1 |
| [0] | [1] | [1] | [1] | [1] | [1] | [1] | [1] |
| Day 1 | 1 | | 1 | 1 | | | |
| [1] | [1] | | [1] | [1] | | | |
| Day 2 | 2<br>[2] | | 2<br>[2] | 2<br>[2] | | | |
| Day 3** | 2 to 5 | 2 to 5 | 3 | 3 | 2 to 5 | 2 to 5 | 2 to 5 |
| [3] | [3] | [3] | [3] | [3] | [3] | [3] | [3] |
| <b>Day 4</b> [4] | 4<br>[4] | | 4<br>[4] | 4<br>[4] | | | |
| Day 5 | 5 | | 5 | 5 | | | |
| [5] | [5] | | [5] | [5] | | | |
| Day 6 | 6 | | 6 | 6 | | | |
| [6]<br>Day 7 | [6]<br>7 | | [6]<br>7 | [6]<br>7 | | | |
| [7] | [7] | | [7] | [7] | | | |
| Day 8** | 8 | 6 to 10 | 8 | 8 | 6 to 10 | 6 to 10 | 6 to 10 |
| [8] | [8] | [8] | [8] | [8] | [8] | [8] | [8] |
| Day 9*** | 9 | | 9~ | 9 | | | |
| [9]<br>Day 10*** | [9]<br>10 | | [9]<br>10 | [9]<br>10 | | | |
| [10] | [10] | | [10] | [10] | | | |
| Day 11*** | 11 | | 11 | 11 | | | |
| [11] | [11] | | [11] | [11] | | | |
| Day 12*** | 12 | | 12 | 12 | | | |
| [12]<br>Day 13*** | [12]<br>13 | | [12]<br>13 | [12]<br>13 | | | |
| [13] | [13] | | [13] | [13] | | | |
| Day 14** | 14 | 11-17 | 13 to 17 | 13 to 17 | 11 to 17 | 11 to 17 | 11 to 17 |
| [14] | [14] | [14] | [14] | [14] | [14] | [14] | [14] |
| Day 15<br>[15] | 15<br>[15] | | | | | | |
| Day 16 | 16 | | | | | | |
| [16] | [16] | | | | | | |
| <b>Day 17</b> [17] | 17<br>[17] | | | | | | |
| Day 18 | 18 | | | | | | |
| [18] | [18]<br>19 | | | | | | |
| <b>Day 19</b><br>[19] | [19] | | | | | | |
| Day 20<br>[20] | 20<br>[20] | | | | | | |
| [3] | [] | | | | | | |

Table 2: Visit Windows

| Day 21** | 21-24 | 18-24 | 18-24 | 18-24 | 18-24 | 18-24 | 18-24 |
|---|---|---|---|---|---|---|---|
| [21] | [21] | [21] | [21] | [21] | [21] | [21] | [21] |
| Day 28 | 25 to +∞ | 25 to +∞ | 25 to +∞ | 25 to +∞ | 25 to +∞ | 25 to +∞ | 25 to +∞ ## |
| [28] | [28] | [28] | [28] | [28] | [28] | [28] | [28] |

<sup>+</sup> Baseline is defined as the last measurement before first study drug intake. Please also see section 2.1.4

Respiratory Infection Patient Reported Outcomes (RI-PRO), Respiratory Infection Intensity and Impact Questionnaire (RiiQ), and Additional Questions about Health and Functioning are collected twice daily (BID) from Day 1 through Day 13. Windows for these assessments are defined relative to the first study drug intake (0h): 12h (+/-6h), 24h (+/-6h), 36h (+/-6h), etc.

Table 3: Visit Windows for ePRO

| Analysis | time* | Target |
|-----------------|------------------------------|--------|
| time | Interval | Time |
| 12h (Day 1.5*) | >0h <sup>\$</sup> ; 17h59min | 12h |
| 24h (Day 2.0) | 18h; 29h 59 min | 24h |
| 36h (Day 2.5) | 30h; 41h 59min | 36h |
| 48h (Day 3.0) | 42h; 53h 59min | 48h |
| 60h (Day 3.5) | 54h; 65h 59min | 60h |
| 72h (Day 4.0) | 66h; 77h 59min | 72h |
| 84h (Day 4.5) | 78h; 89h 59min | 84h |
| 96h (Day 5.0) | 90h; 101h 59min | 96h |
| 108h (Day 5.5) | 102h; 113h 59min | 108h |
| 120h (Day 6.0) | 114h; 125h 59min | 120h |
| 132h (Day 6.5) | 126h; 137h 59min | 132h |
| 144h (Day 7.0) | 138h; 149h 59min | 144h |
| 156h (Day 7.5) | 150h – 161h 59min | 156h |
| 168h (Day 8.0) | 162h; 173h 59min | 168h |
| 180h (Day 8.5) | 174h; 185h 59min | 180h |
| 192h (Day 9.0) | 186h; 197h 59min | 192h |
| 204h (Day 9.5) | 198h; 209h 59min | 204h |
| 216h (Day 10.0) | 210h; 221h 59min | 216h |
| 228h (Day 10.5) | 222h; 233h 59 min | 228h |
| 240h (Day 11.0) | 234h; 245h 59min | 240h |
| 252h (Day 11.5) | 246h; 257h 59min | 252h |
| 264h (Day 12.0) | 258h; 269h 59min | 264h |
| 276h (Day 12.5) | 270h; 281h 59min | 276h |
| 288h (Day 13.0) | 282h; 293h 59 min | 288h |
| 300h (Day 13.5) | 294h; 305h 59min | 300h |
| 312h (Day 14.0) | 306h; 317h 59min | 312h |

<sup>\*</sup>from first drug intake time; \$ post baseline;

For analyses for which we need at most one assessment per day (e.g.: where BID assessments but daily assessment to be used in the analysis) we take the worst over 24 hours according to Table 4.

<sup>\*</sup> Relative to [Study Day 1]; \*\* on site visits \*\*\* only if symptomatic; ## only for hematology and biochemistry if needed \$ visit windows to be applied as well to RI-PRO, Additional Questions about Health and Functioning when QD scheduled is applicable (from Day 14- 312h and onwards) or if treatment discontinued prematurely but follow up visits are performed; If time of assessment between 00:00 to 01:59, it will be considered as if performed within the previous day. For RI-PRO and Additional Questions about Health and Functioning BID please see also Table 3, Table 4 and Table 5.

| Table 4: Worst per Day |
|------------------------|
|------------------------|

| Analysis time | Primary Selection | Secondary Selection<br>TIME INTERVAL (Day)<br>[TARGET TIMEPOINT (Day)] |
|---|---|---|
| Baseline | | |
| Day 2 | Worst [12h; 24h] | |
| Day 3 | Worst [36h; 48h] | 3<br>[3] |
| Day 4 | Worst [60h; 72h] | |
| Day 5 | Worst [84h; 96h] | 4-6<br>[5] |
| Day 6 | Worst [108h; 120h] | |
| Day 7 | Worst [132h; 144h] | |
| Day 8 | Worst [156h; 168h] | 8-9<br>[8] |
| Day 9 | Worst [180h; 192h] | |
| Day 10 | Worst [204h; 216h] | |
| Day 11 | Worst [228h; 240h] | |
| Day 12 | Worst [252h; 264h] | |
| Day 13 | Worst [276h; 288h] | |
| Day 14 | Worst [300h; 312h] | 13-15<br>[14] |

The secondary selection approach will only be considered in the analysis if no record is assigned to Day 3, Day 5, Day 8 and Day 14 according to the rules in the primary selection column. If 'worst per day' as per primary selection is available, same value will be assigned for the secondary selection of 'worst per day'. Otherwise, 'worst per day' as per secondary selection will be derived considering all possible values within the relative day window. The worst possible results will be selected regardless of being the closest one to target day.

Additionally, each BID assessment is defined as a morning or evening assessment based on the timing of the assessment as defined in Table 5.

Table 5: ePRO Time Slot in a Day

| Slot of the Day | Time |
|-----------------|---------------------|
| Morning | 02:00 am – 13:59 pm |
| Evening | 14:00 – 01:59 am* |

<sup>\*</sup>from 00:00 to 01:59 to be considered as if performed within the previous day.

# 2.1.3. Study Day and Relative Day

Study Day 1 is defined as the date of first study medication intake (reference day). All efficacy and safety assessments at all visits will be assigned a day relative to this date.

For visits on or after the reference day (Day 1) the relative day for a visit is defined as:

$$reldy = visit day - reference day + 1$$

and for visits before the reference day (Day 1)

$$reldy = visit day - reference day$$

There is no 'Day 0'.

### 2.1.4. Baseline

In general, the baseline record is defined as the last record before the first intake of the study drug except for the following assessments where additional rules will be applied:

### • RSV RNA viral load:

- Last available assessment within the 24h prior to or at the same time of first drug intake will be considered as baseline.
- If no assessment within the 24h prior to or at the same time of first drug intake, but there is a result available no later than 1h post first study drug intake, the baseline assessment will be the first assessment completed within 1h post first drug intake.
- If none of the above assessments are available, but there is an assessment available before the 24h prior to first drug intake, it will be considered as baseline.

### • ePRO:

- Last available assessment within the 8h prior to first drug intake.
- if no assessment is available within 8 hours prior to first drug intake, but there is an assessment completed within 1-hour post first intake, then baseline assessment will be the assessment completed within 1-hour post first intake.
- If none of the above assessments are available, but there is an assessment available before the 8h prior to first drug intake, it will be considered as baseline.

If no record available at all before first drug intake, baseline will be considered as missing.

## 2.2. Pooling Algorithm for Analysis Centers

Since it is expected that for this trial subjects will be recruited over a large number of centers with a small number of subjects per study center, there is no need to check for treatment by center interactions. In addition, the primary endpoint is an objective endpoint, which is evaluated by a central assay, no heterogeneity across centers is anticipated. Therefore, there is no need for a pooling algorithm for analysis centers.

### 2.3. Analysis Sets

## 2.3.1. All Randomized Analysis Sets

## 2.3.1.1. All Randomized Analysis (RAND) Set

All randomized subjects with a randomization date regardless of being treated or not.

## 2.3.2. Efficacy Analysis Set(s)

## 2.3.2.1. Intent-To-Treat infected (ITT-i) Set

All randomly assigned subjects who received at least 1 dose of study drug and who have an RSV infection confirmed by a PCR-based assay at the central laboratory at baseline (records up to 1 hour after first medication intake can be used in case no pre-treatment observation is available). Subjects in the ITT-i set will be analyzed according to the treatment they were randomly assigned to.

The ITT-i set definition applies also to the interim analysis. However, if a subject has no central lab confirming the RSV infection at baseline, that subject will not be included in the ITT-i set for the interim analysis purpose.

## 2.3.2.2. Modified Intent-To-Treat infected (mITT-i) Set

All subjects in the ITT-i analysis set with RSV viral load  $\geq 1 \log_{10}$  copies/mL above the Lower Limit of Quantification (LLOQ) at baseline.

## 2.3.2.3. Per Protocol Analysis (PP) Set

All subjects in the ITT-i analysis set with the exclusion of any subjects deemed to have a major protocol deviation that may affect the assessment of efficacy. Such major protocol deviations will be identified, revised and documented prior to database lock based on the following criteria:

- Entered but did not satisfy criteria, violation of:
  - inclusion criteria 4 or 5,
    - AND/OR
  - exclusion criteria 1, 4, 7, 8, 9,14 or 16

Please see Section 4.1 and 4.2 of the protocol for full description of the criteria.

- Received wrong treatment or incorrect dose
  - The actual treatment not the same as the planned treatment
  - Subjects missed more than 1 dose.
- Other:
  - Unplanned unblinding has taken place during the study.

- Insufficient post-baseline viral load samples collected (should have at least baseline and 2 post-dose samples between Day 2 and Day 5).
- Received concomitant treatment that may affect the efficacy of the trial medication.

Complete list of concomitant medications to be considered for major protocol violation will be finalized before the database lock.

Note that in the PP set, subjects will be treated as randomized (by definition). Analyses on the PP set will only be performed if >10% subjects in the ITT-i set are excluded from the PP set.

### 2.3.3. Safety Analysis Set

## 2.3.3.1. Safety Analysis Set (SAF)

The safety analysis set includes all subjects who received at least 1 dose of study agent, analyzed as treated.

The actual treatment is determined as the treatment for which the majority of drug dose is taken.

The Safety set will be used to perform the evaluation of all safety variables and will be used for listings.

## 2.4. Definition of Subgroups

The following subgroups will be investigated for efficacy, including the primary endpoint (viral load) and key clinical course endpoints (duration and severity of sign and symptoms, time to resolution of RSV symptoms and respiratory rate, heart rate, body temperature and peripheral capillary oxygen saturation (SpO<sub>2</sub>). For safety, subgroup analyses will be limited to age group and presence of any comorbid disease associated with risk factors for severe RSV disease.

**Table 6:** Subgroups

| Subgroup | Definition |
|---|---|
| Symptom Onset | • Subjects with symptom onset ≤3 days before randomization |
| | • Subjects with symptom onset >3 days before randomization |
| Baseline RSV Viral Subtype | RSV A |
| | RSV B |
| | • RSV A+B |
| Age | • <65 years and >=65 |
| Baseline Viral Load | Central Viral Load (VL) |
| | • VL≥1 log10 copies/mL above the LLOQ at baseline |
| | • otherwise |
| Presence of any Comorbidities | • No |
| | • Yes |
| Presence of any comorbid disease | • No |
| associated with risk for severe RSV | • Yes |
| disease | |

**Table 6:** Subgroups

| Subgroup | Definition |
|---|---|
| Comorbid diseases associated with risk for severe RSV disease | <ul> <li>Asthma [Yes/No]</li> <li>COPD [Yes/No]</li> <li>CHF [Yes/No]</li> <li>CAD (coronary artery disease) [Yes/No]</li> </ul> |
| Other conditions/therapy of potential interest due to risk of infections in general | <ul> <li>Diabetes mellitus [Yes/No]</li> <li>CRF (Chronic Renal Failure) [Yes/No]</li> <li>Use of systemic corticosteroids prior to or during the treatment phase [Yes/No],</li> </ul> |
| Prior use of systemic corticosteroids Note: use in the 7 days prior to randomization and not continued after first dose | <ul><li>No</li><li>Yes</li></ul> |
| Co-infection Note: based on respiratory pathogens panel assay performed at baseline | <ul><li>No</li><li>Yes</li></ul> |

Subgroup analyses will be performed for efficacy primary endpoint and key clinical course endpoints in case at least 15 subjects are enrolled in any of the subgroup categories.

Medical review will be done immediately before database lock on a list with unique coded medical history terms (MedDRA Preferred Terms) to indicate which subjects had comorbidities.

## 2.5. Imputation Rules for Missing AE Date/Time of Onset/Resolution

Partial AE onset dates will be imputed as follows in derivations, but original information should remain in the database:

- If the onset date of an adverse event is missing day only, it will be set to:
  - First day of the month that the AE occurred, if month/year of the onset of AE is different than the month/year of first dosing of the study medication.
  - The day of first dosing of the study medication, if the month/year of the onset of AE is the same as month/year of the first dosing of the study medication and month/year of the AE resolution date is different.
  - The day of first dosing of the study medication or day of AE resolution date, whichever is earliest, if month/year of the onset of AE and month/year of the first dosing of the study medication and month/year of the AE resolution date are same.
- If the onset date of an adverse event is missing both day and month, it will be set to the earliest of:
  - January 1 of the year of onset, as long as this date is on or after the first dosing of the study medication.

- Month and day of the first dosing of the study medication, if this date is the same year that the AE occurred.
- Last day of the year if the year of the AE onset is prior to the year of the first dosing of the study medication.
- The AE resolution date.

Completely missing onset dates will not be imputed.

Partial AE resolution dates not marked as ongoing will be imputed as follows:

- If the resolution date of an adverse event is missing day only, it will be set to the earliest of the last day of the month of occurrence of resolution or the day of the date of death, if the death occurred in that month.
- If the resolution date of an adverse event is missing both day and month, it will be set to the earliest of December 31 of the year or the day and month of the date of death, if the death occurred in that year.

Completely missing resolution dates will not be imputed.

### 3. INTERIM ANALYSIS AND DATA REVIEW COMMITTEE

## 3.1. Interim Analysis

An interim analysis, encompassing efficacy, safety, and pharmacokinetics is planned after at least 36 subjects have been dosed and have completed the assessments of Day 8, or discontinued earlier. Enrollment will not be paused during the interim analysis.

From the subgroup analyses planned for the final analysis, the following will be included for the interim analysis irrespective of the number of subjects within the subgroup:

- Efficacy analysis: Symptoms onset day
- Safety analysis: age group and presence of any comorbid disease associated with risk factors for severe RSV disease.

Exploratory endpoints will not be included in the interim analysis except for an evaluation of the possible effect of the time since onset of symptoms on antiviral activity and clinical course.

Additional interim analyses may be performed at the sponsor's discretion to support decision making for further development of JNJ-53718678 and to support interactions with health authorities. The primary (final) analysis will be performed after the last subject has completed his/her last visit of the study. Since this is an exploratory, hypothesis-generating study, no adjustments for multiplicity will be performed.

### 3.2. Data Review Committee

A Data Review Committee (DRC), comprised of senior sponsor personnel outside of the central sponsor team and not involved in study conduct, will be established. The DRC will monitor

safety data during study conduct on a regular basis and/or ad hoc in case of emergent safety signals identified through medical monitoring.

The central sponsor team, composed by clinical leader, statistician(s), virologist, PK leader, pharmacometrician and statistical programmers will review the unblinded interim efficacy, safety, and pharmacokinetic analyses and will make recommendations to the DRC regarding possible changes to the design of the study. The DRC will decide on the implementation of the recommendations based on the review of the interim results of the study.

Further details of the DRC, eg, composition and activities, are described in the DRC charter.

### 4. SUBJECT INFORMATION

All subject information analyses will be done on the ITT-i Set and the Safety Set, unless specified otherwise for a specific display (in the DPS).

## 4.1. Demographics and Baseline Characteristics

Table 7 presents a list of the demographic variables that will be summarized by treatment group and overall.

**Table 7:** Demographic Variables

| | Summary Type |
|---|---|
| Continuous Variables: | |
| Age (years) | Descriptive statistics (N, mean, |
| Weight at baseline (kg) | standard deviation [SD], median |
| Height at baseline (cm) | and range [minimum and |
| Body Mass Index <sup>b</sup> at baseline (BMI) $(kg/m^2)$ = weight $(kg)/(height (m))^2$ | maximum]). |
| Categorical Variables | |
| Age (<65 years and >=65) | |
| Sex (male, female) | Frequency distribution with the |
| Race <sup>a</sup> (American Indian or Alaska Native, Asian, Black or African | |
| American, Native Hawaiian or other Pacific Islander, White, Other, | number and percentage of subjects |
| Multiple) | in each category. |
| Ethnicity (Hispanic or Latino, not Hispanic or Latino) | |
| Country | |

If multiple race categories are indicated, the Race is recorded as 'Multiple'. The specifications of the categories 'Other' and 'Multiple' will only be listed.

Symptom Onset at Randomization will be calculated by considering:

- Symptom onset start date and time slot of the day
- Randomization date and time slot of the day

as indicated in Table 8.

Rounded to 1 decimal. Even if available in the raw data, BMI will be calculated from baseline weight and height.

**Table 8:** Time Slot in a Day

| Slot of the Day | Time |
|-----------------|---------------------------------|
| Night | 00:00 midnight – 05:59 am |
| Morning | 06:00 am – 11:59 noon |
| Afternoon | 12:00 noon – 17:59 (or 5:59 pm) |
| Evening | 18:00 – 23:59 |

 $symptom \ onset \ days = randomization \ date - reported \ symptom \ onset \ date + correction \ factor \ for \ time \ of \ the \ day$ 

The correction factor is:

- 0: in case time slot on day of randomization  $\leq$  time slot on day of symptoms
- 1: in case time slot on day of randomization > time slot on day of symptoms

**Table 9:** Correction Factor for Time Slot in a Day

| | Randomization Day | | | |
|-------------------|-------------------|---------|-----------|---------|
| Symptom Onset Day | Night | Morning | Afternoon | Evening |
| Night | 0 | 1 | 1 | 1 |
| Morning | 0 | 0 | 1 | 1 |
| Afternoon | 0 | 0 | 0 | 1 |
| Evening | 0 | 0 | 0 | 0 |

In case the time slot of the day of symptom onset is missing, no correction factor will be applied.

Similar definition will be used to calculate time for symptom onset at first treatment.

Table 10 presents a list of the baseline characteristics that will be summarized by treatment group and overall. Baseline characteristics will also be summarized by presence of comorbidities (yes, no) and by symptom onset (≤3 days, >3 days).

**Table 10:** Baseline Characteristics

| | Summary Type |
|---|---|
| Continuous Variables: | |
| Duration of RSV symptoms prior to randomization (days) | |
| Duration of RSV symptoms prior to first treatment (days) | |
| Baseline RSV Viral Load (log <sub>10</sub> copies/ml) | Descriptive statistics (N, mean, |
| Baseline RSV Viral Load (log <sub>10</sub> copies/ml) by RSV Subtype | standard deviation [SD], median |
| Baseline RSV Viral Load (log <sub>10</sub> copies/ml) by symptom onset day | and range [minimum and |
| Respiratory Rate (breaths/min) | maximum]). |
| Heart Rate (beats/min) | |
| Oxygen Saturation (%) | |
| Categorical Variables | |
| Baseline RSV Subtype (RSV A, RSV B, RSV A+B) | |
| Symptom Onset (≤3 days, >3 days) | |
| Co-infection (no, yes) | |
| Presence of ANY Comorbidities (no, yes) | |
| Comorbid disease associated with risk for severe RSV disease (no, yes) | |
| Each of the following diseases (subcategories of the above): | |
| - Asthma | |
| - COPD | Frequency distribution with the |

**Table 10:** Baseline Characteristics

| | Summary Type |
|---|---|
| - CHF | number and percentage of subjects |
| - CAD | in each category. |
| Other conditions/therapy of potential interest due to risk of infections in | |
| general (yes, no) | |
| Each of the following conditions/therapies (subcategories of the above): | |
| - diabetes mellitus | |
| - CRF | |
| - use of systemic corticosteroids prior to or during the treatment | |
| History of wheezing associated with acute respiratory infection? (no, yes) | |
| Contact with HCP before presenting (no, yes) | |
| If Yes, specify the type of HCP (General Practitioner, Other) | |
| History of Tobacco use (current, former, never) | |

## 4.2. Disposition Information

Summaries will be provided for the following disposition information:

- Number of screen failures, randomized (RAND), randomized and not treated, not randomized and treated, safety set (SAF), ITT-i set and PP set (PPS).
- Number of subjects who completed or discontinued treatment and the study, with a breakdown of the reason of discontinuation.
- Number of subjects per phase and per visit in the trial.

## 4.3. Treatment Compliance

Study treatment compliance will be listed as well as the reasons for non-dispensing assigned drug, or for adjusting the dose.

## 4.4. Extent of Exposure

Extent of exposure (days) is defined as (date of the last dose of study treatment – date of the first dose of study treatment) +1.

Note: treatment interruptions will not be taken into account.

Extent of exposure will be summarized descriptively by treatment group.

### 4.5. Protocol Deviations

Only major protocol deviations will be defined in this trial. All major protocol deviations (please see Section 2.3.2.3 for details) will be tabulated and listed. Those that may affect the assessment of efficacy will be documented prior to database lock.

### 4.6. Medical History

The medical history records will be listed; separate listings will be provided for comorbid diseases associated with RSV.

### 4.7. Prior and Concomitant Medications

Medications taken from the date the ICF is signed through to the end of study will be summarized by preferred term using the World Health Organization-Drug Dictionary as frequency tables in 2 parts:

- 1. Prior medication: medication that started before the first dose of study drug, regardless of when dosing of the medication ended
- 2. Concomitant medication: medication received at or after the first dose of study drug, medication that was received before initial dosing and continued after initial dosing of study drug, or medication with missing stop date.

(Medication that started before the first dose of study drug and continued after the first dose of study drug will be summarized as prior medication and separately as concomitant medication.)

The part on concomitant medication will be shown by ATC class level up to level 3.

If a prior/concomitant therapy record missed components of its start and/or stop dates (time and/or day and/or month and/or year), the following actions will be taken:

- 1. In case of partial start or stop datetimes, the concomitant therapy records will be allocated to prior/concomitant using the available partial information, without imputations.
- 2. In case of a completely missing start date, the prior/concomitant therapy will be considered as having started before the trial.
- 3. In case of a completely missing end date, the prior/concomitant therapy will be considered as ongoing at the end of the trial.

### 4.8. Co-Infections

Data on viral (other than RSV) or bacterial pathogens determined in mid-turbinate nasal swabs collected at screening (both by multiplex PCR) will be listed.

Proportions of positive and negative results will be tabulated by treatment group.

#### 5. EFFICACY

All efficacy will be analyzed on the ITT-i set. The primary endpoint will also be analyzed on mITT-i set and PP set.

The efficacy analyses include the following primary, secondary and exploratory endpoints.

### **Primary Endpoints**

To explore the antiviral effect of JNJ-53718678 on RSV, as measured by qRT-PCR assay in mid-turbinate nasal swabs, the following virologic parameters will be assessed:

- AUC from immediately prior to first dose of study drug (baseline) through Day 3, Day 5, Day 8, and Day 14
- RSV viral load and change from baseline over time

- Time to undetectable RSV viral load
- Proportion of subjects with undetectable RSV viral load at each time point throughout the study.

### **Secondary Endpoints**

- Clinical endpoints:
  - Duration and severity of signs and symptoms of RSV infection assessed through an instrument for patient-reported symptoms (either the Respiratory Infection-Patient Reported Outcomes [RI-PRO] questionnaire or the Respiratory Infection Intensity and Impact Questionnaire [RiiQ] questionnaire) and additional questions about health and functioning
  - Time to resolution of selected RSV symptoms as reported by the subject (through either the RI-PRO or RiiQ)
  - Respiratory rate, heart rate, body temperature, and SpO<sub>2</sub> as measured by the investigator.

### **Exploratory Endpoints**

Exploratory endpoints include:

- Antiviral activity and clinical course by
  - time of symptom onset [ $\leq$ 3 days vs >3 days before randomization]
  - presence of comorbidities
  - baseline RSV viral subtype
  - severity of key RSV symptoms at screening, and
  - baseline RSV genotype
- The occurrence of complications associated with onset after treatment initiation that are associated with RSV per the investigator assessment:
  - Bacterial superinfections (eg, pneumonia, sinusitis, bronchitis, bacteremia of presumed respiratory origin per investigator assessment)
  - Exacerbations of underlying pulmonary disease (eg, asthma, chronic obstructive pulmonary disease [COPD])
  - Exacerbations of underlying cardiovascular conditions
- The need for antibiotics related to complications associated with RSV per investigator assessment
- Sequence changes (post baseline) in the RSV F-gene, and other regions of the RSV genome (if applicable), as compared to baseline
- Medical resource utilization collected as medical encounters
- Association between clinical course of RSV and self-rated HRQOL (ie EQ-5D-5L).

### 5.1. Analysis Specifications

All efficacy summaries will be presented with descriptive statistics by treatment group and scheduled visit unless specified otherwise. In addition, descriptive summaries will be presented by the randomization stratification factor, time of symptom onset (≤3 days vs >3 days before randomization). If the endpoint is continuous, the descriptive statistics will include the number of subjects, mean standard deviation, standard error, median, range and interquartile range. If the endpoint is binary or categorical, the frequency distribution with the number and percentage of subjects in each category will be calculated.

For time to event variables, a summary table including number of subjects included in the analysis, number of subjects censored, 25<sup>th</sup> and 75<sup>th</sup> percentiles and median time-to event will be shown by treatment group.

For all the stratified statistical analyses, the derived randomization stratification factor will be used instead of the randomization stratification factor as collected in the IWRS.

## 5.1.1. Level of Significance

Since this is an exploratory, hypothesis-generating study, no hypothesis testing will be performed. However, two-sided 90% confidence intervals may be calculated without adjustments for multiplicity for comparing active dose groups versus placebo.

## 5.1.2. Data Handling Rules

### Viral Load

Rule of maximum: Before any imputation is applied, the value for each Day is defined as the maximum value of all RSV assessments performed on that day. Please notice that this rule doesn't apply for baseline. For baseline details please see Section 2.1.2.

For analysis purposes, the  $log_{10}$  qRT-PCR viral load will be imputed with the midpoint on the log scale between the limit of detection and lower limit of quantification (LLOQ) when the result is 'target detected' (TD) but non-quantifiable.

- For the RSV-A qRT-PCR assay, the LOD is 620 copies/mL and the LLOQ is 1000 copies/mL, a result that is TD will be imputed with 2.90 log<sub>10</sub> copies/mL.
- For the RSV-B qRT-PCR assay, the LOD is 80 copies/mL and the LLOQ is 250 copies/mL, a result that is TD will be imputed with 2.15 log<sub>10</sub> copies/mL.

When the result is 'target not detected' (TND) (i.e., below the LOD), for both RSV A and RSV B the value of TND will be imputed with 0 log<sub>10</sub> copies/mL.

For the overall analysis of viral load, all the viral load results of the RSV type with which the subject has been infected will be used.

In case of co-infection with both subtypes RSV A and B, the rules below will be applied for the overall analyses of viral load from the time the co-infection is detected (i.e. result of TD or >LLOQ):

- In case of two quantifiable results: the log<sub>10</sub> of the sum of the RSV A and RSV B results in copies/mL will be used.
- In case of a quantifiable result and a TD/TND result: use the imputed TD/TND on the original scale and then use the log<sub>10</sub> of the sum of the quantifiable result and the imputed value. copies/mL scale value and then use the log<sub>10</sub> of the sum of the imputed value and quantifiable result.
- In case of two TD results, or one TD and one TND result: use the imputed TD/TND on the copies/mL scale values and then use the log<sub>10</sub> of the sum of the imputed values.
- In case of two TND results: impute the TND as 0 log<sub>10</sub>.

## 5.2. Primary Efficacy Endpoints – Viral Load

#### 5.2.1. Definition

To explore the antiviral effect of JNJ-53718678 on RSV, as measured by qRT-PCR assay in mid-turbinate nasal swabs, the following virologic parameters will be assessed:

- AUC from immediately prior to first dose of study drug (baseline) through Day 3 (48h), Day 5 (96h), Day 8 (168h), and Day 14 (312h);
- RSV viral load and change from baseline over time;
- Time to undetectable RSV viral load;
- Proportion of subjects with undetectable RSV viral load at each time point throughout the study.

The AUC viral load will be analyzed by two different methods:

- using a restricted maximum likelihood based repeated measures approach (mixed model)
- by trapezoidal method

Terminology is clarified in Table 11.

Table 11: AUC viral load

| Method | |
|-------------|-----------------------|
| Mixed model | Trapezoidal |
| AUC Day 3 | AUC <sub>0-48h</sub> |
| AUC Day 5 | AUC <sub>0-96h</sub> |
| AUC Day 8 | AUC <sub>0-168h</sub> |
| | AUC <sub>0-312h</sub> |

Formulae to be used for derived variables, including data conversions, are provided in the table below. Note that for time-to-event variables the actual dates will be used.

| Measurement | Formula |
|---|---|
| Log <sub>10</sub> viral load actual values | Log <sub>10</sub> of the actual values as measured with qRT-PCR, includin both swabs collected at the clinic visits and at home. |
| values | Sould swads conceived at the crime visits and at nome. |
| Log <sub>10</sub> viral load change | Change = $Log_{10}$ viral load actual value – $log_{10}$ baseline value |
| from baseline | |
| RSV viral load AUC <sub>0-48h</sub> | RSV viral load AUC <sub>0-48h</sub> from 0 hours until 48 hours (Day 3) using |
| [trapezoidal method] | the trapezoidal method (see below). |
| RSV viral load AUC <sub>0-96h</sub> | RSV viral load AUC <sub>0-96h</sub> from 0 hours until 96 hours (Day 5) using |
| 0 7011 | the trapezoidal method (see below). |
| [trapezoidal method] | |
| RSV viral load | RSV viral load AUC <sub>0-168h</sub> from 0 hours until 168h (Day 8) hours |
| AUC <sub>0-168h</sub> | using the trapezoidal method (see below). |
| [trapezoidal method] | |
| RSV viral load | RSV viral load AUC <sub>0-312h</sub> from 0 hours until 312h (Day 14) hours |
| AUC <sub>0-312h</sub> | using the trapezoidal method (see below). |
| [trapezoidal method] | |

| Measurement | Formula | |
|---|---|---|
| Time to virus undetectable (hours) [Time-to event] | Time to virus undetectable will be evaluated using two approaches: 1) The time in hours from initiation of study treatment until the first post-baseline time point at which the virus is undetectable and after which time, no more detectable virus assessment (= event). Situation Censoring | |
| | least, two consecutive undetectable virus assessments. Last obtained sample is always considered confirmed. | |
| | Situation Last record is baseline assessment Last available assessment is | Censoring time 0h (right-censored) at last |
| | (Date and time of event or censoring - date and time of first dose of study drug)/3600, rounded to one decimal. | |
| Viral load status at each time point (categorical) | Each RSV viral load measurement will be assigned to one of the 3 categories below: Undetectable (TND) Detectable (TD) Quantifiable | |
| Viral load status at each time point (binary) | Each RSV viral load measurement will be assigned to one of the 2 categories to identify if it is detectable. • Detectable or quantifiable = Yes (1) • Undetectable = No (0) | |

The trapezoidal method will be used to calculate viral load AUC between 0 and xx hours, based on date times of sampling, including the timepoints with (imputed) values available:
$$AUC_{0-xx \ hours} = \frac{1}{2} \sum_{i=1}^{n} (y_i + y_{i-1}) \times (t_i - t_{i-1})$$

where i=1,2,3,... are the time points when post baseline samples are collected,  $y_i$  is the  $log_{10}$  viral load at the time  $t_i$  and  $t_i$  is the time in hours post baseline.  $y_o$  is the (imputed)  $log_{10}$  viral load at baseline,  $t_0$  is time 0 hours,  $t_n$  is time xx.

The following rules will be applied to deal with missing values before calculating the viral load AUC:

- 1. The value at time point 0h, if not exactly at 0h, will be calculated based on linear interpolation between the last observed pre-dose value and the first observed post-dose value.
- 2. In case the first available observation is after 0 hours, the value at 0h will be imputed by carrying backward the first available observation.
- 3. The value at xx hours, if not exactly at xxh, will be calculated based on interpolation between the last observed value before xxh and the first observed value after xxh.
- 4. In case the last available observation is before xxh, the value at xxh will be imputed by carrying forward the last available observation. Carrying forward should only be performed if the time between the available observation and the value at xxh is at most 24 hours.
- 5. Missing values between 0h and xxh will be imputed by interpolation (automatically by trapezoidal rule).
- 6. In case the last observation is before xxh, and the value at xxh cannot be determined, the AUCs through xxh and through any later timepoint will not be derived.

Note that additionally the AUC will be derived using a mixed model approach.

#### 5.2.2. Analysis Methods

Mean  $\log_{10}$  viral load values over time will be analyzed using a restricted maximum likelihood based repeated measures approach. Analysis will include fixed categorical effects of treatment, strata (symptoms onset [ $\leq 3$  days vs > 3 days before randomization), visit, treatment-by-visit interaction, and the continuous covariates of baseline  $\log_{10}$  viral load and baseline  $\log_{10}$  viral load-by-visit interaction as well as a random effect to model the within-subject error covariance. An unstructured covariance structure will be selected. In case this model will not converge, the Toeplitz covariance structure will be applied. The Kenward-Roger approximation will be used to estimate denominator degrees of freedom.

No imputations of missing data from nasal swabs post-baseline will be done in this model, as this mixed model would allow to make inferences under the *missing at random* assumption. Note that for this analysis only values as provided by the central lab will be used.

To evaluate the difference in the AUC between active and placebo, 3 contrasts will be explored: a contrast with no difference between the 2 active doses tested against placebo; a contrast with no difference between low dose and placebo tested against high dose; and a contrast with a linear

dose-response relationship with respect to the active doses. These contrasts will be used to derive the least square mean differences in the AUCs for active versus placebo, and their 90%CIs, with no multiplicity correction.

#### **RSV RNA Viral Load**

Descriptive statistics, mean (SE) graphs and median (IQR) graphs will be shown for the  $log_{10}$  viral load actual values and changes from baseline by visit and by treatment group.

Differences on RSV RNA log<sub>10</sub> viral load by qRT PCR between treatment groups and by analysis visit will be determined by using appropriate contrasts in a similar repeated measure mixed effects model, including 90% 2-sided confidence intervals.

The potential associations with RSV RNA  $log_{10}$  viral load and the following covariates and/or baseline indicators will be explored graphically:

- baseline log<sub>10</sub> viral load
- smoking history (never/current/former)
- history of wheezing (yes/no)
- presence/absence of comorbid diseases associated with risk for severe RSV disease
- presence/absence of other conditions/therapy of potential interest
- days since symptom initiation (0,1,2,3,4,5)
- RSV subtype
- use of corticosteroids
- supplemental oxygen at baseline
- age as continuous variable.
- severity of key RSV symptoms at screening
- baseline RSV genotype;

The homogeneity of treatment effect on the occurrence of AUC viral load from baseline to Days 3, 5, and 8 across subgroups will be examined using the same MMRM model approach for the primary analysis, but also includes the subgroup-by-treatment and subgroup-by-visit interaction terms in the model. A forest plot will present the Least Square means and 90% CI for all subgroups of interest.

#### **RSV Viral Load AUC**

The individual AUC as calculated using the trapezoidal rule will be considered as a supportive analysis and will be analyzed using a linear model with AUC as a dependent variable and treatment group and stratum as fixed factor and baseline  $log_{10}$  viral load as covariate. The differences versus placebo will be estimated using appropriate contrasts with 90% 2-sided confidence intervals.

## Time to virus undetectable [time-to event]

Time-to event variable will be analyzed and plotted using Kaplan-Meier estimates analysis. The estimate of the hazard ratio (HR) and the 90% confidence intervals for the treatment effect will be provided based on a stratified Cox proportional hazard model (derived randomization stratification factor: ≤3 days, >3 days) and including treatment group as a covariate.

A summary table including number of subjects included in the analysis, number of subjects censored, 25<sup>th</sup> and 75<sup>th</sup> percentiles and median time-to event, with 90% confidence intervals based on the Kaplan-Meier method, will be presented by treatment group.

First approach to evaluate virus undetectable, as described in Section 5.2.1 will considered for this analysis.

The potential impact of selected variables that identify the subgroups of interest on the time to virus undetectable will be assessed by the stratified Cox proportional hazard model. The model will be stratified by the randomization stratification factors and include treatment group and subgroup variable as covariates, and the subgroup by treatment interaction term. A forest plot will present the HRs and 90% CI for all subgroups of interest.

#### Proportion of subjects with undetectable RSV viral load

The proportion of subjects within the RSV RNA viral load categories (undetectable, detectable and quantifiable) will be shown in a frequency tabulation, by treatment group and visit. Subjects with missing data on that analysis visit will not be counted in the denominator for the proportion. The difference in proportions for undetectable versus detectable/quantifiable between each active group and placebo, will be tabulated descriptively (n and % per treatment group), for each post baseline timepoint. Summaries of the difference between groups will include 2-sided 90% confidence intervals based on the Wilson score test.

In case of co-infection with both RSV A and B, the worst category will be used for the analysis. As higher viral loads so denote worse degree of infection, the ordering will be from worst to better namely quantifiable – detectable – undetectable.

Information will also be presented graphically.

#### 5.3. Secondary Endpoints - Clinical Course

Clinical course related endpoints are as follows:

- Duration and severity of signs and symptoms of RSV infection assessed through either the Respiratory Infection Patient Reported Outcome (RI-PRO) or the Respiratory Infection Intensity and Impact Questionnaire [RiiQ] questionnaire, and Additional Questions about Health and Functioning.
- Time to resolution of selected RSV symptoms as reported by the subject through either the RI-PRO or RiiQ.
- Respiratory rate, heart rate, body temperature, peripheral capillary oxygen saturation (SpO<sub>2</sub>) as measured by the investigator.

#### 5.3.1. Definition

#### 5.3.1.1. ePROs

RI-PRO, RiiQ, and Additional Questions about Health and Functioning and EQ-5D-5L will be collected from Screening to Day 21. RI-PRO, RiiQ, and Additional Questions about Health and Functioning are completed twice daily (morning and evening) from Day 1 to Day 13.

Note: RiiQ will be completed only by subjects enrolled after the approval of Protocol-Amendment 1. These subjects will complete RI-PRO only at Screening/Baseline and Day 8.

Considering the two scales (RI-PRO and RiiQ) used in the study, the below table reflects the one to one mapping of the key RSV symptom items in RI-PRO to those of the RiiQ that will be used in the analyses.

The RI-PRO key RSV symptoms are as follows: congested or stuffy nose, sore or painful throat, trouble breathing, chest tightness, coughing, coughed up mucus or phlegm, weak or tired.

The RiiQ key RSV symptoms are as follows: nasal congestion, sore throat, short of breath, wheezing, cough, coughing up phlegm (sputum), fatigue (tiredness).

| RI-PRO domain | RI-PRO items<br>(key items) | RiiQ symptom domain items (key items) |
|---|---|---|
| Nose | Runny or dripping nose Congested or stuffy nose Sneezing Sinus pressure | Nasal congestion |
| Throat | Scratchy or itchy throat Sore or painful throat Difficulty swallowing | Sore throat |
| Eyes | Teary or watery eyes Sore or painful eyes Eyes sensitive to light | |
| Chest/Respiratory | Trouble breathing Chest congestion Chest tightness Dry or hacking cough Wet or loose cough Coughing Coughed up mucus or phlegm | Wheezing Short of breath Cough Coughing up phlegm (sputum) |
| Gastrointestinal | Felt nauseous<br>Stomach ache<br>Vomit (frequency)<br>Diarrhea (frequency) | |

| Body/Systemic | Felt dizzy | |
|---------------|--------------------------|----------------------|
| | Head congestion | |
| | Headache | Headache |
| | Lack of appetite | Loss of appetite |
| | Sleeping more than usual | Interrupted sleep |
| | Body aches or pains | Body aches and pains |
| | Weak or tired | Fatigue (tiredness) |
| | Chills or shivering | Feeling feverish |
| | Felt cold | |
| | Felt hot | |
| | Sweating | |
| | | Neck pain |

Formulae to be used for derived variables, including data conversions, are provided in the table below. Note that for time-to-event variables the actual date times will be used.

| Measurement | Formula | |
|---|---|---|
| 1 | PATIENT REPORTED OUTCOMES | |
| RI-PRO | | |
| RI-PRO domain scores + | RI-PRO is a 32 i | items questionnaire computed in six domain |
| change from baseline | scores, representing | g symptom severity in each of the following |
| | body areas as follow | vs: |
| | Domain | Score calculation |
| | Nose | Arithmetic mean of the available items. |
| | | Score will be calculated if at least 3 out of 4 |
| | | items are available, otherwise it will be set to |
| | | missing. |
| | Throat | Arithmetic mean of the available items. |
| | | Score will be calculated if at least 2 out of 3 |
| | | items are available |
| | Eyes | Arithmetic mean of the available items. |
| | | Score will be calculated if at least 2 out of 3 |
| | | items are available, otherwise it will be set to |
| | | missing. |
| | Chest/ | Arithmetic mean of the available items. |
| | Respiratory | Score will be calculated if at least 5 out of 7 |
| | | items are available, otherwise it will be set to |
| | | missing. |
| | Gastrointestinal | Arithmetic mean of the available items. |
| | | Score will be calculated if at least 3 out of 4 |
| | | items are available, otherwise it will be set to |

| Measurement | Formula | | |
|---|---|---|---|
| | Body/Systemic | Score will b | nean of the available items. be calculated if at least 8 out of e available, otherwise it will be g. |
| | Each RI-PRO dom<br>(very severe symptom | ain score ran | ges from 0 (symptom free) to 4 |
| | Please see Attachmo | ent [3]. | |
| RI-PRO key symptom<br>score + change from<br>baseline | nose, sore or pain coughing, coughed | ful throat, tro | 7 key items (congested or stuffy buble breathing, chest tightness, phlegm, weak or tired) will be ms are available, otherwise it will |
| Daily average RI-PRO<br>domain scores + change<br>from baseline | | ulate the avera | ch of the items within a domain, age of the RI-PRO domain scores |
| Time to resolution of selected RSV symptoms | Time (in hours) from resolution of RSV s | | f study drug until the first time of |
| from RI-PRO (hours) [Time-to event] | Resolution of RSV symptoms occurs when items within a selected domain in the RI-PRO are scored as 'Not at all' (score = 0) or 'A little bit' (score =1) (ie alleviated) for at least 24 hours. | | |
| | Selected domains to consider are nose, throat, chest/respiratory and body/systemic symptoms. | | |
| | required, if the before the second Day 13. These 3 over 4 schedule timepoint is allow | e first (of the ond analysis to consecutive to consecutive to wed. | ings indicating resolution are ese 3 consecutive) recording is impoint of the BID schedule at recordings should have been done e analysis timepoints, 1 missing indicating resolution are |
| | required, <b>if the first</b> (of these 2 consecutive) recording is <u>at after</u> the second analysis timepoint of the BID schedule at D 13. These 2 consecutive recordings should have been done ov 3 scheduled consecutive analysis timepoints, 1 missi timepoint is allowed | | 2 consecutive) recording is <u>at or</u> epoint of the BID schedule at Day dings should have been done over |
| | In case RSV symptoms are not resolved, data will be censored. | | |
| | Censoring will be d | | <u>:</u> |
| | Situatio | | Censoring |
| | Last record(s) indi | cate | first record of resolution from |

| Measurement | Formula | |
|---|---|---|
| | resolution of RSV symptoms <b>but</b> insufficient recordings to meet the time to resolution | the last series of recordings of resolution of RSV symptoms |
| | Last record does not indicate resolution of RSV symptoms | after the last observation, at 20:00 on the same day if the last observation was a morning diary entry (from 02:00 until 13:59) |
| | | at 8:00 the next day if the last<br>entry was an evening diary<br>(from 14:00 until 01:59) |
| | Death (without previous | date of death. |
| | resolution) | If time is not available, it will be imputed as per 00:01 of the date of death |
| | missing information to | date of hospitalization |
| | determine resolution or resolution of symptoms because of hospitalization | If time is not available, it will be imputed as per 00:01 of the date of hospitalization |
| | (Date and time of event or censor study drug)/3600, rounded to one | ing - date and time of first dose of decimal |
| Time to complete resolution of selected RSV | Time (in hours) from first dose resolution of RSV symptoms. | of study drug until first complete |
| symptoms from RI-PRO (hours) [Time-to event] | _ | ptoms occurs when items within a are scored as 'Not at all' (score = |
| | Censoring will be applied as defin | ned above. |
| Time to resolution of all RSV symptoms from RI- | Time (in hours) from first dose o resolution of RSV symptoms. | f study drug until the first time of |
| PRO (hours) [Time-to event] | 1 | occurs when all items within a ed as 'Not at all' (score=0) or 'A of for at least 24 hours. |
| | Censoring will be applied as defin | ned above. |
| Time to complete resolution of all RSV | Time (in hours) from first dose resolution of all RSV symptoms. | of study drug until first complete |
| symptoms from RI-PRO (hours) [Time-to event] | | ymptoms occurs when all items are scored as 'Not at all' (score = |

| Measurement | Formula | |
|---|---|---|
| | Censoring will be applied as defined above. | |
| Time to resolution of key RSV symptoms from RI- | Time (in hours) from first dose of study drug until the first time of resolution of key RSV symptoms. | |
| PRO (hours) [Time-to event] | 1 | SV symptoms occurs when all 7 key items are ll' (score = 0) or 'A little bit' (score =1) (ie st 24 hours. |
| | Censoring will be ap | plied as defined above. |
| Time to complete resolution of key RSV | Time (in hours) from resolution of all 7 ke | om first dose of study drug until complete by RSV symptoms. |
| symptoms from RI-PRO (hours) [Time-to event] | Complete resolution of key RSV symptoms occurs when all items within a domain in the RI-PRO are scored as 'Not at all' (score = 0) for at least 24 hours. | |
| | Censoring will be ap | plied as defined above. |
| RiiQ | l | |
| RiiQ symptom score + change from baseline | RiiQ symptom domain is a 13 items questionnaire which ranges from 0 (symptom free) to 3 (severe symptoms). Arithmetic mean will be calculated if at least 9 out of 13 items are available, otherwise it will be set to missing. Please see Attachment [3]. | |
| RiiQ key symptom score + change from baseline | Arithmetic mean of the following 7 key items (nasal congestion, sore throat, short of breath, wheezing, cough, coughing up phlegm [sputum], fatigue [tiredness]) will be calculated if at least 5 out of 7 items are available, otherwise it will be set to missing. | |
| Daily average RiiQ<br>symptom score + RiiQ key<br>symptom score + change<br>from baseline | The worst result observed for each of the items will be used to calculate the average of the RiiQ symptom score per day (in case of BID). | |
| RiiQ impact scores + change from baseline | There are 3 RiiQ impact domains: Daily activity (7 items), Emotions (4 items), and Relationship (5 items). Each item ranges | |
| | from 0 (no impact) to 3 (severe impact). | |
| | Domain | Score calculation |
| | Daily activity | Arithmetic mean will be calculated if at least 5 out of 7 items are available, |
| | | otherwise it will be set to missing. |
| | Emotions | Arithmetic mean will be calculated if at |
| | | least 3 out of 4 items are available, otherwise it will be set to missing. |
| | Relationship | Arithmetic mean will be calculated if at |

| Measurement | Formula |
|---|---|
| | least 3 out of 5 items are available, otherwise it will be set to missing. |
| Time to resolution of all RSV symptoms from RiiQ | Time (in hours) from first dose of study drug until the first time of resolution of all RSV symptoms. |
| (hours) [Time-to event] | Resolution of RSV symptoms occurs when all items within the symptom domain of RiiQ are scored as 'None' (score = 0) or 'Mild' (score = 1) for at least 24 hours. |
| | Censoring will be applied as defined above. |
| Time to complete resolution of all RSV | Time (in hours) from first dose of study drug until first complete resolution of all RSV symptoms. |
| symptoms from RiiQ<br>(hours) [Time-to event] | Complete resolution of RSV symptoms occurs when all items within the symptom domain of the RiiQ are scored as 'None' (score = 0) for at least 24 hours. |
| | Censoring will be applied as defined above. |
| Time to resolution of key RSV symptoms from RiiQ | Time (in hours) from first dose of study drug until the first time of resolution of all 7 key RSV symptoms. |
| (hours) [Time-to event] | Resolution of key RSV symptoms occurs when all 7 key items within the symptom domain of the RiiQ are scored as 'None' (score = 0) or 'Mild' (score = 1) for at least 24 hours. |
| | Censoring will be applied as defined above. |
| Time to complete resolution of key RSV | Time (in hours) from first dose of study drug until first complete resolution of all 7 key RSV symptoms. |
| symptoms from RiiQ<br>(hours) [Time-to event] | Complete resolution of RSV symptoms occurs when all 7 key items within the symptom domain in the RiiQ are scored as 'None' (score = 0) for at least 24 hours. |
| | Censoring will be applied as defined above. |
| Common endpoints for RI-PRO and RiiQ | |
| Key RSV symptom score<br>from either RI-PRO or<br>RiiQ + daily average +<br>change from baseline | Arithmetic mean of the key items from either RI-PRO or RiiQ will be calculated if at least 10 out of 14 items are available, otherwise it will be set to missing. When a key item is available in both RI-PRO and RiiQ, only the key item from RiiQ will be considered. |
| | The worst result observed for each of the items will be used to calculate the average of the RI-PRO or RiiQ symptom score per day (in case of BID). |
| Time to resolution of key<br>RSV symptoms (hours)<br>from either RI-PRO or | Time (in hours) from first dose of study drug until the first time of resolution of all 7 key RSV symptoms from either RI-PRO or |

| Measurement | Formula | |
|---|---|---|
| RiiQ [Time-to event] | RiiQ. | |
| | | ms occurs when all 7 key items scored as 0 or 1 (ie alleviated) for |
| | Censoring will be applied as defin | ned above. |
| Time to complete<br>resolution of key RSV<br>symptoms (hours) from<br>either RI-PRO or RiiQ | | e of study drug until complete<br>emptoms from either RI-PRO or |
| [Time-to event] | _ | RSV symptoms occurs when all 7 r RiiQ are scored as 0 for at least |
| | Censoring will be applied as defin | ned above. |
| Additional Questions Abou | t Health and Functioning | |
| Additional questions about health and functioning | Nine items (please see Attac<br>functioning. | chment [3]) about health and |
| Time to return to usual activity (hours) [Time-to- | Time (in hours) from the first dose of study drug until the time of return to usual activity. | |
| event] | · - | when the response is 'Yes' on RI-<br>ave you returned to your usual<br>hours. |
| | these 3 consecutive) recording timepoint of the BID schedul recordings should have consecutive analysis timepallowed. • Two consecutive recordings 2 consecutive) recording is timepoint of the BID schedul recordings should have consecutive analysis timepoint | ts, 1 missing timepoint is allowed |
| | In case return to usual activit censored. | y is not reached, data will be |
| | Censoring will be done as follows | <u>s</u> : |
| | Situation | Censoring |
| | Last record(s) indicate return to usual activity <b>but</b> insufficient recordings to meet | first record of return from the last series of recordings of return to usual activity. |

| Measurement | Formula | |
|---|---|---|
| | the time to return to usual activity | |
| | Last record does not indicate return to usual activity | after the last observation, at 20:00 on the same day if the last observation was a morning diary entry (from 02:00 until 13:59) |
| | | at 8:00 the next day if the last entry was an evening diary (from 14:00 until 01:59) |
| | Death (without previous return | date of death. |
| | to usual activity) | If time is not available, it will be imputed as per 00:01 of the date of death |
| | missing information to | date of hospitalization |
| | determine return to usual activity because of hospitalization | If time is not available, it will be imputed as per 00:01 of the date of hospitalization |
| | (Date and time of event or censor study drug)/3600, rounded to one | ing - date and time of first dose of decimal |
| Time to return to usual health (hours) [Time-to- | Time (in hours) from the first do return to usual health. | se of study drug until the time of |
| event] | | then the response is 'Yes' on RI-<br>rave you returned to your usual ars. |
| | these 3 consecutive) recording timepoint of the BID schedul recordings should have consecutive analysis timep allowed. • Two consecutive recordings 2 consecutive) recording is | ngs are required, if the first (of the second analysis the at Day 13. These 3 consecutive the been done over 4 scheduled oints, 1 missing timepoint is are required, if the first (of these that or after the second analysis the at Day 13. These 2 consecutive |
| | consecutive analysis timepoin | been done over 3 scheduled its, 1 missing timepoint is allowed |
| | In case return to usual health is no | ot reached, data will be censored. |
| | Censoring will be done as follows | <u>s</u> : |

| Measurement | Formula | |
|---|---|---|
| | Situation | Censoring |
| | Last record(s) indicate return<br>to usual health <b>but</b> insufficient<br>recordings to meet the time to<br>return to usual health | first record of return from the last series of recordings of return to usual health. |
| | Last record does not indicate return to usual health | after the last observation, at 20:00 on the same day if the last observation was a morning diary entry (from 02:00 until 13:59) |
| | | at 8:00 the next day if the last<br>entry was an evening diary<br>(from 14:00 until 01:59) |
| | Death (without previous return | date of death. |
| | to usual health) | If time is not available, it will<br>be imputed as per 00:01 of the<br>date of death |
| | missing information to | date of hospitalization |
| | determine return of usual health because of hospitalization | If time is not available, it will be imputed as per 00:01 of the date of hospitalization |
| | (Date and time of event or censor study drug)/3600, rounded to one | ing - date and time of first dose of<br>decimal |
| 5-level EuroQol 5-Dimension | on Questionnaire (EQ-5D-5L) | |
| EQ-5D dimension parameters: Mobility, | | ed by the following dimensions: vities, pain/discomfort, anxiety/evel score from 1 to 5. |
| Self-care, | • no problems (level code = | 1), |
| Usual activities, | slight problems (level cod | e = 2), |
| Pain/discomfort, | moderate problems (level | code = 3), |
| Anxiety/depression | severe problems (level cod | de = 4), |
| | extreme problems (level c | ode = 5)). |
| | Please see Attachment [4]: EQ | -5D-5L for further details. |
| EQ-5D VAS | EQ-5D VAS is a continuous sec<br>you can imagine) to 100 (best hea | ore ranging from 0 (worst health alth you can imagine). |
| EQ-5D Valuation index | EQ-5D Valuation index summ | narizes the information of the |

| Measurement | Formula |
|---|---|
| | 5 dimensions of the descriptive system. |
| | O Assign the level code 1, 2, 3, 4 and 5 to each level of the 5 dimensions (see Attachment [4]: EQ-5D-5L) |
| | <ul> <li>Create a health state for each patient-time point combination.</li> <li>A health state is a combination of 5 level codes; one level code for each dimension. The dimensions are ordered as described in the table above.</li> </ul> |
| | E.g. health state 12543 indicates 'no problems walking, slight problems washing or dressing myself, unable to do my usual activities, severe pain or discomfort, moderately anxious or depressed'. |
| | Assign an index value to each health state as defined in Respiratory where EQ-5D health state is converted to a single summary index by applying a formula that essentially attaches weights to each of the levels in each dimension. The algorithm is based on the valuation of EQ-5D health states using the UK TTO (=time trade-off method) based value set. |

# 5.3.1.2. Clinical Course Endpoints related to Respiratory, Heart Rate and Body Temperature

# 5.3.1.2.1. Respiratory Rate, Heart Rate, Oxygen Saturation and Body Temperature

| Measurement | Formula |
|---|---|
| Clinical Course Endpoints | related to Respiratory, Heart Rate and Body Temperature |
| Respiratory Rate actual values + changes from baseline | Actual values of Respiratory Rate measured at baseline/Day 1, Day 3, Day 8, Day 14 and Day 21. |
| Respiratory Rate status at each visit (binary) | Each measurement will be assigned to one of the 2 categories to identify if the respiratory rate is normalized to the pre-RSV disease status, rated by the investigator at baseline/Day 1, Day 3, Day 8, Day 14 and Day 21. Normalization of respiratory rate (RR) will be derived from the |
| | answer to the corresponding question in the eCRF "Is this value similar to the pre-RSV infection value for this patient?" • Yes → Normalized (0) |

| Measurement | Formula |
|---|---|
| | No → Abnormal (1) |
| Heart Rate actual values + changes from baseline | Heart Rate measured at baseline, Day 3, Day 8, Day 14 and Day 21. |
| Heart Rate status at each visit (binary) | Each measurement will be assigned to one of the 2 categories to identify if the heart rate is normalized to the pre-RSV disease status, rated by the investigator at baseline, Day 3, Day 8, Day 14 and Day 21. Normalization of heart rate (HR) will be derived from the answer to the corresponding question in the eCRF "Is this value similar to the pre-RSV infection value for this patient?" • Yes → Normalized (0) |
| | • No $\rightarrow$ Abnormal (1) |
| Oxygen Saturation actual values + changes from baseline | Oxygen Saturation measured at baseline, Day 3, Day 8, Day 14 and Day 21. |
| Oxygen Saturation status at each visit (binary) | Each measurement will be assigned to one of the 2 categories to identify if the oxygen saturation is normalized to the pre-RSV disease status, rated by the investigator at baseline/Day 1, Day 3, Day 8, Day 14 and Day 21. |
| | Normalization of oxygen saturation (SpO2) will be derived from the answer to the corresponding question in the eCRF "Is this value similar to the pre-RSV infection value for this patient?" |
| | • Yes → Normalized (0) |
| | • No → Abnormal (1) |
| Body Temperature actual values + changes from baseline | Body Temperature measured at on-site clinic visits (baseline, Day 3, Day 8, Day 14 and Day 21), as well as measured at home. |

# 5.3.1.2.2. Other Clinical Course Parameters

| Measurement | Formula |
|---|---|
| Other Clinical Course Para | ameters |
| Need for Oxygen<br>supplementation | Subjects who required supplemental oxygen after first dose of study drug and who's answer to the question "Has supplemental oxygen administration returned to that level provided prior to the current respiratory infection?" is 'No', will receive code 1. Subjects who did not require supplemental oxygen or for who the level returned to the level provided prior to the current respiratory infection, will receive code 0. |
| Respiratory infection complication | Subjects who experienced a respiratory infection complication after first dose of study drug will receive code 1, subjects who did not experience a complication will receive code 0. |
| | The overall category will consist of any complication (answer to the question: "Is this AE a complication related to the current respiratory infection?"). |
| | The following subcategories will also be analyzed: Respiratory complications, including Bacterial complications Viral complications Non-respiratory infectious complications, including Bacterial complications Viral complications |
| | <ul><li>Metabolic complications</li><li>Other</li></ul> |
| Wheezing status | Investigator will evaluate the subject's wheezing at on-site visits Screening/baseline, Day 3, Day 8, Day 14 and Day 21 as per information collected in the eCRF under: |
| | "Describe the subject's wheezing now" |
| | <ul> <li>No wheezing</li> <li>Terminal expiratory wheezing or only with stethoscope</li> <li>Entire expiration or audible during expiration without stethoscope</li> <li>Inspiration and expiration without stethoscope</li> </ul> |

| Measurement | Formula |
|---|---|
| | "On auscultation are the following present" |
| | <ul> <li>Rales (crackles) → Yes/No</li> <li>Ronchi → Yes/No</li> </ul> |

# 5.3.2. Analysis Methods

# 5.3.2.1. Endpoint-specific analysis methods

#### RI-PRO and RiiQ domain scores and daily average domain scores

Descriptive statistics, mean (SE) graphs and median (IQR) graphs will be shown for the actual values and changes from baseline for both Ri-PRO and RiiQ scores.

Changes from baseline on each of the RI-PRO and RiiQ domain scores will be analyzed using a restricted maximum likelihood based repeated measures approach as per Section 5.2.2. An unstructured covariance structure will be selected.

# **Additional Questions about Health and Functioning**

Frequency tabulations for the 9 additional questions about health and functioning will provided.

## EQ-5D-5L VAS

Frequency tabulations of the EQ-5D-5 L dimensions will be provided.

EQ-5D VAS descriptive statistics for the actual values and changes from baseline will be summarized.

Changes from baseline at each day of assessment will be analyzed using a restricted maximum likelihood based repeated measures approach as per Section 5.2.2. An unstructured covariance structure will be selected

#### Respiration Rate, Heart Rate, Oxygen Saturation and Body Temperature

Descriptive statistics, mean (SE) graphs and median (IQR) graphs will be shown for the actual values and changes from baseline by visit and by treatment group.

#### Respiration Rate Status, Heart Rate Status and Oxygen Saturation Status

The proportion of subjects within the two categories (abnormal, normalized) for each status (respiration rate, heart rate, and oxygen saturation) will be shown in a frequency tabulation by treatment group and analysis time point. The difference in proportions for abnormal status between each active group and placebo will be tabulated, and summaries will include 2-sided 90% confidence intervals based on the Wilson score test.

Subjects with missing data on that analysis visit will not be counted in the denominator for the proportion.

## Need of Oxygen supplementation

The requirement for oxygen supplementation will only be calculated for those subjects that don't require oxygen supplementation before first dose of study drug.

The proportion of subjects with oxygen supplementation (yes and no) will be shown in a frequency tabulation by treatment group. The difference in proportions between each active group and placebo will be tabulated, summaries will include 2-sided 90% confidence intervals based on the Wilson score test.

Note that these incidences are only analyzed if any subjects require oxygen supplementation.

## **Respiratory infection complication**

The proportion of subjects with presence/absence of complications (overall category and subcategories) will be shown in a frequency tabulation by treatment group including a column for the total JNJ-8678 irrespective of the doses.

Note that these incidences are only analyzed if any subjects have complications occur.

# <u>Time to resolution of symptoms, Time to return to usual health and Time to return to usual activity</u>

Time-to event variable will be analyzed and plotted using Kaplan-Meier estimates analysis. The estimate of the hazard ratio (HR) and the 90% confidence intervals for the treatment effect will be provided based on a stratified Cox proportional hazard model (derived randomization stratification factor: ≤3 days, >3 days) and including treatment group as a covariate. Due to limited available RiiQ data, these analyses will not be applied to the RiiQ time to event variables.

A summary table including number of subjects included in the analysis, number of subjects censored, 25<sup>th</sup> and 75<sup>th</sup> percentiles and median time-to event, with 90% confidence intervals based on the Kaplan-Meier method, will be presented by treatment group.

The potential impact of selected variables that identify the subgroups of interest on the time to resolution of symptoms will be assessed by the stratified Cox proportional hazard model. The model will be stratified by the randomization stratification factors and include treatment group and subgroup variable as covariates, and the subgroup by treatment interaction term. A forest plot will present the HRs and 90% CI for all subgroups of interest.

#### **Breathing Sounds**

Frequency tabulations of each wheezing status will be provided by treatment group and visit.

The proportion of subjects with Rales and Ronchi (yes and no) will be shown in a frequency tabulation by treatment group. The difference in proportions between each active group and

placebo will be tabulated, summaries will include 2-sided 90% confidence intervals based on the Wilson score test

# 5.4. Sensitivity Analyses

As a sensitivity analysis, the analysis on change from baseline on Day 3 and Day 8 will be repeated but excluding viral load data not collected by a Health Care Professional (HCP). If different results will be observed from this sensitivity and the primary analysis, then additional analyses may be performed to investigate further.

Time to virus undetectable will be also repeated but considering the second approach (please see Section 5.2.1) to evaluate virus undetectable.

Sensitivity analyses to assess the robustness of the primary efficacy analysis of viral load AUC will be performed by including the stratification factor, RSV symptom onset ( $\leq$ 3 days or > 3 days), as collected by the IWRS in the mixed-effects model. Additionally, the primary efficacy analysis will be repeated on the mITT-I set.

For the time to resolution of selected RSV symptoms of RI-PRO, sensitivity analyses will be performed considering 4 different imputation methods:

- Method 1: from first resolution (score 0 or 1) after last unresolved value onwards, impute missing data as resolution.
- Method 2: impute all missing values as unresolved (score >1).
- Method 3: impute all missing values in-between resolved observations (score 0 or 1) as resolved
- Method 4: impute all missing values as unresolved (score >1), except when in-between resolved values where resolved is imputed.

# 5.5. Other Efficacy Variable(s)

#### 5.5.1. Definition

| Measurement | Formula |
|---|---|
| Need for antibiotics related to complications associated with RSV | Need for antibiotics is defined as 'Yes' if the answers to the following 4 questions on the AE page in the eCRF are answered with 'Yes' to all of them. |
| | • Is this AE a complication related to the current respiratory infection? |
| | • Is this an infection? |
| | • If yes, was infection treated with oral or parenteral antibiotics? |
| | If yes, specify the type of complication "Respiratory Complications" |

54

## 5.5.2. Analysis Methods

Summary tables will be presented by treatment group, stratification factor and visits.

# Need for antibiotics related to complications associated with RSV

The proportion of subjects with a need for antibiotics (yes and no) will be shown in a frequency tabulation. The difference in proportions between each active group and placebo will be tabulated, summaries will include 2-sided 90% confidence intervals based on the Wilson score test

# 5.6. Exploratory Analyses

Relationships between primary antiviral effect endpoints and clinical course endpoints will be investigated as follows

Antiviral activity endpoints:

- RSV RNA log<sub>10</sub> viral load AUCs.
- Time to virus undetectable.
- Time to virus confirmed undetectable

Clinical course endpoints:

- RI-PRO score per domain
- Key RSV symptom score from RI-PRO
- Key RSV symptom score from either RI-PRO or RiiQ (if available RiiQ data)
- Time to resolution of selected RSV symptoms from RI-PRO
- Time to resolution of key RSV symptoms from RI-PRO
- Time to resolution of key RSV symptoms from either RI-PRO or RiiQ (if available RiiQ data)
- Time to resolution of all RSV symptoms from RI-PRO
- EQ-5D-5L each dimension and Visual Analog Scale

The relationships for each pair of variables described above will be explored using the Spearman's rank correlation coefficients. Scatterplots with smoother curve per treatment group will be used for continuous and time-to-event variables (ignoring censoring). Boxplots will be created to graphically present the association between continuous and binary variables. For association between time-to-event clinical course parameters and continuous or binary variables, Kaplan-Meier plots will be generated by quartiles of the continuous variable, or by yes/no status of the binary variable, respectively.

The association between each EQ-5D-5L dimension and time to alleviation will also be explore using the spearman's rank correlation coefficient and graphically.

#### 6. SAFETY

All safety analyses will be done on the Safety Set.

#### 6.1. Adverse Events

All safety analyses will be done on the Safety Set.

#### 6.1.1. Definitions

#### **Coding of AE**

The verbatim terms used in the eCRF by investigators to identify AEs will be coded using the Medical Dictionary for Regulatory Activities. Events are looked at on the level of their preferred term.

#### **Emergent Adverse Event**

Emergent AEs are AEs with onset after first study medication intake or that are a consequence of a pre-existing condition that has worsened since baseline. All reported emergent AEs will be included in the analysis. For each AE, the percentage of subjects who experience at least 1 occurrence of the given event will be summarized by treatment group.

#### **Phase allocation of AE**

Adverse events present in the SDTM database are allocated to phases based on their start date. If the start date of an event falls between (or on) the start and stop date of a phase, the AE is attributed to that phase (emergent principle).

Incomplete dates (i.e. time and/or day and/or month and/or year missing) are imputed according to the rules in Section 2.5.

## 6.1.2. Analysis Methods

Treatment-emergent adverse events will be summarized by body system, preferred term and treatment group (including a column for total JNJ-8678).

A summary will be provided for the following emergent adverse events by phase (treatment phase, follow-up phase) and by treatment:

- any adverse events,
- serious adverse events,
- deaths due to AE,
- adverse events by toxicity grade,
- AEs at least possibly related to study medication,
- AEs for which study medication was permanently stopped,
- AEs for which study was discontinues prematurely.
- serious adverse events that were at least possibly related to study medication.

There will be no formal statistical testing.

Incidence tabulations will be provided for individual adverse events in the above categories (in case there are at least 5 events). Additionally, tabulation of AEs of at least grade 2 and considered related to study drug will be provided.

Listings will be provided for at least the following categories: all AEs, serious AEs, AEs leading to death, AEs leading to permanent stop, grade 3-4 AEs.

The summary, incidence tabulation for the individual preferred terms and subject listing will be provided for the RSV-related complications.

The following adverse events will be tabulated; or listed (in case there are less than 5 events) by subgroups (see Section 2.4): any AE, any RSV-related complications, any grade 3-4 AE, AEs that are at least possibly related to study medication, AEs leading to death, serious AEs, AEs leading to permanent stop of study medication.

## 6.2. Clinical Laboratory Tests

#### 6.2.1. Definitions

Laboratory parameters of hematology, serum chemistry and urinalysis will be investigated: All analyses will be done on SI-converted values as available in the database.

**Coagulation function** will be monitored during this study through evaluation of partial thromboplastin time (PTT) activated partial thromboplastin time (aPTT) in seconds and of the International normalized ratio

**Renal Function** will be monitored during the study through evaluation of the estimated Glomerular Filtration (eGFR) based on:

- Serum creatinine by Cockcroft-Gault formula
   C<sub>Cr</sub> (mL/min) = sex \* [(140 age) \* weight(kg) / 72 \* S<sub>Cr</sub>(mg/dL)]; if female, correction factor is 0.85
- Serum cystatin C GFR (mL/min/1.73m<sup>2</sup>) = 84.69 \* cystatin C (mg/L)<sup>-1.680</sup>

#### **Toxicity grades and abnormalities for laboratory parameters:**

The laboratory abnormalities will be determined according to the DMID adult toxicity grading scale (see Attachment [3]), available toxicity grades provided by the central lab (Covance) will be used. In case no toxicity grades are defined for a test, the abnormalities (above/below normal range) will be used.

In determining toxicity grades/abnormalities for each subject the following rules are applied:

- Worst grades/abnormalities are determined over the whole observational period, per phase (treatment, follow-up and combination treatment + follow-up), including unscheduled measurements.
- The abnormalities "abnormally low" and "abnormally high" are considered equally important, i.e. if a subject has as well an abnormally low as an abnormally high value post-baseline, both abnormalities are shown in the tables. (This means that the sum of the percentages can be more than 100%).
- If, for a specific test, the grading list provides distinct limits for abnormally low (=hypo) values as well as for abnormally high (=hyper) values, this test should be repeated for hyper and hypo limits separately in cross-tabulations.

#### **Emergent definition for toxicity grades and abnormalities**

An abnormality (toxicity grade or abnormality based on normal ranges) will be considered emergent if it is worse than the baseline abnormality. If the baseline abnormality is missing, the abnormality is always considered as emergent. A shift from "abnormally low" at baseline to "abnormally high" post baseline (or vice versa) is also emergent. The emergent definition is applicable in both, the treatment and follow-up phase.

# In case of missing date or partial dates

Laboratory records with missing assessment date- or partially missing (any: day, month or year) will not be used in descriptive statistics, unless the scheduled target day or time is known, and a unique phase allocation is possible taking this additional information into account. These assessments will be allocated to the correct phase using the available date information, and the information on their assessment schedule. In case it is not possible to assign a unique phase (e.g. unscheduled time points), the assessment will be assigned to all possible active phases based on the available date and time information. These cases will be flagged in the respective listings.

# **Imputations of numerical values expressed as characters**

In case a laboratory test result is censored (no numeric value is available, but only a verbatim term), the following rules are applied:

- '<x' or '>x': a numeric value will be imputed by a value exceeding the cut-off value with one unit
- ' $\leq$ x' or ' $\geq$ x': imputation by x.

This also applies to normal limits expressed as such.

No such imputations will be done for urinalysis parameters as these are usually character/categorical expressions

#### 6.2.2. Analysis Methods

Laboratory data will be summarized by type of laboratory test. Actual values and changes from baseline will be summarized by treatment group at each scheduled time point.

A cross-tabulation of the worst toxicity/abnormality versus baseline will be presented per phase (treatment phase, follow-up phase) and for the combination of treatment and follow-up phase. This table will also show the number and percentage of subjects per worst toxicity/abnormality, the number and percentage of subjects per emergent worst toxicity/abnormality and the cumulative number of subjects per emergent toxicity/abnormality or worse.

Mean  $\pm$  SE graphs over time for the actual values and changes from baseline will be generated for all tests performed by treatment group.

A listing of abnormal individual subject hematology and clinical chemistry values from scheduled and unscheduled time points will be provided. This listing will include all other time points for the corresponding subject/parameter. Grade 2 or higher toxicity laboratory values will be listed separately. Urinalysis results will be listed.

## 6.3. Vital Signs and Physical Examination Findings

Systolic and Diastolic blood pressure, heart rate, respiratory rate, body temperature and oxygen saturation (SpO<sub>2</sub>) will be investigated.

#### 6.3.1. Definitions

The vital signs abnormalities will be defined as indicated in Table 12. In determining the abnormalities, the following rules are applied:

- Worst grades/abnormalities are determined over the whole observational period for each trial phase separately, including post-baseline scheduled and unscheduled measurements of that phase.
- The abnormalities 'abnormally low' and 'abnormally high'/grades are considered equally important, i.e. if a subject has as well an abnormally low as an abnormally high or graded value post-baseline, both abnormalities are shown in the tables. (This means that the sum of the percentages can be more than 100%).

**Table 12:** Clinically Important Abnormalities in Vital Signs

| Vital Sign | Abnormality Code | Criteria |
|---|---|---|
| Systolic blood | Abnormally low | ≤ 90 mmHg |
| pressure | - | |
| | Grade 1 or mild | > 140 mmHg - < 160 mmHg |
| | Grade 2 or moderate | ≥ 160 mmHg - < 180 mmHg |
| | Grade 3 or severe | ≥ 180 mmHg |
| Diastolic blood pressure | Abnormally low | ≤ 50 mmHg |
| | Grade 1 or mild | > 90 mmHg - < 100 mmHg |
| | Grade 2 or moderate | ≥ 100 mmHg - < 110 mmHg |
| | Grade 3 or severe | ≥ 110 mmHg |
| Respiratory rate | Grade 1 or mild | 17-20 breaths per minute |
| | Grade 2 or moderate | 21-25 breaths per minute |
| | Grade 3 or severe | > 25 breaths per minute |
| | Grade 4 or potentially life threatening | Intubation |
| Oxygen Saturation | Abnormally low | < 95% |
| Temperature (oral) | Abnormally high | > 38.0 ° C |
| Pulse/Heart Rate | Abnormally low | ≤ 45 bpm |
| | Abnormally high | ≥ 120 bpm |

# **Emergent definition for abnormalities**

An abnormality will be considered emergent if it is worse than baseline. If baseline is missing, the abnormality is always considered emergent. A shift from 'abnormally low' at baseline to 'abnormally high' post baseline (or vice versa) is also emergent.

# 6.3.2. Analysis Methods

Actual values and changes from baseline will be summarized by treatment group at each scheduled time point.

A cross-tabulation of the worst toxicity/abnormality versus baseline will be presented per phase (treatment phase, follow-up phase) and for the combination of treatment and follow-up phase. This table will also show the number and percentage of subjects per worst toxicity/abnormality, the number and percentage of subjects per emergent worst toxicity/abnormality and the cumulative number of subjects per emergent toxicity/abnormality or worse.

Mean  $\pm$  SE graphs over time for the actual values and changes from baseline will be generated for all tests performed by treatment group.

A listing of abnormal (or grade 2 or higher) individual subject vital signs values will be provided. This listing will include all other time points for the corresponding subject/parameter.

# 6.4. Electrocardiogram

PR, QT, QRS, QTc intervals and heart rate will be investigated. QTcB and QTcF values will be used as reported by the central ECG provider, they will not be recalculated.

#### 6.4.1. Definitions

The ECG abnormalities will be defined as indicated in Table 13. In determining the abnormalities, the following rules are applied:

- Worst grades/abnormalities are determined over the whole observational period and for each trial phase separately, including post-baseline scheduled and unscheduled measurements of that phase.
- The abnormalities 'abnormally low' and 'abnormally high'/grades are considered equally important, i.e. if a subject has as well an abnormally low as an abnormally high or graded value post-baseline, both abnormalities are shown in the tables. (This means that the sum of the percentages can be more than 100%).

**Table 13:** ECG Abnormalities

| ECG parameter | Abnormality Code | Criteria |
|---|---|---|
| Abnormalities on actual values | | |
| Pulse/Heart Rate | Abnormally low | ≤ 45 bpm |
| | Abnormally high | ≥ 120 bpm |
| PR | Abnormally high | ≥ 210 ms |
| QRS | Abnormally high | ≥ 120 ms |
| QT <sub>corrected</sub> | Borderline prolonged QT | 450 ms < QTc ≤ 480 ms |
| | Prolonged QT | $480 \text{ ms} < \text{QTc} \le 500 \text{ ms}$ |
| | Pathologically prolonged QT | QTc > 500 ms |
| Abnormalities on | changes from baseline ( $\Delta QTc$ ) | |
| QT <sub>corrected</sub> | Normal QTc change | $\Delta QTc < 30 \text{ ms}$ |
| | Borderline QTc change | $30 \text{ ms} \le \Delta QTc \le 60 \text{ ms}$ |
| | Abnormally high QTc change | $\Delta QTc > 60 \text{ ms}$ |

#### **Emergent definition for abnormalities**

An abnormality will be considered emergent if it is worse than baseline. If baseline is missing, the abnormality is always considered as emergent. A shift from 'abnormally low' at baseline to 'abnormally high' or 'grade ...' post baseline (or vice versa) is also emergent.

# **Triplicate ECG assessments**

For time points on which triplicate ECGs apply (expected for all time points), a mean value per triplet cluster, will be calculated per time point before any further handling. This mean value will be used through the entire analysis. In the analysis dataset, the time of the first triplet member will be retained for this average record.

## **Rounding**

When ECG parameters need to be derived or any operations should be performed (e.g. averaging over many assessments/triplicates), no rounding to the integer/unit will be performed; the maximum stored resolution of these vales in the derived dataset(s) will be limited to 8 decimal positions. When used in tables, these values will be presented using formats reflecting the resolution of the unit applicable to the respective parameter (milliseconds, beats per minute).

# 6.4.2. Analysis Methods

Actual values and changes from baseline will be summarized by treatment group at each scheduled time point.

A cross-tabulation of the worst toxicity/abnormality versus baseline will be presented per phase (treatment phase, follow-up phase) and for the combination of treatment and follow-up phase. This table will also show the number and percentage of subjects per worst toxicity/abnormality, the number and percentage of subjects per emergent worst toxicity/abnormality.

A tabulation of the worst QT/QTc change versus baseline per treatment per phase (treatment phase, follow-up phase) and for the combination of treatment and follow-up phase will be presented

Mean  $\pm$  SE graphs over time for the actual values and changes from baseline will be generated for all tests performed by treatment group.

A listing of abnormal individual subject ECG values will be provided. This listing will include all other time points for the corresponding subject/parameter.

#### 7. HEALTH ECONOMICS

#### 7.1. Definitions

Medical Resource Utilization will be assessed by the number and duration of medical care encounters for RSV infection or complications associated with RSV per investigator assessment.

Information will be provided as:

- Number of medical encounters and rationale (AE, Other)
- Type of encounter such as medical practitioner office, emergency room, hospitalization, intensive care unit, palliative care unit among others
- Specialist involved
- Frequency of visits.

#### 7.2. Analysis Methods

The proportion of subjects requiring any medical encounter will be shown in a frequency tabulation by treatment group with the corresponding 90% confidence interval (exact Clopper-Pearson method).

Similar frequency tables will be provided for type of medical encounter. Data will also be summarized stratifying by presence of any comorbidity.

Additional information on medical encounters (frequency of visits, type of practitioner) will be listed.

#### 8. VIROLOGY

The sequencing results of the F-gene (and other regions of the RSV genome at the request of the protocol virologist) and changes from baseline will be summarized. Sequencing results may be presented in a separate report.

#### 8.1. Definitions

## **Viral Strain Typing**

The RSV subtype is determined at baseline using the RSV-A/B RT-qPCR assay performed in the central lab.

## **Viral Sequencing**

Viral resistance will be evaluated by next-generation sequencing (NGS) of the RSV Fusion (F) gene using a read frequency cut-off that will be defined in the Data Presentation Sheet.

Baseline samples from all subjects will be sequenced to identify pre-existing polymorphisms in the F gene. Post-baseline sequencing will be performed on the last evaluable on-treatment sample and/or during follow-up for all subjects (if viral load is high enough) to identify emerging amino acid substitutions in the F gene. Additional post-baseline sequencing can be performed on request of the sponsor virologist.

#### **Genetic variations**

Genetic variations are defined as changes (on amino acid or nucleotide level) in the subject's virus's sequence compared to a reference sequence. Genetic variations can include substitutions, insertions and deletions. The reference sequences used will be RSV-A Long strain (GenBank Accession number AY911262) for RSV-A samples and RSV-B strain 9320 (GenBank Accession number AY353550) for RSV-B samples. Genetic variations will be reported on amino acid level.

- **Baseline polymorphism**: amino acid difference from the RSV-A or RSV-B reference strain detected at baseline above a certain NGS read frequency cut-off, which is to be defined.
- **Emerging genetic variation:** a genetic variation (amino acid substitution, insertion or deletion) that is absent (i.e. below a to be defined NGS read frequency cut-off) at baseline but present above a certain to be defined NGS read frequency cut-off at a later post-baseline time point.
- Enriched genetic variation: a genetic variation (amino acid substitution, insertion or deletion) that is present at baseline with an NGS read frequency cut-off that will be defined and detected post-baseline with an increase in NGS read frequency compared to baseline.

The minimum increase in NGS read frequency to meet the definition of enriched genetic variation will be defined.

- **Genetic variation profile**: a specific genetic variation or combination of genetic variations at one or more time points.
- RSV F-gene amino acid positions of interest:
  - O Short list of 8 F-gene positions of interest for JNJ-53718678, based on in vitro selection experiments with JNJ-53718678 and/or in vitro reduced susceptibility to JNJ-53718678: positions 141, 143, 394, 398, 400, 486, 488, and 489.
  - Long list of 20 F-gene positions of interest for the class of RSV fusion inhibitors, based on in vitro selection experiments, clinical observations, and/or in vitro reduced susceptibility to RSV fusion inhibitors: positions 127, 138, 140, 141, 143, 144, 323, 338, 392, 394, 398, 399, 400, 401, 474, 486, 487, 488, 489, and 517.

The read frequency cut-off that will be used for reporting RSV F-gene NGS data, as well as the read frequency cut-offs used in the definitions of baseline polymorphisms, emerging and enriched genetic variations will be defined in the Data Presentation Specifications.

# **Analysis Time Points**

Virology results will be assigned to the visit windows as described in Sections 2.1.2 Phase Definitions and 2.1.4 Visit Windows. In addition to the time points corresponding to the visits at which samples for RSV F gene sequencing are collected, the below time points will be considered:

- Baseline (BL): Time point with sequencing data available closest prior to the first dose. This will be the Day 1 pre-treatment sample; however, if RSV F gene sequencing data cannot be obtained from this sample, the screening sample may be used for sequencing.
- Last Evaluable On-Treatment Time Point: Last available post-baseline time point during the treatment phase with sequencing data available. In case no On-Treatment assessment is available, the first assessment during Follow-Up is selected instead.
- Time Point of Sequence during the Follow-Up phase: Last available post-baseline time point during the follow-up phase with sequencing data available.
- Entire post-baseline phase: Aggregate of all available post-baseline time points in the study with sequencing data available

# 8.2. Analysis Methods

# 8.2.1. Viral Strain Typing

The number of subjects by RSV subtype will be tabulated in frequency outputs (n, %).

#### 8.2.2. Viral Sequencing

#### **Baseline**

The prevalence of baseline polymorphisms in the RSV F-gene, ie the number of subjects with baseline polymorphisms in the RSV F-gene, will be tabulated in frequency outputs (n, %).

Amino acid changes from reference sequence at baseline will be listed for all subjects using a defined NGS read frequency cut-off (will be defined in the Data Presentation Specifications).

# **Post-baseline**

Emerging and enriched genetic variations will be tabulated by analysis time point in frequency outputs (n, %). Amino acid changes from reference sequence will be listed for all subjects with post-baseline sequencing data using a defined NGS read frequency cut-off (will be defined in the Data Presentation Specifications).

## **REFERENCES**

- Duncan CB, Walsh EE et al. Risk Factors for Respiratory Failure Associated with Respiratory Syncytial Virus Infection in Adults. *J Infect Dis*. 2009 October 15; 200(8): 1242–1246.
- Walsh EE, Peterson DR et al. Risk Factors for Severe Respiratory Syncytial Virus Infection in Elderly Persons. *J Infect Dis*. 2004; 189:233–8
- EQ-5D-5L User Guide. Basic information on how to use the EQ-5D-5L instrument, Version 2.1, April 2015, Mandy van Reenen / Bas Janssen, EuroQol Research Foundation, www.euroqol.org
- E.D. Bacci, K. Kim, S. Stringer, N. K. Leidy, User Manual for the InFLUenza Patient-Reported Outcome (FLU-PRO) Diary, Version 1.1
- Akaike H., A new look at the statistical model identification, IEEE Transactions on Automatic Control, 1974: 19 (6): 716–723.
- Kaplan E. L., Meier P. Nonparametric estimation from incomplete observations. Journal of the American Statistical Association, 1958; 53 (282): 457–481.
- Mehta CR. and Patel NR, Exact Logistic Regression: Theory and Examples, Statistics in Medicine, 1995: 14, 2143–2160.

#### **ATTACHMENTS**

Attachment [1]: Division of Microbiology and Infectious Diseases (DMID) Adult Toxicity Table – November 2007

**ABBREVIATIONS**: Abbreviations utilized in the Table:

ULN = Upper Limit of Normal LLN = Lower Limit of Normal

 $R_x$  = Therapy Req = Required Mod = Moderate IV = Intravenous ADL = Activities of Daily Living Dec = Decreased

#### **ESTIMATING SEVERITY GRADE**

For abnormalities NOT found elsewhere in the Toxicity Tables use the scale below to estimate grade of severity:

- **GRADE 1** Mild Transient or mild discomfort (< 48 hours); no medical intervention/therapy required
- **GRADE 2 Moderate** Mild to moderate limitation in activity some assistance may be needed; no or minimal medical intervention/therapy required
- **GRADE 3 Severe** Marked limitation in activity, some assistance usually required; medical intervention/therapy required, hospitalizations possible
- **GRADE 4 Life-threatening** Extreme limitation in activity, significant assistance required; significant medical intervention/therapy required, hospitalization or hospice care probable

#### **SERIOUS OR LIFE-THREATENING AES**

ANY clinical event deemed by the clinician to be serious or life-threatening should be considered a grade 4 event. Clinical events considered to be serious or life-threatening include, but are not limited to: seizures, coma, tetany, diabetic ketoacidosis, disseminated intravascular coagulation, diffuse petechiae, paralysis, acute psychosis, severe depression.

#### **COMMENTS REGARDING THE USE OF THESE TABLES**

- Standardized and commonly used toxicity tables (Division of AIDS, NCI's Common Toxicity Criteria (CTC), and World Health Organization [WHO]) have been adapted for use by the Division of Microbiology and Infectious Diseases (DMID) and modified to better meet the needs of participants in DMID trials.
- For parameters not included in the following Toxicity Tables, sites should refer to the "Guide For Estimating Severity Grade" located above.
- Criteria are generally grouped by body system.
- Some protocols may have additional protocol-specific grading criteria, which will supersede the use of these tables for specified criteria.

| HEMATOLOGY | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Hemoglobin | 9.5 - 10.5 gm/dL | 8.0 - 9.4gm/dL | 6.5 - 7.9 gm/dL | < 6.5 gm/dL |
| Absolute Neutrophil Count | 1,000-1,500/ mm <sup>3</sup> | 750-999/ mm <sup>3</sup> | 500-749/ mm <sup>3</sup> | <500/ mm <sup>3</sup> |
| Platelets | 75,000-<br>99,999/ mm <sup>3</sup> | 50,000-<br>74,999/ mm <sup>3</sup> | 20,000-49,999/ mm <sup>3</sup> | <20,000/ mm <sup>3</sup> |
| WBCs | 11,000-13,000/<br>mm <sup>3</sup> | 13,000-<br>15,000 / mm <sup>3</sup> | 15,000-<br>30,000/ mm <sup>3</sup> | >30,000 or<br><1,000 / mm <sup>3</sup> |
| % Polymorphonuclear<br>Leucocytes + Band Cells | > 80% | 90 – 95% | >95% | |
| Abnormal Fibrinogen | Low:<br>100-200 mg/dL<br>High:<br>400-600 mg/dL | Low:<br><100 mg/dL<br>High:<br>>600 mg/dL | Low:<br>< 50 mg/dL | Fibrinogen<br>associated with gross<br>bleeding or with<br>disseminated<br>coagulation |
| Fibrin Split Product | 20-40 mcg/ mL | 41-50 mcg/ mL | 51-60 mcg/ mL | > 60 mcg/ mL |
| Prothrombin Time (PT) | 1.01 - 1.25 x ULN | 1.26-1.5 x ULN | 1.51 -3.0 x ULN | >3 x ULN |
| Activated Partial<br>Thromboplastin (APPT) | 1.01 -1.66 x ULN | 1.67 - 2.33 x ULN | 2.34 - 3 x ULN | > 3 x ULN |
| Methemoglobin | 5.0 - 9.9 % | 10.0 - 14.9 % | 15.0 - 19.9% | > 20.0 % |

| CHEMISTRIES | 3 | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Hyponatremia | 130-135 mEq/ L | 123-129 mEq/ L | 116-122 mEq/ L | < 116 mEq/ L or abnormal sodium<br>with mental<br>status changes or seizures |
| Hypernatremia | 146-150 mEq/ L | 151-157 mEq/ L | 158-165 mEq/ L | > 165 mEq/ L or abnormal sodium<br>with mental<br>status changes or seizures |
| Hypokalemia | 3.0 - 3.4 mEq/ L | 2.5 - 2.9 mEq/ L | 2.0 - 2.4 mEq/ L or<br>intensive replacement<br>therapy or<br>hospitalization<br>required | < 2.0 mEq/ L or abnormal<br>potassium with<br>paresis, ileus or life-threatening<br>arrhythmia |
| Hyperkalemia | 5.6 - 6.0 mEq/ L | 6.1 - 6.5 mEq/ L | 6.6 - 7.0 mEq/l | > 7.0 mEq/ L or abnormal potassium <i>with</i> life-threatening arrhythmia |
| Hypoglycemia | 55-64 mg/dL | 40-54 mg/dL | 30-39 mg/dL | <30 mg/dL or abnormal glucose<br>with mental<br>status changes or coma |
| Hyperglycemia (nonfasting and no prior diabetes) | 116 - 160 mg/dL | 161- 250 mg/d L | 251 - 500 mg/dL | > 500 mg/dL or abnormal glucose with ketoacidosis or seizures |
| Hypocalcemia<br>(corrected for<br>albumin) | 8.4 - 7.8 mg/dL | 7.7 - 7.0 mg/dL | 6.9 - 6.1 mg/dL | < 6.1 mg/dL or abnormal calcium with life-threatening arrhythmia or tetany |

| CHEMISTRIES (continued) | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Hypercalcemia (correct for albumin) | 10.6 - 11.5 mg/dL | 11.6 - 12.5<br>mg/d L | 12.6 - 13.5 mg/dL | > 13.5 mg/dL or abnormal calcium <i>with</i> life-threatening arrhythmia |
| Hypomagnesemia | 1.4 - 1.2 mEq/ L | 1.1 - 0.9 mEq/ L | 0.8 - 0.6 mEq/ L | < 0.6 mEq/ L or abnormal<br>magnesium <i>with</i> life-<br>threatening arrhythmia |
| Hypophosphatemia | 2.0 - 2.4 mg/dL | 1.5 -1.9 mg/dL or<br>replacement Rx<br>required | 1.0 -1.4 mg/dL<br>intensive therapy or<br>hospitalization<br>required | < 1.0 mg/dL or abnormal<br>phosphate <i>with</i> life-<br>threatening arrhythmia |
| Hyperbilirubinemia (when accompanied by any increase in other liver function test) | 1.1 - <1.25 x ULN | 1.25 - <1.5 x<br>ULN | 1.5 – 1.75 x ULN | > 1.75 x ULN |
| Hyperbilirubinemia (when other liver function are in the normal range) | 1.1 - <1.5 x ULN | 1.5 - <2.0 x ULN | 2.0 – 3.0 x ULN | > 3.0 x ULN |
| BUN | 1.25 - 2.5 x ULN | 2.6 - 5 x ULN | 5.1 - 10 x ULN | > 10 x ULN |
| Hyperuricemia (uric acid) | 7.5 – 10.0 mg/dL | 10.1 – 12.0<br>mg/dL | 12.1 – 15.0 mg/d L | >15.0 mg/d L |
| Creatinine | 1.1 - 1.5 x ULN | 1.6 - 3.0 x ULN | 3.1 - 6 x ULN | >6 x ULN or dialysis required |

| ENZYMES | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| AST (SGOT) | 1.1 - <2.0 x ULN | 2.0 – <3.0 x ULN | 3.0 – 8.0 x ULN | > 8 x ULN |
| ALT (SGPT) | 1.1 - <2.0 x ULN | 2.0 – <3.0 x ULN | 3.0 – 8.0 x ULN | > 8 x ULN |
| GGT | 1.1 - <2.0 x ULN | 2.0 – <3.0 x ULN | 3.0 – 8.0 x ULN | > 8 x ULN |
| Alkaline Phosphatase | 1.1 - <2.0 x ULN | 2.0 – <3.0 x ULN | 3.0 – 8.0 x ULN | > 8 x ULN |
| Amylase | 1.1 - 1.5 x ULN | 1.6 - 2.0 x ULN | 2.1 - 5.0 x ULN | > 5.1 x ULN |
| Lipase | 1.1 - 1.5 x ULN | 1.6 - 2.0 x ULN | 2.1 - 5.0 x ULN | > 5.1 x ULN |

| URINALYSIS | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Proteinuria | 1+ | 2-3+ | 4+ | nephrotic syndrome |
| | or<br>200 mg - 1 gm<br>loss/day | or<br>1-2 gm loss/day | or<br>2-3.5 gm loss/day | or<br>>3.5 gm loss/day |
| Hematuria | microscopic only<br><10 rbc/hpf | gross, no clots<br>>10 rbc/hpf | gross, with or without clots, OR RBC casts | obstructive or<br>required<br>transfusion |

| CARDIOVASCULAR | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Cardiac Rhythm | | asymptomatic,<br>transient signs, no<br>Rx required | recurrent/persistent;<br>symptomatic Rx<br>required | unstable dysrythmia;<br>hospitalization<br>and treatment<br>required |
| Hypertension | transient increase >20 mm/ Hg; no treatment | recurrent, chronic<br>increase<br>> 20mm/ Hg<br>/treatment required | acute treatment<br>required; outpatient<br>treatment or<br>hospitalization<br>possible | end organ damage or<br>hospitalization<br>required |
| Hypotension | transient orthostatic hypotension with heart rate increased by <20 beat/min or decreased by <10 mm Hg systolic BP, No treatment required | symptoms due to orthostatic hypotension or BP decreased by <20 mm Hg systolic; correctable with oral flu id treatment | hospitalization required | mean arterial pressure <60mm/ Hg or end organ damage or shock; requires hospitalization and vasopressor treatment |
| Pericarditis | minimal effusion | mild/ moderate<br>asymptomatic<br>effusion, no treatment | symptomatic<br>effusion; pain; EKG<br>changes | tamponade;<br>pericardiocentesis or<br>surgery required |
| Hemorrhage, Blood Loss | microscopic/occult | mild, no transfusion | gross blood loss;<br>1-2 units transfused | massive blood loss; >3 units transfused |

| RESPIRATORY | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Cough | transient- no<br>treatment | persistent cough;<br>treatment responsive | Paroxysmal cough;<br>uncontrolled with<br>treatment | |
| Bronchospasm, Acute | transient; no<br>treatment;<br>70% - 80% FEV1<br>of peak flow | requires<br>treatment; normalizes<br>with bronchodilator;<br>FEV1 50% -<br>70%<br>(of peak flow) | no normalization<br>with bronchodilator;<br>FEV1 25% - 50%<br>of peak flow; or<br>retractions present | cyanosis: FEV1<br><25%<br>of peak flow or<br>intubation necessary |
| Dyspnea | dyspnea on exertion | dyspnea with normal activity | dyspnea at rest | dyspnea requiring oxygen therapy |

| GASTROINTESTINAL | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Nausea | mild or transient;<br>maintains<br>reasonable intake | moderate discomfort;<br>intake decreased<br>significantly; some<br>activity limited | no significant intake;<br>requires IV flu ids | hospitalization<br>required; |
| Vomiting | 1 episode in 24 hours | 2-5 episodes in<br>24 hours | >6 episodes in<br>24 hours or needing<br>IV fluids | physiologic<br>consequences<br>requiring<br>hospitalization or<br>requiring parenteral<br>nutrition |
| Constipation | requiring stool<br>softener or dietary<br>modification | requiring<br>laxatives | obstipation<br>requiring manual<br>evacuation or enema | obstruction or toxic megacolon |
| Diarrhea | mild or transient; 3-4<br>loose<br>stools/day or mild<br>diarrhea last <1 week | stools/day or diarrhea | >7 loose stools/day<br>or bloody diarrhea; or<br>orthostatic<br>hypotension or<br>electrolyte imbalance<br>or >2L IV fluids<br>required | consequences requiring |
| Oral Discomfort/Dysphagia | mild discomfort; no<br>difficulty<br>swallowing | some limits on<br>eating/drinking | eating/talking very<br>limited; unable to<br>swallow solid foods | unable to drink flu<br>ids; requires IV fluids |

| NEUROLOGICAL | | | | | | |
|---|---|---|---|---|--|--|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 | | |
| Neuro-Cerebellar | slight incoordination<br>dysdiadochokinesis | intention tremor,<br>dysmetria,<br>slurred speech;<br>nystagmus | locomotor ataxia | incapacitated | | |
| Psychiatric | mild anxiety or<br>depression | moderate anxiety or<br>depression; therapy<br>required; change in<br>normal routine | severe mood changes<br>requiring therapy; or<br>suicidal ideation; or<br>aggressive ideation | acute psychosis requiring hospitalization; or suicidal gesture/attempt or hallucinations | | |
| Muscle Strength | subjective weakness<br>no objective<br>symptoms/ signs | mild objective<br>signs/symptoms no<br>decrease in function | objective weakness function limited | paralysis | | |
| Paresthesia (burning, tingling, etc.) | mild discomfort; no treatment required | moderate discomfort;<br>non-narcotic<br>analgesia required | severe discomfort; or<br>narcotic analgesia<br>required with<br>symptomatic<br>improvement | incapacitating; or not<br>responsive to narcotic<br>analgesia | | |
| Neuro-sensory | mild impairment in sensation (decreased sensation, eg, vibratory, pinprick, hot/cold in great toes) in focal area or symmetrical distribution; or change in taste, smell, vision and/or hearing | moderate impairment (mod decreased sensation, eg, vibratory, pinprick, hot/cold to ankles) and/or joint position or mild impairment that is not symmetrical | severe impairment (decreased or loss of sensation to knees or wrists) or loss of sensation of at least mod degree in multiple different body areas (ie, upper and lower extremities) | / | | |
| MUSCULOSKELATEL | | | | | | | |
|---|---|---|---|---|--|--|--|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 | | | |
| Arthralgia (joint pain) | mild pain not<br>interfering with<br>function | moderate pain,<br>analgesics and/or pain<br>interfering with<br>function but not with<br>activities of daily<br>living | severe pain; pain<br>and/or analgesics<br>interfering with<br>activities of daily<br>living | disabling pain | | | |
| Arthritis | mild pain with inflammation, erythema or joint swelling – but not interfering with function | moderate pain with inflammation, erythema or joint swelling – interfering with function, but not with activities of daily living | severe pain with<br>inflammation,<br>erythema or joint<br>swelling –and<br>interfering with<br>activities of daily<br>living | permanent and/or<br>disabling joint<br>destruction | | | |
| Myalgia | Myalgia with no limitation of activity | muscle<br>tenderness (at other<br>than injection site) or<br>with moderate<br>impairment of activity | activity | frank<br>myonecrosis | | | |

| SKIN | SKIN | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Mucocutaneous | erythema; pruritus | diffuse,<br>maculopapular rash,<br>dry desquamation | vesiculation or<br>moist desquamation<br>or ulceration | exfoliative dermatitis, mucous membrane involvement or erythema, multiforme or suspected Stevens-Johnson or necrosis requiring surgery |
| Induration | <15mm | 15-30 mm | >30mm | |
| Erythema | <15mm | 15-30 mm | >30mm | |
| Edema | <15mm | 15-30 mm | >30mm | |
| Rash at Injection Site | <15mm | 15-30 mm | >30mm | |
| Pruritus | slight itching at injection site | moderate itching at injection extremity | itching over entire body | |

| SYSTEMIC | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Allergic Reaction | pruritus without rash | localized urticaria | generalized urticaria;<br>angioedema | anaphylaxis |
| Headache | mild, no treatment required | transient, moderate;<br>treatment required | severe; responds to<br>initial narcotic<br>therapy | intractable; requires<br>repeated narcotic<br>therapy |
| Fever: oral | 37.7 - 38.5 C or<br>100.0 - 101.5 F | 38.6 - 39.5 C or<br>101.6 - 102.9 F | 39.6 - 40.5 C or 103 -<br>105 F | >40 C or<br>>105 F |
| Fatigue | normal activity<br>reduced < 48 hours | normal activity<br>decreased 25-<br>50% > 48 hours | normal activity<br>decreased > 50%<br>can't work | unable to care for self |

## Attachment [2]: Inclusion/exclusion criteria

#### Inclusion Criteria

Each potential subject must satisfy all of the following criteria to be enrolled in the study:

- 1. Male or female.
- 2.  $\geq 18$  years of age.
- 3. Must sign an ICF indicating they understand the purpose of, and procedures required for, the study and is willing to participate in the study.

**Note**: Prior to signing the main consent form for the study, subjects may specifically allow for the collection and testing of nasal mid-turbinate swabs by signing the pre-screening (diagnostic) ICF.

4. Subjects must have an acute respiratory illness with signs and symptoms consistent with a viral infection (eg, fever, cough, nasal congestion, runny nose, sore throat, myalgia, lethargy, shortness of breath, or wheezing) with onset ≤5 days from the anticipated time of randomization. Onset of symptoms is defined as the time the subject becomes aware of the first sign and/or symptom consistent with a viral infection. Efforts should be made to determine the time of onset of symptoms as accurately as possible (in relation to routine daily activities).

**Note**: The viral infection may present in any way as long as the underlying precipitant of the illness is considered by the investigator to be due to RSV infection. Examples of such an illness include:

- An upper or lower viral respiratory tract infection (eg, "flu-like illness");
- Pneumonia;
- Respiratory distress;
- Asthma exacerbation;
- COPD exacerbation.
- 5. Subject has been diagnosed with RSV infection using a rapid PCR-based (preferably locally available) or rapid-antigen-detection test.

*Note*: If a patient has a positive similar diagnostic test from another study and meets all eligibility criteria for inclusion in this study, this diagnostic test result can be used for confirmation of eligibility.

- 6. Before randomization, a woman must be not of childbearing potential defined as:
  - Premenarchal
     A premenarchal state is one in which menarche has not yet occurred.

- Postmenopausal
  - A postmenopausal state is defined as no menses for 12 months without an alternative medical cause. An available high follicle-stimulating hormone level (>40 IU/L or mIU/mL) in the postmenopausal range may be used to confirm a postmenopausal state in women not using hormonal contraception or hormonal replacement therapy, however in the absence of 12 months of amenorrhea, a single follicle-stimulating hormone measurement is insufficient.
- Permanently sterile
   Permanent sterilization methods include hysterectomy, bilateral salpingectomy, bilateral tubal occlusion/ligation procedures, and bilateral oophorectomy.
- 7. A woman must agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction during the study and for a period of 30 days after the last dose of study drug.
- 8. All women must have a negative urine  $\beta$ -human chorionic gonadotropin pregnancy test at screening.
- 9. A male subject must wear a condom when engaging in any activity that allows for passage of ejaculate to another person. Male subjects should also be advised of the benefit for a female partner to use a highly effective method of contraception as a condom may break or leak.

*Note*: Contraceptive (birth control) use by subjects should be consistent with local regulations regarding the acceptable methods of contraception for those participating in clinical studies.

- 10. A male subject must agree not to donate sperm for the purpose of reproduction during the study and for a minimum of 90 days after receiving the last dose of study drug.
- 11. Willing and able to adhere to the lifestyle restrictions specified in this protocol (please see protocol Section 4.3).
- 12. With the exception of the RSV-related illness the subject must be medically stable on the basis of physical examination, medical history, vital signs, and ECG performed at screening. If there are abnormalities, they must be consistent with the underlying condition (RSV disease and/or comorbid condition) in the study population as evaluated by the investigator (with exception of QTcF interval >500 ms, see exclusion criterion 13). This determination must be recorded in the subject's source documents and initialed by the investigator.

### **Exclusion Criteria**

Any potential subject who meets any of the following criteria will be excluded from participating in the study:

- 1. Hospitalized subjects or subjects expected to be hospitalized within 24 hours of screening.
  - *Note*: Any stay in the emergency room or in the observational unit of at least 24 hours will be considered hospitalization for the purposes of the study.
- 2. History of or concurrent illness (beyond a comorbid condition) that in the opinion of the investigator, might confound the results of the study or pose an additional risk in administering study drug to the subject or that could prevent, limit, or confound the protocol-specified assessments.
- 3. Subjects who had major surgery within the 28 days prior to randomization or have planned major surgery through the course of the study.
- 4. Subjects who are considered by the investigator to be immunocompromised within the past 12 months, whether due to underlying medical condition (eg, malignancy or genetic disorder other than immunoglobulin A deficiency, or human immunodeficiency virus [HIV] infection) or medical therapy (eg, medications other than corticosteroids for the treatment of COPD or asthma exacerbations, chemotherapy, radiation, stem cell or solid organ transplant).
- 5. Subject has known or suspected chronic or acute hepatitis B or C infection.
- 6. Subject has known allergies, hypersensitivity, or intolerance to JNJ-53718678 or to any of the excipients of the JNJ-53718678 or placebo formulation (refer to the IB).
- 7. Subject with current or planned participation in another clinical study where study drug/investigational device is being administered while participating in the current study.
- 8. Subjects unwilling to undergo mid-turbinate nasal swab procedures or with any physical abnormality which limits the ability to collect regular nasal specimens.
- 9. Subjects unable to take medications orally or with a known gastrointestinal-related condition that is considered by the sponsor or investigator to be likely to interfere with study drug ingestion or absorption.
- 10. Women who are pregnant or breastfeeding.

- 11. Men who plan to father a child while enrolled in this study or within 90 days after the last dose of study drug.
- 12. Subject with clinically significant abnormal ECG findings (other than QTcF interval >500 ms, see exclusion criterion 13) not consistent with the underlying condition in the study population, as judged by the investigator.
- 13. Confirmed QTcF interval >500 ms per the machine read parameter result at screening. Confirmation needs to be obtained by repeat triplicate ECG recording prior to dosing.
- 14. Subjects who are using any disallowed medication as listed in Section 8 of the protocol.
- 15. Subjects with history of drug or alcohol abuse according to Diagnostic and Statistical Manual of Mental Disorders (5<sup>th</sup> edition) criteria within 1 year before screening.
- 16. Subjects who received an investigational drug, an investigational vaccine, or used an invasive investigational medical device within 30 days or 5 elimination half-lives (whichever is longer) before the planned first dose of study drug or is currently enrolled in an investigational study.
- 17. Subject is a family member of the employees of the investigator or study-site with direct involvement in the proposed study or other studies under the direction of that investigator or study-site or of the investigator.

78

# Attachment [3]:

# Respiratory infection-patient reported outcomes (ri-pro $\ensuremath{\mathbb{G}}$ ) symptom questionnaire

| Domain | Items | Scoring and Minimum Data Requirement |
|---|---|---|
| Nose | Runny or dripping nose | Arithmetic mean of 4 items |
| | Congested or stuffy nose | Daily score for 3 of 4 items |
| | Sneezing | must be present to calculate domain score |
| | Sinus pressure | domain score |
| Throat | Scratchy or itchy throat | Arithmetic mean of 3 items |
| | Sore or painful throat | Daily score for 2 of 3 items |
| | Difficulty swallowing | must be present to calculate domain score |
| Eyes | Teary or watery eyes | Arithmetic mean of 3 items |
| | Sore or painful eyes | Daily score for 2 of 3 items |
| | Eyes sensitive to light | must be present to calculate domain score |
| Chest/Respiratory | Trouble breathing | Arithmetic mean of 7 items |
| | Chest congestion | Daily score for 5 of 7 items |
| | Chest tightness | must be present to calculat domain score |
| | Dry or hacking cough | WOMANI DOOLO |
| | Wet or loose cough | |
| | Coughing | |
| | Coughed up mucus or phlegm | |
| Gastrointestinal | Felt nauseous | Arithmetic mean of 4 items |
| | Stomach ache | Daily score for 3 of 4 items |
| | Vomit (frequency) | must be present to calculate domain score |
| | Diarrhea (frequency) | domain score |
| Body/Systemic | Felt dizzy | Arithmetic mean of 11 items |
| | Head congestion | Daily score for 8 of 11 items |
| | Headache | must be present to calculate domain score |
| | Lack of appetite | domain score |
| | Sleeping more than usual | |
| | Body aches or pains | |

| Domain | Items | Scoring and Minimum Data<br>Requirement |
|--------|---------------------|-----------------------------------------|
| | Weak or tired | |
| | Chills or shivering | |
| | Felt cold | |
| | Felt hot | |
| | Sweating | |

# Adult RSV additional questions

| Addit | ional Questions About Health and Functioning | |
|---|---|---|
| 1. | Did you take any medicine for our respiratory infection | Yes |
| | symptoms today? | No |
| 2. | Did you use any rescue medicine today for asthma or COPD? | I do not take medicine for asthma or COPD |
| | | Yes |
| | | No |
| 3. | Since this time yesterday, how much of the time did you | None of the time |
| | breathe oxygen from an oxygen tank? | Less than an hour |
| | | 1 to 4 hours |
| | | More than 4 hours |
| 4. | Overall, how severe were your respiratory infection symptoms today? | No respiratory infection symptoms today |
| | | Mild |
| | | Moderate |
| | | Severe |
| | | Very Severe |
| 5. | Overall, how were your respiratory infection symptoms | Much better |
| | today compared to yesterday? | Somewhat better |
| | | A little better |
| | | About the same |
| | | A little worse |
| | | Somewhat worse |
| | | Much worse |
| 6. | How much did your respiratory infection symptoms | Not at all |
| | interfere with your usual activities? | A little bit |
| | | Somewhat |
| | | Quite a bit |
| | | Very Much |

| 7. Have you returned to your usual activities today? | Yes |
|--------------------------------------------------------|-----------|
| | No |
| 8. In general, how would you rate your physical health | Excellent |
| today? | Very good |
| | Good |
| | Fair |
| | Poor |
| 9. Have you returned to your usual health today? | Yes |
| | No |

# Respiratory Infection Intensity and Impact Questionnaire (RiiQ™)







# Attachment [4]: EQ-5D-5L

# **EQ-5D-5L Dimensions**

| Dimension | | sion Level | | Interpretation |
|---|---|---|---|---|
| 1 | Mobility | 1 | No problems | I have no problems walking |
| | | 2 | Slight problems | I have slight problems walking |
| | | 3 | Moderate problems | I have moderate problems walking |
| | | 4 | Severe problems | I have severe problems walking |
| | | 5 | Extreme problems | I am unable to walk |
| 2 | Self-care | 1 | No problems | I have no problems washing or dressing myself |
| | | 2 | Slight problems | I have slight problems washing or dressing myself |
| | | 3 | Moderate problems | I have moderate problems washing or dressing myself |
| | | 4 | Severe problems | I have severe problems washing or dressing myself |
| | | 5 | Extreme problems | I am unable to wash or dress myself |
| 3 | Usual activities | 1 | No problems | I have no problems doing my usual activities |
| | | 2 | Slight problems | I have slight problems doing my usual activities |
| | | 3 | Moderate problems | I have moderate problems doing my usual activities |
| | | 4 | Severe problems | I have severe problems doing my usual activities |
| | | 5 | Extreme problems | I am unable to do my usual activities |
| 4 | Pain/discomfort | 1 | No problems | I have no pain or discomfort |
| | | 2 | Slight problems | I have slight pain or discomfort |
| | | 3 | Moderate problems | I have moderate pain or discomfort |
| | | 4 | Severe problems | I have severe pain or discomfort |
| | | 5 | Extreme problems | I have extreme pain or discomfort |
| 5 | Anxiety/depression | 1 | No problems | I am not anxious or depressed |
| | | 2 | Slight problems | I am slightly anxious or depressed |
| | | 3 | Moderate problems | I am moderately anxious or depressed |
| | | 4 | Severe problems | I am severely anxious or depressed |
| | | 5 | Extreme problems | I am extremely anxious or depressed |

The best health you can imagine

## **EQ-5D-5L VAS**

- We would like to know how good or bad your health is TODAY.
- This scale is numbered from 0 to 100.
- 100 means the <u>best</u> health you can imagine.
   0 means the <u>worst</u> health you can imagine.
- Mark an X on the scale to indicate how your health is TODAY.
- Now, please write the number you marked on the scale in the box below.

YOUR HEALTH TODAY =

 $\textit{USA (English)} © 2009 \; \textit{EuroQol Group. EQ-5D}{}^{\text{TM}} \textit{is a trade mark of the EuroQol Group}$ 

## **Valuation Index**

| Health state | Index Value | Health state | Index Value | Health state | Index Value | Health state | Index Value |
|---|---|---|---|---|---|---|---|
| 11111 | 1 | 11242 | 0,498 | 11423 | 0,606 | 11554 | 0,018 |
| 11112 | 0,879 | 11243 | 0,484 | 11424 | 0,437 | 11555 | -0,066 |
| 11113 | 0,848 | 11244 | 0,323 | 11425 | 0,26 | 12111 | 0,846 |
| 11114 | 0,635 | 11245 | 0,157 | 11431 | 0,653 | 12112 | 0,779 |
| 11115 | 0,414 | 11251 | 0,235 | 11432 | 0,596 | 12113 | 0,761 |
| 11121 | 0,837 | 11252 | 0,179 | 11433 | 0,582 | 12114 | 0,548 |
| 11122 | 0,768 | 11253 | 0,164 | 11434 | 0,412 | 12115 | 0,327 |
| 11123 | 0,75 | 11254 | 0,083 | 11435 | 0,236 | 12121 | 0,737 |
| 11124 | 0,537 | 11255 | -0,001 | 11441 | 0,475 | 12122 | 0,678 |
| 11125 | 0,316 | 11311 | 0,883 | 11442 | 0,419 | 12123 | 0,663 |
| 11131 | 0,796 | 11312 | 0,827 | 11443 | 0,404 | 12124 | 0,45 |
| 11132 | 0,74 | 11313 | 0,812 | 11444 | 0,27 | 12125 | 0,229 |
| 11133 | 0,725 | 11314 | 0,599 | 11445 | 0,131 | 12131 | 0,709 |
| 11134 | 0,512 | 11315 | 0,378 | 11451 | 0,209 | 12132 | 0,653 |
| 11135 | 0,291 | 11321 | 0,785 | 11452 | 0,153 | 12133 | 0,638 |
| 11141 | 0,584 | 11322 | 0,728 | 11453 | 0,138 | 12134 | 0,425 |
| 11142 | 0,527 | 11323 | 0,714 | 11454 | 0,057 | 12135 | 0,204 |
| 11143 | 0,513 | 11324 | 0,501 | 11455 | -0,027 | 12141 | 0,497 |
| 11144 | 0,352 | 11325 | 0,28 | 11511 | 0,556 | 12142 | 0,441 |
| 11145 | 0,186 | 11331 | 0,76 | 11512 | 0,5 | 12143 | 0,426 |
| 11151 | 0,264 | 11332 | 0,704 | 11513 | 0,485 | 12144 | 0,266 |
| 11152 | 0,208 | 11333 | 0,689 | 11514 | 0,404 | 12145 | 0,099 |
| 11153 | 0,193 | 11334 | 0,476 | 11515 | 0,32 | 12151 | 0,177 |
| 11154 | 0,112 | 11335 | 0,255 | 11521 | 0,458 | 12152 | 0,121 |
| 11155 | 0,028 | 11341 | 0,548 | 11522 | 0,401 | 12153 | 0,106 |
| 11211 | 0,906 | 11342 | 0,491 | 11523 | 0,387 | 12154 | 0,025 |
| 11212 | 0,837 | 11343 | 0,477 | 11524 | 0,306 | 12155 | -0,059 |
| 11213 | 0,819 | 11344 | 0,316 | 11525 | 0,222 | 12211 | 0,806 |
| 11214 | 0,606 | 11345 | 0,15 | 11531 | 0,433 | 12212 | 0,748 |
| 11215 | 0,385 | 11351 | 0,228 | 11532 | 0,377 | 12213 | 0,733 |
| 11221 | 0,795 | 11352 | 0,172 | 11533 | 0,362 | 12214 | 0,52 |
| 11222 | 0,736 | 11353 | 0,157 | 11534 | 0,281 | 12215 | 0,299 |
| 11223 | 0,721 | 11354 | 0,076 | 11535 | 0,197 | 12221 | 0,706 |
| 11224 | 0,508 | 11355 | -0,008 | 11541 | 0,328 | 12222 | 0,649 |
| 11225 | 0,287 | 11411 | 0,776 | 11542 | 0,272 | 12223 | 0,634 |
| 11231 | 0,767 | 11412 | 0,719 | 11543 | 0,257 | 12224 | 0,421 |
| 11232 | 0,711 | 11413 | 0,705 | 11544 | 0,176 | 12225 | 0,2 |
| 11233 | 0,696 | 11414 | 0,535 | 11545 | 0,092 | 12231 | 0,681 |
| 11234 | 0,483 | 11415 | 0,359 | 11551 | 0,17 | 12232 | 0,624 |
| 11235 | 0,262 | 11421 | 0,677 | 11552 | 0,114 | 12233 | 0,61 |
| 11241 | 0,555 | 11422 | 0,621 | 11553 | 0,099 | 12234 | 0,397 |
| 12235 | 0,176 | 12424 | 0,35 | 13113 | 0,744 | 13252 | 0,075 |

| | | | | | | • | |
|---|---|---|---|---|---|---|---|
| Health state | Index Value | Health state | Index Value | Health state | Index Value | Health state | Index Value |
| 12241 | 0,468 | 12425 | 0,174 | 13114 | 0,531 | 13253 | 0,06 |
| 12242 | 0,412 | 12431 | 0,566 | 13115 | 0,31 | 13254 | -0,021 |
| 12243 | 0,397 | 12432 | 0,51 | 13121 | 0,717 | 13255 | -0,105 |
| 12244 | 0,237 | 12433 | 0,495 | 13122 | 0,66 | 13311 | 0,779 |
| 12245 | 0,071 | 12434 | 0,325 | 13123 | 0,646 | 13312 | 0,723 |
| 12251 | 0,149 | 12435 | 0,149 | 13124 | 0,433 | 13313 | 0,708 |
| 12252 | 0,092 | 12441 | 0,389 | 13125 | 0,212 | 13314 | 0,495 |
| 12253 | 0,078 | 12442 | 0,332 | 13131 | 0,692 | 13315 | 0,274 |
| 12254 | -0,003 | 12443 | 0,318 | 13132 | 0,636 | 13321 | 0,681 |
| 12255 | -0,088 | 12444 | 0,184 | 13133 | 0,621 | 13322 | 0,624 |
| 12311 | 0,796 | 12445 | 0,044 | 13134 | 0,408 | 13323 | 0,61 |
| 12312 | 0,74 | 12451 | 0,122 | 13135 | 0,187 | 13324 | 0,397 |
| 12313 | 0,725 | 12452 | 0,066 | 13141 | 0,48 | 13325 | 0,176 |
| 12314 | 0,512 | 12453 | 0,051 | 13142 | 0,423 | 13331 | 0,656 |
| 12315 | 0,291 | 12454 | -0,03 | 13143 | 0,409 | 13332 | 0,6 |
| 12321 | 0,698 | 12455 | -0,114 | 13144 | 0,248 | 13333 | 0,585 |
| 12322 | 0,642 | 12511 | 0,469 | 13145 | 0,082 | 13334 | 0,372 |
| 12323 | 0,627 | 12512 | 0,413 | 13151 | 0,16 | 13335 | 0,151 |
| 12324 | 0,414 | 12513 | 0,398 | 13152 | 0,104 | 13341 | 0,444 |
| 12325 | 0,193 | 12514 | 0,317 | 13153 | 0,089 | 13342 | 0,387 |
| 12331 | 0,673 | 12515 | 0,233 | 13154 | 0,008 | 13343 | 0,373 |
| 12332 | 0,617 | 12521 | 0,371 | 13155 | -0,076 | 13344 | 0,212 |
| 12333 | 0,602 | 12522 | 0,315 | 13211 | 0,786 | 13345 | 0,046 |
| 12334 | 0,389 | 12523 | 0,3 | 13212 | 0,73 | 13351 | 0,124 |
| 12335 | 0,168 | 12524 | 0,219 | 13213 | 0,715 | 13352 | 0,068 |
| 12341 | 0,461 | 12525 | 0,135 | 13214 | 0,502 | 13353 | 0,053 |
| 12342 | 0,405 | 12531 | 0,346 | 13215 | 0,281 | 13354 | -0,028 |
| 12343 | 0,39 | 12532 | 0,29 | 13221 | 0,688 | 13355 | -0,112 |
| 12344 | 0,23 | 12533 | 0,275 | 13222 | 0,631 | 13411 | 0,672 |
| 12345 | 0,063 | 12534 | 0,194 | 13223 | 0,617 | 13412 | 0,615 |
| 12351 | 0,141 | 12535 | 0,11 | 13224 | 0,404 | 13413 | 0,601 |
| 12352 | 0,085 | 12541 | 0,241 | 13225 | 0,183 | 13414 | 0,431 |
| 12353 | 0,07 | 12542 | 0,185 | 13231 | 0,663 | 13415 | 0,255 |
| 12354 | -0,011 | 12543 | 0,17 | 13232 | 0,607 | 13421 | 0,573 |
| 12355 | -0,095 | 12544 | 0,089 | 13233 | 0,592 | 13422 | 0,517 |
| 12411 | 0,689 | 12545 | 0,005 | 13234 | 0,379 | 13423 | 0,502 |
| 12412 | 0,633 | 12551 | 0,083 | 13235 | 0,158 | 13424 | 0,333 |
| 12413 | 0,618 | 12552 | 0,027 | 13241 | 0,451 | 13425 | 0,156 |
| 12414 | 0,448 | 12553 | 0,012 | 13242 | 0,394 | 13431 | 0,549 |
| 12415 | 0,272 | 12554 | -0,069 | 13243 | 0,38 | 13432 | 0,492 |
| 12421 | 0,591 | 12555 | -0,153 | 13244 | 0,219 | 13433 | 0,478 |
| 12422 | 0,534 | 13111 | 0,815 | 13245 | 0,053 | 13434 | 0,308 |
| 12423 | 0,52 | 13112 | 0,759 | 13251 | 0,131 | 13435 | 0,132 |
| 13441 | 0,371 | 14125 | 0,185 | 14314 | 0,435 | 14453 | 0,007 |
| 13442 | 0,315 | 14131 | 0,6 | 14315 | 0,247 | 14454 | -0,074 |

| Health state | Index Value | Health state | Index Value | Health state | Index Value | Health state | Index Value |
|---|---|---|---|---|---|---|---|
| 13443 | 0,3 | 14132 | 0,544 | 14321 | 0,588 | 14455 | -0,158 |
| 13444 | 0,166 | 14133 | 0,529 | 14322 | 0,532 | 14511 | 0,425 |
| 13445 | 0,027 | 14134 | 0,348 | 14323 | 0,517 | 14512 | 0,369 |
| 13451 | 0,105 | 14135 | 0,16 | 14324 | 0,337 | 14513 | 0,354 |
| 13452 | 0,049 | 14141 | 0,414 | 14325 | 0,149 | 14514 | 0,273 |
| 13453 | 0,034 | 14142 | 0,357 | 14331 | 0,564 | 14515 | 0,189 |
| 13454 | -0,047 | 14143 | 0,343 | 14332 | 0,508 | 14521 | 0,327 |
| 13455 | -0,131 | 14144 | 0,202 | 14333 | 0,493 | 14522 | 0,27 |
| 13511 | 0,452 | 14145 | 0,055 | 14334 | 0,312 | 14523 | 0,256 |
| 13512 | 0,396 | 14151 | 0,133 | 14335 | 0,124 | 14524 | 0,175 |
| 13513 | 0,381 | 14152 | 0,077 | 14341 | 0,378 | 14525 | 0,091 |
| 13514 | 0,3 | 14153 | 0,062 | 14342 | 0,321 | 14531 | 0,302 |
| 13515 | 0,216 | 14154 | -0,019 | 14343 | 0,307 | 14532 | 0,246 |
| 13521 | 0,354 | 14155 | -0,103 | 14344 | 0,166 | 14533 | 0,231 |
| 13522 | 0,297 | 14211 | 0,694 | 14345 | 0,019 | 14534 | 0,15 |
| 13523 | 0,283 | 14212 | 0,638 | 14351 | 0,097 | 14535 | 0,066 |
| 13524 | 0,202 | 14213 | 0,623 | 14352 | 0,041 | 14541 | 0,197 |
| 13525 | 0,118 | 14214 | 0,442 | 14353 | 0,026 | 14542 | 0,141 |
| 13531 | 0,329 | 14215 | 0,254 | 14354 | -0,055 | 14543 | 0,126 |
| 13532 | 0,273 | 14221 | 0,596 | 14355 | -0,139 | 14544 | 0,045 |
| 13533 | 0,258 | 14222 | 0,539 | 14411 | 0,601 | 14545 | -0,039 |
| 13534 | 0,177 | 14223 | 0,525 | 14412 | 0,545 | 14551 | 0,039 |
| 13535 | 0,093 | 14224 | 0,344 | 14413 | 0,53 | 14552 | -0,017 |
| 13541 | 0,224 | 14225 | 0,156 | 14414 | 0,382 | 14553 | -0,032 |
| 13542 | 0,168 | 14231 | 0,571 | 14415 | 0,228 | 14554 | -0,113 |
| 13543 | 0,153 | 14232 | 0,515 | 14421 | 0,502 | 14555 | -0,197 |
| 13544 | 0,072 | 14233 | 0,5 | 14422 | 0,446 | 15111 | 0,436 |
| 13545 | -0,012 | 14234 | 0,319 | 14423 | 0,431 | 15112 | 0,38 |
| 13551 | 0,066 | 14235 | 0,131 | 14424 | 0,283 | 15113 | 0,365 |
| 13552 | 0,01 | 14241 | 0,385 | 14425 | 0,13 | 15114 | 0,284 |
| 13553 | -0,005 | 14242 | 0,328 | 14431 | 0,478 | 15115 | 0,2 |
| 13554 | -0,086 | 14243 | 0,314 | 14432 | 0,422 | 15121 | 0,338 |
| 13555 | -0,17 | 14244 | 0,173 | 14433 | 0,407 | 15122 | 0,281 |
| 14111 | 0,723 | 14245 | 0,026 | 14434 | 0,259 | 15123 | 0,267 |
| 14112 | 0,667 | 14251 | 0,104 | 14435 | 0,105 | 15124 | 0,186 |
| 14113 | 0,652 | 14252 | 0,048 | 14441 | 0,318 | 15125 | 0,102 |
| 14114 | 0,471 | 14253 | 0,033 | 14442 | 0,262 | 15131 | 0,313 |
| 14115 | 0,283 | 14254 | -0,048 | 14443 | 0,247 | 15132 | 0,257 |
| 14121 | 0,624 | 14255 | -0,132 | 14444 | 0,126 | 15133 | 0,242 |
| 14122 | 0,568 | 14311 | 0,687 | 14445 | 0 | 15134 | 0,161 |
| 14123 | 0,553 | 14312 | 0,631 | 14451 | 0,078 | 15135 | 0,077 |
| 14124 | 0,373 | 14313 | 0,616 | 14452 | 0,022 | 15141 | 0,208 |
| 15142 | 0,152 | 15331 | 0,277 | 21115 | 0,357 | 21254 | 0,026 |
| 15143 | 0,137 | 15332 | 0,221 | 21121 | 0,767 | 21255 | -0,058 |
| 15144 | 0,056 | 15333 | 0,206 | 21122 | 0,708 | 21311 | 0,826 |

| Health state | Index Value | Health state | Index Value | Health state | Index Value | Health state | Index Value |
|---|---|---|---|---|---|---|---|
| 15145 | -0,028 | 15334 | 0,125 | 21123 | 0,693 | 21312 | 0,77 |
| 15151 | 0,05 | 15335 | 0,041 | 21124 | 0,48 | 21313 | 0,755 |
| 15152 | -0,006 | 15341 | 0,172 | 21125 | 0,259 | 21314 | 0,542 |
| 15153 | -0,021 | 15342 | 0,116 | 21131 | 0,739 | 21315 | 0,321 |
| 15154 | -0,102 | 15343 | 0,101 | 21132 | 0,683 | 21321 | 0,728 |
| 15155 | -0,186 | 15344 | 0,02 | 21133 | 0,668 | 21322 | 0,671 |
| 15211 | 0,407 | 15345 | -0,064 | 21134 | 0,455 | 21323 | 0,657 |
| 15212 | 0,351 | 15351 | 0,014 | 21135 | 0,234 | 21324 | 0,444 |
| 15213 | 0,336 | 15352 | -0,042 | 21141 | 0,527 | 21325 | 0,223 |
| 15214 | 0,255 | 15353 | -0,057 | 21142 | 0,47 | 21331 | 0,703 |
| 15215 | 0,171 | 15354 | -0,138 | 21143 | 0,456 | 21332 | 0,647 |
| 15221 | 0,309 | 15355 | -0,222 | 21144 | 0,296 | 21333 | 0,632 |
| 15222 | 0,252 | 15411 | 0,381 | 21145 | 0,129 | 21334 | 0,419 |
| 15223 | 0,238 | 15412 | 0,325 | 21151 | 0,207 | 21335 | 0,198 |
| 15224 | 0,157 | 15413 | 0,31 | 21152 | 0,151 | 21341 | 0,491 |
| 15225 | 0,073 | 15414 | 0,229 | 21153 | 0,136 | 21342 | 0,434 |
| 15231 | 0,284 | 15415 | 0,145 | 21154 | 0,055 | 21343 | 0,42 |
| 15232 | 0,228 | 15421 | 0,282 | 21155 | -0,029 | 21344 | 0,26 |
| 15233 | 0,213 | 15422 | 0,226 | 21211 | 0,836 | 21345 | 0,093 |
| 15234 | 0,132 | 15423 | 0,211 | 21212 | 0,778 | 21351 | 0,171 |
| 15235 | 0,048 | 15424 | 0,13 | 21213 | 0,762 | 21352 | 0,115 |
| 15241 | 0,179 | 15425 | 0,046 | 21214 | 0,549 | 21353 | 0,1 |
| 15242 | 0,123 | 15431 | 0,258 | 21215 | 0,328 | 21354 | 0,019 |
| 15243 | 0,108 | 15432 | 0,202 | 21221 | 0,735 | 21355 | -0,065 |
| 15244 | 0,027 | 15433 | 0,187 | 21222 | 0,679 | 21411 | 0,719 |
| 15245 | -0,057 | 15434 | 0,106 | 21223 | 0,664 | 21412 | 0,663 |
| 15251 | 0,021 | 15435 | 0,022 | 21224 | 0,451 | 21413 | 0,648 |
| 15252 | -0,035 | 15441 | 0,153 | 21225 | 0,23 | 21414 | 0,478 |
| 15253 | -0,05 | 15442 | 0,097 | 21231 | 0,71 | 21415 | 0,302 |
| 15254 | -0,131 | 15443 | 0,082 | 21232 | 0,654 | 21421 | 0,62 |
| 15255 | -0,215 | 15544 | -0,038 | 21233 | 0,639 | 21422 | 0,564 |
| 15311 | 0,4 | 15545 | -0,122 | 21234 | 0,426 | 21423 | 0,549 |
| 15312 | 0,344 | 15551 | -0,044 | 21235 | 0,205 | 21424 | 0,38 |
| 15313 | 0,329 | 15552 | -0,1 | 21241 | 0,498 | 21425 | 0,204 |
| 15314 | 0,248 | 15553 | -0,115 | 21242 | 0,442 | 21431 | 0,596 |
| 15315 | 0,164 | 15554 | -0,196 | 21243 | 0,427 | 21432 | 0,54 |
| 15321 | 0,302 | 15555 | -0,28 | 21244 | 0,267 | 21433 | 0,525 |
| 15322 | 0,245 | 21111 | 0,877 | 21245 | 0,1 | 21434 | 0,355 |
| 15323 | 0,231 | 21112 | 0,809 | 21251 | 0,178 | 21435 | 0,179 |
| 15324 | 0,15 | 21113 | 0,791 | 21252 | 0,122 | 21441 | 0,419 |
| 15325 | 0,066 | 21114 | 0,578 | 21253 | 0,107 | 21442 | 0,362 |
| 21443 | 0,348 | 22132 | 0,596 | 22321 | 0,641 | 22455 | -0,17 |
| 21444 | 0,213 | 22133 | 0,582 | 22322 | 0,585 | 22511 | 0,413 |
| 21445 | 0,074 | 22134 | 0,369 | 22323 | 0,57 | 22512 | 0,356 |
| 21451 | 0,152 | 22135 | 0,148 | 22324 | 0,357 | 22513 | 0,342 |

| Health state | Index Value | Health state | Index Value | Health state | Index Value | Health state | Index Value |
|---|---|---|---|---|---|---|---|
| 21452 | 0,096 | 22141 | 0,44 | 22325 | 0,136 | 22514 | 0,261 |
| 21453 | 0,081 | 22142 | 0,384 | 22331 | 0,617 | 22515 | 0,177 |
| 21454 | 0 | 22143 | 0,369 | 22332 | 0,56 | 22521 | 0,314 |
| 21455 | -0,084 | 22144 | 0,209 | 22333 | 0,546 | 22522 | 0,258 |
| 21511 | 0,499 | 22145 | 0,043 | 22334 | 0,333 | 22523 | 0,243 |
| 21512 | 0,443 | 22151 | 0,121 | 22335 | 0,112 | 22524 | 0,162 |
| 21513 | 0,428 | 22152 | 0,064 | 22341 | 0,404 | 22525 | 0,078 |
| 21514 | 0,347 | 22153 | 0,05 | 22342 | 0,348 | 22531 | 0,29 |
| 21515 | 0,263 | 22154 | -0,031 | 22343 | 0,333 | 22532 | 0,233 |
| 21521 | 0,401 | 22155 | -0,115 | 22344 | 0,173 | 22533 | 0,219 |
| 21522 | 0,344 | 22211 | 0,747 | 22345 | 0,007 | 22534 | 0,138 |
| 21523 | 0,33 | 22212 | 0,691 | 22351 | 0,085 | 22535 | 0,054 |
| 21524 | 0,249 | 22213 | 0,676 | 22352 | 0,028 | 22541 | 0,185 |
| 21525 | 0,165 | 22214 | 0,463 | 22353 | 0,014 | 22542 | 0,128 |
| 21531 | 0,376 | 22215 | 0,242 | 22354 | -0,067 | 22543 | 0,114 |
| 21532 | 0,32 | 22221 | 0,648 | 22355 | -0,151 | 22544 | 0,033 |
| 21533 | 0,305 | 22222 | 0,592 | 22411 | 0,632 | 22545 | -0,051 |
| 21534 | 0,224 | 22223 | 0,577 | 22412 | 0,576 | 22551 | 0,027 |
| 21535 | 0,14 | 22224 | 0,364 | 22413 | 0,561 | 22552 | -0,03 |
| 21541 | 0,271 | 22225 | 0,143 | 22414 | 0,392 | 22553 | -0,044 |
| 21542 | 0,215 | 22231 | 0,624 | 22415 | 0,216 | 22554 | -0,125 |
| 21543 | 0,2 | 22232 | 0,567 | 22421 | 0,534 | 22555 | -0,209 |
| 21544 | 0,119 | 22233 | 0,553 | 22422 | 0,477 | 23111 | 0,758 |
| 21545 | 0,035 | 22234 | 0,34 | 22423 | 0,463 | 23112 | 0,702 |
| 21551 | 0,113 | 22235 | 0,119 | 22424 | 0,293 | 23113 | 0,687 |
| 21552 | 0,057 | 22241 | 0,411 | 22425 | 0,117 | 23114 | 0,474 |
| 21553 | 0,042 | 22242 | 0,355 | 22431 | 0,509 | 23115 | 0,253 |
| 21554 | -0,039 | 22243 | 0,34 | 22432 | 0,453 | 23121 | 0,66 |
| 21555 | -0,123 | 22244 | 0,18 | 22433 | 0,438 | 23122 | 0,603 |
| 22111 | 0,778 | 22245 | 0,014 | 22434 | 0,269 | 23123 | 0,589 |
| 22112 | 0,72 | 22251 | 0,092 | 22435 | 0,093 | 23124 | 0,376 |
| 22113 | 0,705 | 22252 | 0,035 | 22441 | 0,332 | 23125 | 0,155 |
| 22114 | 0,492 | 22253 | 0,021 | 22442 | 0,276 | 23131 | 0,635 |
| 22115 | 0,271 | 22254 | -0,06 | 22443 | 0,261 | 23132 | 0,579 |
| 22121 | 0,678 | 22255 | -0,144 | 22444 | 0,127 | 23133 | 0,564 |
| 22122 | 0,621 | 22311 | 0,74 | 22445 | -0,013 | 23134 | 0,351 |
| 22123 | 0,606 | 22312 | 0,683 | 22451 | 0,066 | 23135 | 0,13 |
| 22124 | 0,393 | 22313 | 0,669 | 22452 | 0,009 | 23141 | 0,423 |
| 22125 | 0,172 | 22314 | 0,456 | 22453 | -0,005 | 23142 | 0,366 |
| 22131 | 0,653 | 22315 | 0,235 | 22454 | -0,086 | 23143 | 0,352 |
| 23144 | 0,192 | 23333 | 0,528 | 23522 | 0,24 | 24155 | -0,16 |
| 23145 | 0,025 | 23334 | 0,315 | 23523 | 0,226 | 24211 | 0,637 |
| 23151 | 0,103 | 23335 | 0,094 | 23524 | 0,145 | 24212 | 0,581 |
| 23152 | 0,047 | 23341 | 0,387 | 23525 | 0,061 | 24213 | 0,566 |
| 23153 | 0,032 | 23342 | 0,33 | 23531 | 0,272 | 24214 | 0,385 |

| | | | | | | <u> </u> | |
|---|---|---|---|---|---|---|---|
| Health state | Index Value | Health state | Index Value | Health state | Index Value | Health state | Index Value |
| 23154 | -0,049 | 23343 | 0,316 | 23532 | 0,216 | 24215 | 0,198 |
| 23155 | -0,133 | 23344 | 0,156 | 23533 | 0,201 | 24221 | 0,539 |
| 23211 | 0,729 | 23345 | -0,011 | 23534 | 0,12 | 24222 | 0,482 |
| 23212 | 0,673 | 23351 | 0,067 | 23535 | 0,036 | 24223 | 0,468 |
| 23213 | 0,658 | 23352 | 0,011 | 23541 | 0,167 | 24224 | 0,287 |
| 23214 | 0,445 | 23353 | -0,004 | 23542 | 0,111 | 24225 | 0,099 |
| 23215 | 0,224 | 23354 | -0,085 | 23543 | 0,096 | 24231 | 0,514 |
| 23221 | 0,631 | 23355 | -0,169 | 23544 | 0,015 | 24232 | 0,458 |
| 23222 | 0,575 | 23411 | 0,615 | 23545 | -0,069 | 24233 | 0,443 |
| 23223 | 0,56 | 23412 | 0,559 | 23551 | 0,009 | 24234 | 0,262 |
| 23224 | 0,347 | 23413 | 0,544 | 23552 | -0,047 | 24235 | 0,075 |
| 23225 | 0,126 | 23414 | 0,374 | 23553 | -0,062 | 24241 | 0,328 |
| 23231 | 0,606 | 23415 | 0,198 | 23554 | -0,143 | 24242 | 0,272 |
| 23232 | 0,55 | 23421 | 0,516 | 23555 | -0,227 | 24243 | 0,257 |
| 23233 | 0,535 | 23422 | 0,46 | 24111 | 0,666 | 24244 | 0,116 |
| 23234 | 0,322 | 23423 | 0,445 | 24112 | 0,61 | 24245 | -0,03 |
| 23235 | 0,101 | 23424 | 0,276 | 24113 | 0,595 | 24251 | 0,048 |
| 23241 | 0,394 | 23425 | 0,1 | 24114 | 0,414 | 24252 | -0,009 |
| 23242 | 0,338 | 23431 | 0,492 | 24115 | 0,227 | 24253 | -0,023 |
| 23243 | 0,323 | 23432 | 0,436 | 24121 | 0,568 | 24254 | -0,104 |
| 23244 | 0,163 | 23433 | 0,421 | 24122 | 0,511 | 24255 | -0,188 |
| 23245 | -0,004 | 23434 | 0,251 | 24123 | 0,497 | 24311 | 0,63 |
| 23251 | 0,074 | 23435 | 0,075 | 24124 | 0,316 | 24312 | 0,574 |
| 23252 | 0,018 | 23441 | 0,315 | 24125 | 0,128 | 24313 | 0,559 |
| 23253 | 0,003 | 23442 | 0,258 | 24131 | 0,543 | 24314 | 0,378 |
| 23254 | -0,078 | 23443 | 0,244 | 24132 | 0,487 | 24315 | 0,191 |
| 23255 | -0,162 | 23444 | 0,109 | 24133 | 0,472 | 24321 | 0,532 |
| 23311 | 0,722 | 23445 | -0,03 | 24134 | 0,291 | 24322 | 0,475 |
| 23312 | 0,666 | 23451 | 0,048 | 24135 | 0,104 | 24323 | 0,461 |
| 23313 | 0,651 | 23452 | -0,008 | 24141 | 0,357 | 24324 | 0,28 |
| 23314 | 0,438 | 23453 | -0,023 | 24142 | 0,3 | 24325 | 0,092 |
| 23315 | 0,217 | 23454 | -0,104 | 24143 | 0,286 | 24331 | 0,507 |
| 23321 | 0,624 | 23455 | -0,188 | 24144 | 0,145 | 24332 | 0,451 |
| 23322 | 0,567 | 23511 | 0,395 | 24145 | -0,002 | 24333 | 0,436 |
| 23323 | 0,553 | 23512 | 0,339 | 24151 | 0,077 | 24334 | 0,255 |
| 23324 | 0,34 | 23513 | 0,324 | 24152 | 0,02 | 24335 | 0,068 |
| 23325 | 0,119 | 23514 | 0,243 | 24153 | 0,006 | 24341 | 0,321 |
| 23331 | 0,599 | 23515 | 0,159 | 24154 | -0,076 | 24342 | 0,264 |
| 23332 | 0,543 | 23521 | 0,297 | 24155 | -0,16 | 24343 | 0,25 |
| 24344 | 0,109 | 24533 | 0,175 | 25222 | 0,196 | 25411 | 0,324 |
| 24345 | -0,038 | 24534 | 0,094 | 25223 | 0,181 | 25412 | 0,268 |
| 24351 | 0,041 | 24535 | 0,01 | 25224 | 0,1 | 25413 | 0,253 |
| 24352 | -0,016 | 24541 | 0,14 | 25225 | 0,016 | 25414 | 0,172 |
| 24353 | -0,031 | 24542 | 0,084 | 25231 | 0,227 | 25415 | 0,088 |
| 24354 | -0,112 | 24543 | 0,069 | 25232 | 0,171 | 25421 | 0,226 |

| Health state | Index Value | Health state | Index Value | Health state | Index Value | Health state | Index Value |
|---|---|---|---|---|---|---|---|
| 24355 | -0,196 | 24544 | -0,012 | 25233 | 0,156 | 25422 | 0,169 |
| 24411 | 0,544 | 24545 | -0,096 | 25234 | 0,075 | 25423 | 0,155 |
| 24412 | 0,488 | 24551 | -0,018 | 25235 | -0,009 | 25424 | 0,074 |
| 24413 | 0,473 | 24552 | -0,074 | 25241 | 0,122 | 25425 | -0,01 |
| 24414 | 0,325 | 24553 | -0,089 | 25242 | 0,066 | 25431 | 0,201 |
| 24415 | 0,172 | 24554 | -0,17 | 25243 | 0,051 | 25432 | 0,145 |
| 24421 | 0,446 | 24555 | -0,254 | 25244 | -0,03 | 25433 | 0,13 |
| 24422 | 0,389 | 25111 | 0,379 | 25245 | -0,114 | 25434 | 0,049 |
| 24423 | 0,375 | 25112 | 0,323 | 25251 | -0,036 | 25435 | -0,035 |
| 24424 | 0,227 | 25113 | 0,308 | 25252 | -0,092 | 25441 | 0,096 |
| 24425 | 0,073 | 25114 | 0,227 | 25253 | -0,107 | 25442 | 0,04 |
| 24431 | 0,421 | 25115 | 0,143 | 25254 | -0,188 | 25443 | 0,025 |
| 24432 | 0,365 | 25121 | 0,281 | 25255 | -0,272 | 25444 | -0,056 |
| 24433 | 0,35 | 25122 | 0,224 | 25311 | 0,343 | 25445 | -0,14 |
| 24434 | 0,202 | 25123 | 0,21 | 25312 | 0,287 | 25451 | -0,062 |
| 24435 | 0,049 | 25124 | 0,129 | 25313 | 0,272 | 25452 | -0,118 |
| 24441 | 0,262 | 25125 | 0,045 | 25314 | 0,191 | 25453 | -0,133 |
| 24442 | 0,205 | 25131 | 0,256 | 25315 | 0,107 | 25454 | -0,214 |
| 24443 | 0,191 | 25132 | 0,2 | 25321 | 0,245 | 25455 | -0,298 |
| 24444 | 0,069 | 25133 | 0,185 | 25322 | 0,188 | 25511 | 0,285 |
| 24445 | -0,057 | 25134 | 0,104 | 25323 | 0,174 | 25512 | 0,229 |
| 24451 | 0,022 | 25135 | 0,02 | 25324 | 0,093 | 25513 | 0,214 |
| 24452 | -0,035 | 25141 | 0,151 | 25325 | 0,009 | 25514 | 0,133 |
| 24453 | -0,05 | 25142 | 0,095 | 25331 | 0,22 | 25515 | 0,049 |
| 24454 | -0,131 | 25143 | 0,08 | 25332 | 0,164 | 25521 | 0,187 |
| 24455 | -0,215 | 25144 | -0,001 | 25333 | 0,149 | 25522 | 0,13 |
| 24511 | 0,369 | 25145 | -0,085 | 25334 | 0,068 | 25523 | 0,116 |
| 24512 | 0,312 | 25151 | -0,007 | 25335 | -0,016 | 25524 | 0,035 |
| 24513 | 0,298 | 25152 | -0,063 | 25341 | 0,115 | 25525 | -0,049 |
| 24514 | 0,217 | 25153 | -0,078 | 25342 | 0,059 | 25531 | 0,162 |
| 24515 | 0,133 | 25154 | -0,159 | 25343 | 0,044 | 25532 | 0,106 |
| 24521 | 0,27 | 25155 | -0,243 | 25344 | -0,037 | 25533 | 0,091 |
| 24522 | 0,214 | 25211 | 0,35 | 25345 | -0,121 | 25534 | 0,01 |
| 24523 | 0,199 | 25212 | 0,294 | 25351 | -0,043 | 25535 | -0,074 |
| 24524 | 0,118 | 25213 | 0,279 | 25352 | -0,099 | 25541 | 0,057 |
| 24525 | 0,034 | 25214 | 0,198 | 25353 | -0,114 | 25542 | 0,001 |
| 24531 | 0,246 | 25215 | 0,114 | 25354 | -0,195 | 25543 | -0,014 |
| 24532 | 0,189 | 25221 | 0,252 | 25355 | -0,279 | 25544 | -0,095 |
| 25545 | -0,179 | 31234 | 0,414 | 31423 | 0,537 | 32112 | 0,707 |
| 25551 | -0,101 | 31235 | 0,193 | 31424 | 0,368 | 32113 | 0,692 |
| 25552 | -0,157 | 31241 | 0,486 | 31425 | 0,191 | 32114 | 0,479 |
| 25553 | -0,172 | 31242 | 0,429 | 31431 | 0,584 | 32115 | 0,258 |
| 25554 | -0,253 | 31243 | 0,415 | 31432 | 0,527 | 32121 | 0,665 |
| 25555 | -0,337 | 31244 | 0,254 | 31433 | 0,513 | 32122 | 0,609 |
| 31111 | 0,85 | 31245 | 0,088 | 31434 | 0,343 | 32123 | 0,594 |

| Health state | Index Value | Health state | Index Value | Health state | Index Value | Health state | Index Value |
|---|---|---|---|---|---|---|---|
| 31112 | 0,794 | 31251 | 0,166 | 31435 | 0,167 | 32124 | 0,381 |
| 31113 | 0,779 | 31252 | 0,11 | 31441 | 0,406 | 32125 | 0,16 |
| 31114 | 0,566 | 31253 | 0,095 | 31442 | 0,35 | 32131 | 0,64 |
| 31115 | 0,345 | 31254 | 0,014 | 31443 | 0,335 | 32132 | 0,584 |
| 31121 | 0,752 | 31255 | -0,07 | 31444 | 0,201 | 32133 | 0,569 |
| 31122 | 0,695 | 31311 | 0,814 | 31445 | 0,062 | 32134 | 0,356 |
| 31123 | 0,681 | 31312 | 0,758 | 31451 | 0,14 | 32135 | 0,135 |
| 31124 | 0,468 | 31313 | 0,743 | 31452 | 0,084 | 32141 | 0,428 |
| 31125 | 0,247 | 31314 | 0,53 | 31453 | 0,069 | 32142 | 0,372 |
| 31131 | 0,727 | 31315 | 0,309 | 31454 | -0,012 | 32143 | 0,357 |
| 31132 | 0,671 | 31321 | 0,716 | 31455 | -0,096 | 32144 | 0,197 |
| 31133 | 0,656 | 31322 | 0,659 | 31511 | 0,487 | 32145 | 0,03 |
| 31134 | 0,443 | 31323 | 0,645 | 31512 | 0,431 | 32151 | 0,108 |
| 31135 | 0,222 | 31324 | 0,432 | 31513 | 0,416 | 32152 | 0,052 |
| 31141 | 0,515 | 31325 | 0,211 | 31514 | 0,335 | 32153 | 0,037 |
| 31142 | 0,458 | 31331 | 0,691 | 31515 | 0,251 | 32154 | -0,044 |
| 31143 | 0,444 | 31332 | 0,635 | 31521 | 0,389 | 32155 | -0,128 |
| 31144 | 0,283 | 31333 | 0,62 | 31522 | 0,332 | 32211 | 0,735 |
| 31145 | 0,117 | 31334 | 0,407 | 31523 | 0,318 | 32212 | 0,678 |
| 31151 | 0,195 | 31335 | 0,186 | 31524 | 0,237 | 32213 | 0,664 |
| 31152 | 0,139 | 31341 | 0,479 | 31525 | 0,153 | 32214 | 0,451 |
| 31153 | 0,124 | 31342 | 0,422 | 31531 | 0,364 | 32215 | 0,23 |
| 31154 | 0,043 | 31343 | 0,408 | 31532 | 0,308 | 32221 | 0,636 |
| 31155 | -0,041 | 31344 | 0,247 | 31533 | 0,293 | 32222 | 0,58 |
| 31211 | 0,821 | 31345 | 0,081 | 31534 | 0,212 | 32223 | 0,565 |
| 31212 | 0,765 | 31351 | 0,159 | 31535 | 0,128 | 32224 | 0,352 |
| 31213 | 0,75 | 31352 | 0,103 | 31541 | 0,259 | 32225 | 0,131 |
| 31214 | 0,537 | 31353 | 0,088 | 31542 | 0,203 | 32231 | 0,612 |
| 31215 | 0,316 | 31354 | 0,007 | 31543 | 0,188 | 32232 | 0,555 |
| 31221 | 0,723 | 31355 | -0,077 | 31544 | 0,107 | 32233 | 0,541 |
| 31222 | 0,666 | 31411 | 0,707 | 31545 | 0,023 | 32234 | 0,328 |
| 31223 | 0,652 | 31412 | 0,65 | 31551 | 0,101 | 32235 | 0,107 |
| 31224 | 0,439 | 31413 | 0,636 | 31552 | 0,045 | 32241 | 0,399 |
| 31225 | 0,218 | 31414 | 0,466 | 31553 | 0,03 | 32242 | 0,343 |
| 31231 | 0,698 | 31415 | 0,29 | 31554 | -0,051 | 32243 | 0,328 |
| 31232 | 0,642 | 31421 | 0,608 | 31555 | -0,135 | 32244 | 0,168 |
| 31233 | 0,627 | 31422 | 0,552 | 32111 | 0,763 | 32245 | 0,002 |
| 32251 | 0,08 | 32435 | 0,08 | 33124 | 0,364 | 33313 | 0,639 |
| 32252 | 0,023 | 32441 | 0,32 | 33125 | 0,143 | 33314 | 0,426 |
| 32253 | 0,009 | 32442 | 0,263 | 33131 | 0,623 | 33315 | 0,205 |
| 32254 | -0,072 | 32443 | 0,249 | 33132 | 0,567 | 33321 | 0,612 |
| 32255 | -0,157 | 32444 | 0,115 | 33133 | 0,552 | 33322 | 0,555 |
| 32311 | 0,727 | 32445 | -0,025 | 33134 | 0,339 | 33323 | 0,541 |
| 32312 | 0,671 | 32451 | 0,053 | 33135 | 0,118 | 33324 | 0,328 |
| 32313 | 0,656 | 32452 | -0,003 | 33141 | 0,411 | 33325 | 0,107 |

| Health state | Index Value | Health state | Index Value | Health state | Index Value | Health state | Index Value |
|---|---|---|---|---|---|---|---|
| 32314 | 0,443 | 32453 | -0,018 | 33142 | 0,354 | 33331 | 0,587 |
| 32315 | 0,222 | 32454 | -0,099 | 33143 | 0,34 | 33332 | 0,531 |
| 32321 | 0,629 | 32455 | -0,183 | 33144 | 0,179 | 33333 | 0,516 |
| 32322 | 0,573 | 32511 | 0,4 | 33145 | 0,013 | 33334 | 0,303 |
| 32323 | 0,558 | 32512 | 0,344 | 33151 | 0,091 | 33335 | 0,082 |
| 32324 | 0,345 | 32513 | 0,329 | 33152 | 0,035 | 33341 | 0,375 |
| 32325 | 0,124 | 32514 | 0,248 | 33153 | 0,02 | 33342 | 0,318 |
| 32331 | 0,604 | 32515 | 0,164 | 33154 | -0,061 | 33343 | 0,304 |
| 32332 | 0,548 | 32521 | 0,302 | 33155 | -0,145 | 33344 | 0,143 |
| 32333 | 0,533 | 32522 | 0,246 | 33211 | 0,717 | 33345 | -0,023 |
| 32334 | 0,32 | 32523 | 0,231 | 33212 | 0,661 | 33351 | 0,055 |
| 32335 | 0,099 | 32524 | 0,15 | 33213 | 0,646 | 33352 | -0,001 |
| 32341 | 0,392 | 32525 | 0,066 | 33214 | 0,433 | 33353 | -0,016 |
| 32342 | 0,336 | 32531 | 0,277 | 33215 | 0,212 | 33354 | -0,097 |
| 32343 | 0,321 | 32532 | 0,221 | 33221 | 0,619 | 33355 | -0,181 |
| 32344 | 0,161 | 32533 | 0,206 | 33222 | 0,562 | 33411 | 0,603 |
| 32345 | -0,006 | 32534 | 0,125 | 33223 | 0,548 | 33412 | 0,546 |
| 32351 | 0,072 | 32535 | 0,041 | 33224 | 0,335 | 33413 | 0,532 |
| 32352 | 0,016 | 32541 | 0,172 | 33225 | 0,114 | 33414 | 0,362 |
| 32353 | 0,001 | 32542 | 0,116 | 33231 | 0,594 | 33415 | 0,186 |
| 32354 | -0,08 | 32543 | 0,101 | 33232 | 0,538 | 33421 | 0,504 |
| 32355 | -0,164 | 32544 | 0,02 | 33233 | 0,523 | 33422 | 0,448 |
| 32411 | 0,62 | 32545 | -0,064 | 33234 | 0,31 | 33423 | 0,433 |
| 32412 | 0,564 | 32551 | 0,014 | 33235 | 0,089 | 33424 | 0,264 |
| 32413 | 0,549 | 32552 | -0,042 | 33241 | 0,382 | 33425 | 0,087 |
| 32414 | 0,379 | 32553 | -0,057 | 33242 | 0,325 | 33431 | 0,48 |
| 32415 | 0,203 | 32554 | -0,138 | 33243 | 0,311 | 33432 | 0,423 |
| 32421 | 0,522 | 32555 | -0,222 | 33244 | 0,15 | 33433 | 0,409 |
| 32422 | 0,465 | 33111 | 0,746 | 33245 | -0,016 | 33434 | 0,239 |
| 32423 | 0,451 | 33112 | 0,69 | 33251 | 0,062 | 33435 | 0,063 |
| 32424 | 0,281 | 33113 | 0,675 | 33252 | 0,006 | 33441 | 0,302 |
| 32425 | 0,105 | 33114 | 0,462 | 33253 | -0,009 | 33442 | 0,246 |
| 32431 | 0,497 | 33115 | 0,241 | 33254 | -0,09 | 33443 | 0,231 |
| 32432 | 0,441 | 33121 | 0,648 | 33255 | -0,174 | 33444 | 0,097 |
| 32433 | 0,426 | 33122 | 0,591 | 33311 | 0,71 | 33445 | -0,042 |
| 32434 | 0,256 | 33123 | 0,577 | 33312 | 0,654 | 33451 | 0,036 |
| 33452 | -0,02 | 34141 | 0,345 | 34325 | 0,08 | 34514 | 0,204 |
| 33453 | -0,035 | 34142 | 0,288 | 34331 | 0,495 | 34515 | 0,12 |
| 33454 | -0,116 | 34143 | 0,274 | 34332 | 0,439 | 34521 | 0,258 |
| 33455 | -0,2 | 34144 | 0,133 | 34333 | 0,424 | 34522 | 0,201 |
| 33511 | 0,383 | 34145 | -0,014 | 34334 | 0,243 | 34523 | 0,187 |
| 33512 | 0,327 | 34151 | 0,064 | 34335 | 0,055 | 34524 | 0,106 |
| 33513 | 0,312 | 34152 | 0,008 | 34341 | 0,309 | 34525 | 0,022 |
| 33514 | 0,231 | 34153 | -0,007 | 34342 | 0,252 | 34531 | 0,233 |
| 33515 | 0,147 | 34154 | -0,088 | 34343 | 0,238 | 34532 | 0,177 |

| Health state | Index Value | Health state | Index Value | Health state | Index Value | Health state | Index Value |
|---|---|---|---|---|---|---|---|
| 33521 | 0,285 | 34155 | -0,172 | 34344 | 0,097 | 34533 | 0,162 |
| 33522 | 0,228 | 34211 | 0,625 | 34345 | -0,05 | 34534 | 0,081 |
| 33523 | 0,214 | 34212 | 0,569 | 34351 | 0,028 | 34535 | -0,003 |
| 33524 | 0,133 | 34213 | 0,554 | 34352 | -0,028 | 34541 | 0,128 |
| 33525 | 0,049 | 34214 | 0,373 | 34353 | -0,043 | 34542 | 0,072 |
| 33531 | 0,26 | 34215 | 0,185 | 34354 | -0,124 | 34543 | 0,057 |
| 33532 | 0,204 | 34221 | 0,527 | 34355 | -0,208 | 34544 | -0,024 |
| 33533 | 0,189 | 34222 | 0,47 | 34411 | 0,532 | 34545 | -0,108 |
| 33534 | 0,108 | 34223 | 0,456 | 34412 | 0,476 | 34551 | -0,03 |
| 33535 | 0,024 | 34224 | 0,275 | 34413 | 0,461 | 34552 | -0,086 |
| 33541 | 0,155 | 34225 | 0,087 | 34414 | 0,313 | 34553 | -0,101 |
| 33542 | 0,099 | 34231 | 0,502 | 34415 | 0,159 | 34554 | -0,182 |
| 33543 | 0,084 | 34232 | 0,446 | 34421 | 0,433 | 34555 | -0,266 |
| 33544 | 0,003 | 34233 | 0,431 | 34422 | 0,377 | 35111 | 0,367 |
| 33545 | -0,081 | 34234 | 0,25 | 34423 | 0,362 | 35112 | 0,311 |
| 33551 | -0,003 | 34235 | 0,062 | 34424 | 0,214 | 35113 | 0,296 |
| 33552 | -0,059 | 34241 | 0,316 | 34425 | 0,061 | 35114 | 0,215 |
| 33553 | -0,074 | 34242 | 0,259 | 34431 | 0,409 | 35115 | 0,131 |
| 33554 | -0,155 | 34243 | 0,245 | 34432 | 0,353 | 35121 | 0,269 |
| 33555 | -0,239 | 34244 | 0,104 | 34433 | 0,338 | 35122 | 0,212 |
| 34111 | 0,654 | 34245 | -0,043 | 34434 | 0,19 | 35123 | 0,198 |
| 34112 | 0,598 | 34251 | 0,035 | 34435 | 0,036 | 35124 | 0,117 |
| 34113 | 0,583 | 34252 | -0,021 | 34441 | 0,249 | 35125 | 0,033 |
| 34114 | 0,402 | 34253 | -0,036 | 34442 | 0,193 | 35131 | 0,244 |
| 34115 | 0,214 | 34254 | -0,117 | 34443 | 0,178 | 35132 | 0,188 |
| 34121 | 0,555 | 34255 | -0,201 | 34444 | 0,057 | 35133 | 0,173 |
| 34122 | 0,499 | 34311 | 0,618 | 34445 | -0,069 | 35134 | 0,092 |
| 34123 | 0,484 | 34312 | 0,562 | 34451 | 0,009 | 35135 | 0,008 |
| 34124 | 0,304 | 34313 | 0,547 | 34452 | -0,047 | 35141 | 0,139 |
| 34125 | 0,116 | 34314 | 0,366 | 34453 | -0,062 | 35142 | 0,083 |
| 34131 | 0,531 | 34315 | 0,178 | 34454 | -0,143 | 35143 | 0,068 |
| 34132 | 0,475 | 34321 | 0,519 | 34455 | -0,227 | 35144 | -0,013 |
| 34133 | 0,46 | 34322 | 0,463 | 34511 | 0,356 | 35145 | -0,097 |
| 34134 | 0,279 | 34323 | 0,448 | 34512 | 0,3 | 35151 | -0,019 |
| 34135 | 0,091 | 34324 | 0,268 | 34513 | 0,285 | 35152 | -0,075 |
| 35153 | -0,09 | 35342 | 0,047 | 35531 | 0,15 | 41215 | 0,299 |
| 35154 | -0,171 | 35343 | 0,032 | 35532 | 0,094 | 41221 | 0,686 |
| 35155 | -0,255 | 35344 | -0,049 | 35533 | 0,079 | 41222 | 0,629 |
| 35211 | 0,338 | 35345 | -0,133 | 35534 | -0,002 | 41223 | 0,615 |
| 35212 | 0,282 | 35351 | -0,055 | 35535 | -0,086 | 41224 | 0,411 |
| 35213 | 0,267 | 35352 | -0,111 | 35541 | 0,045 | 41225 | 0,2 |
| 35214 | 0,186 | 35353 | -0,126 | 35542 | -0,011 | 41231 | 0,661 |
| 35215 | 0,102 | 35354 | -0,207 | 35543 | -0,026 | 41232 | 0,605 |
| 35221 | 0,24 | 35355 | -0,291 | 35544 | -0,107 | 41233 | 0,59 |
| 35222 | 0,183 | 35411 | 0,312 | 35545 | -0,191 | 41234 | 0,387 |

| | | | | | 5 (41)51144 | 1 1 11101 ) 515 1 10 | |
|---|---|---|---|---|---|---|---|
| Health state | Index Value | Health state | Index Value | Health state | Index Value | Health state | Index Value |
| 35223 | 0,169 | 35412 | 0,256 | 35551 | -0,113 | 41235 | 0,176 |
| 35224 | 0,088 | 35413 | 0,241 | 35552 | -0,169 | 41241 | 0,456 |
| 35225 | 0,004 | 35414 | 0,16 | 35553 | -0,184 | 41242 | 0,4 |
| 35231 | 0,215 | 35415 | 0,076 | 35554 | -0,265 | 41243 | 0,385 |
| 35232 | 0,159 | 35421 | 0,213 | 35555 | -0,349 | 41244 | 0,231 |
| 35233 | 0,144 | 35422 | 0,157 | 41111 | 0,813 | 41245 | 0,07 |
| 35234 | 0,063 | 35423 | 0,142 | 41112 | 0,757 | 41251 | 0,149 |
| 35235 | -0,021 | 35424 | 0,061 | 41113 | 0,742 | 41252 | 0,092 |
| 35241 | 0,11 | 35425 | -0,023 | 41114 | 0,539 | 41253 | 0,078 |
| 35242 | 0,054 | 35431 | 0,189 | 41115 | 0,327 | 41254 | -0,004 |
| 35243 | 0,039 | 35432 | 0,133 | 41121 | 0,714 | 41255 | -0,088 |
| 35244 | -0,042 | 35433 | 0,118 | 41122 | 0,658 | 41311 | 0,777 |
| 35245 | -0,126 | 35434 | 0,037 | 41123 | 0,643 | 41312 | 0,721 |
| 35251 | -0,048 | 35435 | -0,047 | 41124 | 0,44 | 41313 | 0,706 |
| 35252 | -0,104 | 35441 | 0,084 | 41125 | 0,229 | 41314 | 0,503 |
| 35253 | -0,119 | 35442 | 0,028 | 41131 | 0,69 | 41315 | 0,291 |
| 35254 | -0,2 | 35443 | 0,013 | 41132 | 0,634 | 41321 | 0,678 |
| 35255 | -0,284 | 35444 | -0,068 | 41133 | 0,619 | 41322 | 0,622 |
| 35311 | 0,331 | 35445 | -0,152 | 41134 | 0,416 | 41323 | 0,607 |
| 35312 | 0,275 | 35451 | -0,074 | 41135 | 0,204 | 41324 | 0,404 |
| 35313 | 0,26 | 35452 | -0,13 | 41141 | 0,485 | 41325 | 0,193 |
| 35314 | 0,179 | 35453 | -0,145 | 41142 | 0,429 | 41331 | 0,654 |
| 35315 | 0,095 | 35454 | -0,226 | 41143 | 0,414 | 41332 | 0,598 |
| 35321 | 0,233 | 35455 | -0,31 | 41144 | 0,26 | 41333 | 0,583 |
| 35322 | 0,176 | 35511 | 0,273 | 41145 | 0,099 | 41334 | 0,38 |
| 35323 | 0,162 | 35512 | 0,217 | 41151 | 0,177 | 41335 | 0,168 |
| 35324 | 0,081 | 35513 | 0,202 | 41152 | 0,121 | 41341 | 0,449 |
| 35325 | -0,004 | 35514 | 0,121 | 41153 | 0,106 | 41342 | 0,393 |
| 35331 | 0,208 | 35515 | 0,037 | 41154 | 0,025 | 41343 | 0,378 |
| 35332 | 0,152 | 35521 | 0,175 | 41155 | -0,059 | 41344 | 0,224 |
| 35333 | 0,137 | 35522 | 0,118 | 41211 | 0,784 | 41345 | 0,063 |
| 35334 | 0,056 | 35523 | 0,104 | 41212 | 0,728 | 41351 | 0,141 |
| 35335 | -0,028 | 35524 | 0,023 | 41213 | 0,713 | 41352 | 0,085 |
| 35341 | 0,103 | 35525 | -0,062 | 41214 | 0,51 | 41353 | 0,07 |
| 41354 | -0,011 | 41543 | 0,17 | 42232 | 0,518 | 42421 | 0,491 |
| 41355 | -0,095 | 41544 | 0,089 | 42233 | 0,504 | 42422 | 0,434 |
| 41411 | 0,676 | 41545 | 0,005 | 42234 | 0,3 | 42423 | 0,42 |
| 41412 | 0,62 | 41551 | 0,083 | 42235 | 0,089 | 42424 | 0,257 |
| 41413 | 0,605 | 41552 | 0,027 | 42241 | 0,37 | 42425 | 0,087 |
| 41414 | 0,442 | 41553 | 0,012 | 42242 | 0,313 | 42431 | 0,466 |
| 41415 | 0,272 | 41554 | -0,069 | 42243 | 0,299 | 42432 | 0,41 |
| 41421 | 0,577 | 41555 | -0,153 | 42244 | 0,144 | 42433 | 0,395 |
| 41422 | 0,521 | 42111 | 0,726 | 42245 | -0,016 | 42434 | 0,232 |
| 41423 | 0,506 | 42112 | 0,67 | 42251 | 0,062 | 42435 | 0,063 |
| 41424 | 0,343 | 42113 | 0,655 | 42252 | 0,006 | 42441 | 0,294 |

| Health state | Index Value | Health state | Index Value | Health state | Index Value | Health state | Index Value |
|---|---|---|---|---|---|---|---|
| 41425 | 0,174 | 42114 | 0,452 | 42253 | -0,009 | 42442 | 0,238 |
| 41431 | 0,553 | 42115 | 0,241 | 42254 | -0,09 | 42443 | 0,223 |
| 41432 | 0,497 | 42121 | 0,628 | 42255 | -0,174 | 42444 | 0,093 |
| 41433 | 0,482 | 42122 | 0,572 | 42311 | 0,69 | 42445 | -0,042 |
| 41434 | 0,319 | 42123 | 0,557 | 42312 | 0,634 | 42451 | 0,036 |
| 41435 | 0,149 | 42124 | 0,353 | 42313 | 0,619 | 42452 | -0,021 |
| 41441 | 0,381 | 42125 | 0,142 | 42314 | 0,416 | 42453 | -0,035 |
| 41442 | 0,325 | 42131 | 0,603 | 42315 | 0,205 | 42454 | -0,116 |
| 41443 | 0,31 | 42132 | 0,547 | 42321 | 0,592 | 42455 | -0,2 |
| 41444 | 0,18 | 42133 | 0,532 | 42322 | 0,536 | 42511 | 0,383 |
| 41445 | 0,044 | 42134 | 0,329 | 42323 | 0,521 | 42512 | 0,326 |
| 41451 | 0,122 | 42135 | 0,118 | 42324 | 0,317 | 42513 | 0,312 |
| 41452 | 0,066 | 42141 | 0,399 | 42325 | 0,106 | 42514 | 0,231 |
| 41453 | 0,051 | 42142 | 0,342 | 42331 | 0,567 | 42515 | 0,147 |
| 41454 | -0,03 | 42143 | 0,328 | 42332 | 0,511 | 42521 | 0,284 |
| 41455 | -0,114 | 42144 | 0,173 | 42333 | 0,496 | 42522 | 0,228 |
| 41511 | 0,469 | 42145 | 0,013 | 42334 | 0,293 | 42523 | 0,213 |
| 41512 | 0,413 | 42151 | 0,091 | 42335 | 0,082 | 42524 | 0,132 |
| 41513 | 0,398 | 42152 | 0,034 | 42341 | 0,363 | 42525 | 0,048 |
| 41514 | 0,317 | 42153 | 0,02 | 42342 | 0,306 | 42531 | 0,26 |
| 41515 | 0,233 | 42154 | -0,061 | 42343 | 0,292 | 42532 | 0,203 |
| 41521 | 0,371 | 42155 | -0,145 | 42344 | 0,137 | 42533 | 0,189 |
| 41522 | 0,315 | 42211 | 0,698 | 42345 | -0,023 | 42534 | 0,108 |
| 41523 | 0,3 | 42212 | 0,641 | 42351 | 0,055 | 42535 | 0,024 |
| 41524 | 0,219 | 42213 | 0,627 | 42352 | -0,002 | 42541 | 0,155 |
| 41525 | 0,135 | 42214 | 0,423 | 42353 | -0,016 | 42542 | 0,098 |
| 41531 | 0,346 | 42215 | 0,212 | 42354 | -0,097 | 42543 | 0,084 |
| 41532 | 0,29 | 42221 | 0,599 | 42355 | -0,181 | 42544 | 0,003 |
| 41533 | 0,275 | 42222 | 0,543 | 42411 | 0,589 | 42545 | -0,081 |
| 41534 | 0,194 | 42223 | 0,528 | 42412 | 0,533 | 42551 | -0,003 |
| 41535 | 0,11 | 42224 | 0,325 | 42413 | 0,518 | 42552 | -0,06 |
| 41541 | 0,241 | 42225 | 0,113 | 42414 | 0,355 | 42553 | -0,074 |
| 41542 | 0,185 | 42231 | 0,575 | 42415 | 0,186 | 42554 | -0,155 |
| 42555 | -0,239 | 43244 | 0,127 | 43433 | 0,378 | 44122 | 0,467 |
| 43111 | 0,709 | 43245 | -0,034 | 43434 | 0,215 | 44123 | 0,452 |
| 43112 | 0,653 | 43251 | 0,045 | 43435 | 0,045 | 44124 | 0,278 |
| 43113 | 0,638 | 43252 | -0,012 | 43441 | 0,277 | 44125 | 0,098 |
| 43114 | 0,435 | 43253 | -0,027 | 43442 | 0,221 | 44131 | 0,499 |
| 43115 | 0,223 | 43254 | -0,108 | 43443 | 0,206 | 44132 | 0,442 |
| 43121 | 0,61 | 43255 | -0,192 | 43444 | 0,076 | 44133 | 0,428 |
| 43122 | 0,554 | 43311 | 0,673 | 43445 | -0,06 | 44134 | 0,254 |
| 43123 | 0,539 | 43312 | 0,617 | 43451 | 0,018 | 44135 | 0,074 |
| 43124 | 0,336 | 43313 | 0,602 | 43452 | -0,038 | 44141 | 0,318 |
| 43125 | 0,125 | 43314 | 0,399 | 43453 | -0,053 | 44142 | 0,262 |
| 43131 | 0,586 | 43315 | 0,187 | 43454 | -0,134 | 44143 | 0,247 |

| Health state | Index Value | Health state | Index Value | Health state | Index Value | Health state | Index Value |
|---|---|---|---|---|---|---|---|
| 43132 | 0,53 | 43321 | 0,574 | 43455 | -0,218 | 44144 | 0,11 |
| 43133 | 0,515 | 43322 | 0,518 | 43511 | 0,365 | 44145 | -0,032 |
| 43134 | 0,312 | 43323 | 0,503 | 43512 | 0,309 | 44151 | 0,047 |
| 43135 | 0,1 | 43324 | 0,3 | 43513 | 0,294 | 44152 | -0,01 |
| 43141 | 0,381 | 43325 | 0,089 | 43514 | 0,213 | 44153 | -0,024 |
| 43142 | 0,325 | 43331 | 0,55 | 43515 | 0,129 | 44154 | -0,105 |
| 43143 | 0,31 | 43332 | 0,494 | 43521 | 0,267 | 44155 | -0,189 |
| 43144 | 0,156 | 43333 | 0,479 | 43522 | 0,211 | 44211 | 0,593 |
| 43145 | -0,005 | 43334 | 0,276 | 43523 | 0,196 | 44212 | 0,536 |
| 43151 | 0,073 | 43335 | 0,064 | 43524 | 0,115 | 44213 | 0,522 |
| 43152 | 0,017 | 43341 | 0,345 | 43525 | 0,031 | 44214 | 0,348 |
| 43153 | 0,002 | 43342 | 0,289 | 43531 | 0,242 | 44215 | 0,168 |
| 43154 | -0,079 | 43343 | 0,274 | 43532 | 0,186 | 44221 | 0,494 |
| 43155 | -0,163 | 43344 | 0,12 | 43533 | 0,171 | 44222 | 0,438 |
| 43211 | 0,68 | 43345 | -0,041 | 43534 | 0,09 | 44223 | 0,423 |
| 43212 | 0,624 | 43351 | 0,037 | 43535 | 0,006 | 44224 | 0,249 |
| 43213 | 0,609 | 43352 | -0,019 | 43541 | 0,137 | 44225 | 0,069 |
| 43214 | 0,406 | 43353 | -0,034 | 43542 | 0,081 | 44231 | 0,47 |
| 43215 | 0,195 | 43354 | -0,115 | 43543 | 0,066 | 44232 | 0,413 |
| 43221 | 0,582 | 43355 | -0,199 | 43544 | -0,015 | 44233 | 0,399 |
| 43222 | 0,525 | 43411 | 0,572 | 43545 | -0,099 | 44234 | 0,225 |
| 43223 | 0,511 | 43412 | 0,516 | 43551 | -0,021 | 44235 | 0,045 |
| 43224 | 0,307 | 43413 | 0,501 | 43552 | -0,077 | 44241 | 0,289 |
| 43225 | 0,096 | 43414 | 0,338 | 43553 | -0,092 | 44242 | 0,233 |
| 43231 | 0,557 | 43415 | 0,168 | 43554 | -0,173 | 44243 | 0,218 |
| 43232 | 0,501 | 43421 | 0,473 | 43555 | -0,257 | 44244 | 0,082 |
| 43233 | 0,486 | 43422 | 0,417 | 44111 | 0,622 | 44245 | -0,06 |
| 43234 | 0,283 | 43423 | 0,402 | 44112 | 0,565 | 44251 | 0,018 |
| 43235 | 0,072 | 43424 | 0,239 | 44113 | 0,551 | 44252 | -0,039 |
| 43241 | 0,352 | 43425 | 0,07 | 44114 | 0,377 | 44253 | -0,053 |
| 43242 | 0,296 | 43431 | 0,449 | 44115 | 0,197 | 44254 | -0,134 |
| 43243 | 0,281 | 43432 | 0,393 | 44121 | 0,523 | 44255 | -0,218 |
| 44311 | 0,586 | 44445 | -0,087 | 45134 | 0,074 | 45323 | 0,144 |
| 44312 | 0,529 | 44451 | -0,009 | 45135 | -0,01 | 45324 | 0,063 |
| 44313 | 0,515 | 44452 | -0,065 | 45141 | 0,121 | 45325 | -0,021 |
| 44314 | 0,341 | 44453 | -0,08 | 45142 | 0,065 | 45331 | 0,19 |
| 44315 | 0,161 | 44454 | -0,16 | 45143 | 0,05 | 45332 | 0,134 |
| 44321 | 0,487 | 44455 | -0,245 | 45144 | -0,031 | 45333 | 0,119 |
| 44322 | 0,431 | 44511 | 0,339 | 45145 | -0,115 | 45334 | 0,038 |
| 44323 | 0,416 | 44512 | 0,282 | 45151 | -0,037 | 45335 | -0,046 |
| 44324 | 0,242 | 44513 | 0,268 | 45152 | -0,093 | 45341 | 0,085 |
| 44325 | 0,062 | 44514 | 0,187 | 45153 | -0,108 | 45342 | 0,029 |
| 44331 | 0,463 | 44515 | 0,103 | 45154 | -0,189 | 45343 | 0,014 |
| 44332 | 0,406 | 44521 | 0,24 | 45155 | -0,273 | 45344 | -0,067 |
| 44333 | 0,392 | 44522 | 0,184 | 45211 | 0,321 | 45345 | -0,151 |

| | | | | | | - | |
|---|---|---|---|---|---|---|---|
| Health state | Index Value | Health state | Index Value | Health state | Index Value | Health state | Index Value |
| 44334 | 0,218 | 44523 | 0,169 | 45212 | 0,264 | 45351 | -0,073 |
| 44335 | 0,038 | 44524 | 0,088 | 45213 | 0,25 | 45352 | -0,129 |
| 44341 | 0,282 | 44525 | 0,004 | 45214 | 0,169 | 45353 | -0,144 |
| 44342 | 0,226 | 44531 | 0,216 | 45215 | 0,085 | 45354 | -0,225 |
| 44343 | 0,211 | 44532 | 0,159 | 45221 | 0,222 | 45355 | -0,309 |
| 44344 | 0,074 | 44533 | 0,145 | 45222 | 0,166 | 45411 | 0,294 |
| 44345 | -0,068 | 44534 | 0,064 | 45223 | 0,151 | 45412 | 0,238 |
| 44351 | 0,011 | 44535 | -0,02 | 45224 | 0,07 | 45413 | 0,223 |
| 44352 | -0,046 | 44541 | 0,111 | 45225 | -0,014 | 45414 | 0,142 |
| 44353 | -0,06 | 44542 | 0,054 | 45231 | 0,198 | 45415 | 0,058 |
| 44354 | -0,141 | 44543 | 0,04 | 45232 | 0,141 | 45421 | 0,196 |
| 44355 | -0,225 | 44544 | -0,041 | 45233 | 0,127 | 45422 | 0,139 |
| 44411 | 0,504 | 44545 | -0,126 | 45234 | 0,046 | 45423 | 0,125 |
| 44412 | 0,448 | 44551 | -0,047 | 45235 | -0,039 | 45424 | 0,044 |
| 44413 | 0,433 | 44552 | -0,104 | 45241 | 0,092 | 45425 | -0,04 |
| 44414 | 0,29 | 44553 | -0,118 | 45242 | 0,036 | 45431 | 0,171 |
| 44415 | 0,142 | 44554 | -0,199 | 45243 | 0,021 | 45432 | 0,115 |
| 44421 | 0,406 | 44555 | -0,283 | 45244 | -0,06 | 45433 | 0,1 |
| 44422 | 0,35 | 45111 | 0,349 | 45245 | -0,144 | 45434 | 0,019 |
| 44423 | 0,335 | 45112 | 0,293 | 45251 | -0,066 | 45435 | -0,065 |
| 44424 | 0,192 | 45113 | 0,278 | 45252 | -0,122 | 45441 | 0,066 |
| 44425 | 0,043 | 45114 | 0,197 | 45253 | -0,137 | 45442 | 0,01 |
| 44431 | 0,381 | 45115 | 0,113 | 45254 | -0,218 | 45443 | -0,005 |
| 44432 | 0,325 | 45121 | 0,251 | 45255 | -0,302 | 45444 | -0,086 |
| 44433 | 0,31 | 45122 | 0,195 | 45311 | 0,313 | 45445 | -0,17 |
| 44434 | 0,167 | 45123 | 0,18 | 45312 | 0,257 | 45451 | -0,092 |
| 44435 | 0,019 | 45124 | 0,099 | 45313 | 0,242 | 45452 | -0,148 |
| 44441 | 0,226 | 45125 | 0,015 | 45314 | 0,161 | 45453 | -0,163 |
| 44442 | 0,169 | 45131 | 0,226 | 45315 | 0,077 | 45454 | -0,244 |
| 44443 | 0,155 | 45132 | 0,17 | 45321 | 0,215 | 45455 | -0,328 |
| 44444 | 0,036 | 45133 | 0,155 | 45322 | 0,159 | 45511 | 0,255 |
| 45512 | 0,199 | 51151 | -0,05 | 51335 | -0,059 | 51524 | -0,009 |
| 45513 | 0,184 | 51152 | -0,106 | 51341 | 0,072 | 51525 | -0,093 |
| 45514 | 0,103 | 51153 | -0,121 | 51342 | 0,016 | 51531 | 0,119 |
| 45515 | 0,019 | 51154 | -0,202 | 51343 | 0,001 | 51532 | 0,063 |
| 45521 | 0,157 | 51155 | -0,286 | 51344 | -0,08 | 51533 | 0,048 |
| 45522 | 0,101 | 51211 | 0,307 | 51345 | -0,164 | 51534 | -0,033 |
| 45523 | 0,086 | 51212 | 0,251 | 51351 | -0,086 | 51535 | -0,117 |
| 45524 | 0,005 | 51213 | 0,236 | 51352 | -0,142 | 51541 | 0,014 |
| 45525 | -0,079 | 51214 | 0,155 | 51353 | -0,157 | 51542 | -0,042 |
| 45531 | 0,132 | 51215 | 0,071 | 51354 | -0,238 | 51543 | -0,057 |
| 45532 | 0,076 | 51221 | 0,209 | 51355 | -0,322 | 51544 | -0,138 |
| 45533 | 0,061 | 51222 | 0,152 | 51411 | 0,281 | 51545 | -0,222 |
| 45534 | -0,02 | 51223 | 0,138 | 51412 | 0,225 | 51551 | -0,144 |
| 45535 | -0,104 | 51224 | 0,057 | 51413 | 0,21 | 51552 | -0,2 |

| Health state | Index Value | Health state | Index Value | Health state | Index Value | Health state | Index Value |
|---|---|---|---|---|---|---|---|
| 45541 | 0,027 | 51225 | -0,027 | 51414 | 0,129 | 51553 | -0,215 |
| 45542 | -0,029 | 51231 | 0,184 | 51415 | 0,045 | 51554 | -0,296 |
| 45543 | -0,044 | 51232 | 0,128 | 51421 | 0,182 | 51555 | -0,38 |
| 45544 | -0,125 | 51233 | 0,113 | 51422 | 0,126 | 52111 | 0,249 |
| 45545 | -0,209 | 51234 | 0,032 | 51423 | 0,111 | 52112 | 0,193 |
| 45551 | -0,131 | 51235 | -0,052 | 51424 | 0,03 | 52113 | 0,178 |
| 45552 | -0,187 | 51241 | 0,079 | 51425 | -0,054 | 52114 | 0,097 |
| 45553 | -0,202 | 51242 | 0,023 | 51431 | 0,158 | 52115 | 0,013 |
| 45554 | -0,283 | 51243 | 0,008 | 51432 | 0,102 | 52121 | 0,151 |
| 45555 | -0,367 | 51244 | -0,073 | 51433 | 0,087 | 52122 | 0,095 |
| 51111 | 0,336 | 51245 | -0,157 | 51434 | 0,006 | 52123 | 0,08 |
| 51112 | 0,28 | 51251 | -0,079 | 51435 | -0,078 | 52124 | -0,001 |
| 51113 | 0,265 | 51252 | -0,135 | 51441 | 0,053 | 52125 | -0,085 |
| 51114 | 0,184 | 51253 | -0,15 | 51442 | -0,003 | 52131 | 0,126 |
| 51115 | 0,1 | 51254 | -0,231 | 51443 | -0,018 | 52132 | 0,07 |
| 51121 | 0,238 | 51255 | -0,315 | 51444 | -0,099 | 52133 | 0,055 |
| 51122 | 0,181 | 51311 | 0,3 | 51445 | -0,183 | 52134 | -0,026 |
| 51123 | 0,167 | 51312 | 0,244 | 51451 | -0,105 | 52135 | -0,11 |
| 51124 | 0,086 | 51313 | 0,229 | 51452 | -0,161 | 52141 | 0,021 |
| 51125 | 0,002 | 51314 | 0,148 | 51453 | -0,176 | 52142 | -0,035 |
| 51131 | 0,213 | 51315 | 0,064 | 51454 | -0,257 | 52143 | -0,05 |
| 51132 | 0,157 | 51321 | 0,202 | 51455 | -0,341 | 52144 | -0,131 |
| 51133 | 0,142 | 51322 | 0,145 | 51511 | 0,242 | 52145 | -0,215 |
| 51134 | 0,061 | 51323 | 0,131 | 51512 | 0,186 | 52151 | -0,137 |
| 51135 | -0,023 | 51324 | 0,05 | 51513 | 0,171 | 52152 | -0,193 |
| 51141 | 0,108 | 51325 | -0,035 | 51514 | 0,09 | 52153 | -0,208 |
| 51142 | 0,052 | 51331 | 0,177 | 51515 | 0,006 | 52154 | -0,289 |
| 51143 | 0,037 | 51332 | 0,121 | 51521 | 0,144 | 52155 | -0,373 |
| 51144 | -0,044 | 51333 | 0,106 | 51522 | 0,087 | 52211 | 0,221 |
| 51145 | -0,128 | 51334 | 0,025 | 51523 | 0,073 | 52212 | 0,164 |
| 52213 | 0,15 | 52352 | -0,229 | 52541 | -0,073 | 53225 | -0,131 |
| 52214 | 0,069 | 52353 | -0,244 | 52542 | -0,129 | 53231 | 0,08 |
| 52215 | -0,016 | 52354 | -0,325 | 52543 | -0,144 | 53232 | 0,024 |
| 52221 | 0,122 | 52355 | -0,409 | 52544 | -0,225 | 53233 | 0,009 |
| 52222 | 0,066 | 52411 | 0,194 | 52545 | -0,309 | 53234 | -0,072 |
| 52223 | 0,051 | 52412 | 0,138 | 52551 | -0,231 | 53235 | -0,156 |
| 52224 | -0,03 | 52413 | 0,123 | 52552 | -0,287 | 53241 | -0,025 |
| 52225 | -0,114 | 52414 | 0,042 | 52553 | -0,302 | 53242 | -0,081 |
| 52231 | 0,098 | 52415 | -0,042 | 52554 | -0,383 | 53243 | -0,096 |
| 52232 | 0,041 | 52421 | 0,096 | 52555 | -0,467 | 53244 | -0,177 |
| 52233 | 0,027 | 52422 | 0,04 | 53111 | 0,232 | 53245 | -0,261 |
| 52234 | -0,054 | 52423 | 0,025 | 53112 | 0,176 | 53251 | -0,183 |
| 52235 | -0,139 | 52424 | -0,056 | 53113 | 0,161 | 53252 | -0,239 |
| 52241 | -0,008 | 52425 | -0,14 | 53114 | 0,08 | 53253 | -0,254 |
| 52242 | -0,064 | 52431 | 0,071 | 53115 | -0,004 | 53254 | -0,335 |

| Health state | Index Value | Health state | Index Value | Health state | Index Value | Health state | Index Value |
|---|---|---|---|---|---|---|---|
| 52243 | -0,079 | 52432 | 0,015 | 53121 | 0,134 | 53255 | -0,419 |
| 52244 | -0,16 | 52433 | 0 | 53122 | 0,077 | 53311 | 0,196 |
| 52245 | -0,244 | 52434 | -0,081 | 53123 | 0,063 | 53312 | 0,14 |
| 52251 | -0,166 | 52435 | -0,165 | 53124 | -0,019 | 53313 | 0,125 |
| 52252 | -0,222 | 52441 | -0,034 | 53125 | -0,103 | 53314 | 0,044 |
| 52253 | -0,237 | 52442 | -0,09 | 53131 | 0,109 | 53315 | -0,04 |
| 52254 | -0,317 | 52443 | -0,105 | 53132 | 0,053 | 53321 | 0,098 |
| 52255 | -0,402 | 52444 | -0,186 | 53133 | 0,038 | 53322 | 0,041 |
| 52311 | 0,213 | 52445 | -0,27 | 53134 | -0,043 | 53323 | 0,027 |
| 52312 | 0,157 | 52451 | -0,192 | 53135 | -0,127 | 53324 | -0,055 |
| 52313 | 0,142 | 52452 | -0,248 | 53141 | 0,004 | 53325 | -0,139 |
| 52314 | 0,061 | 52453 | -0,263 | 53142 | -0,052 | 53331 | 0,073 |
| 52315 | -0,023 | 52454 | -0,344 | 53143 | -0,067 | 53332 | 0,017 |
| 52321 | 0,115 | 52455 | -0,428 | 53144 | -0,148 | 53333 | 0,002 |
| 52322 | 0,059 | 52511 | 0,155 | 53145 | -0,232 | 53334 | -0,079 |
| 52323 | 0,044 | 52512 | 0,099 | 53151 | -0,154 | 53335 | -0,163 |
| 52324 | -0,037 | 52513 | 0,084 | 53152 | -0,21 | 53341 | -0,032 |
| 52325 | -0,121 | 52514 | 0,003 | 53153 | -0,225 | 53342 | -0,088 |
| 52331 | 0,09 | 52515 | -0,081 | 53154 | -0,306 | 53343 | -0,103 |
| 52332 | 0,034 | 52521 | 0,057 | 53155 | -0,39 | 53344 | -0,184 |
| 52333 | 0,019 | 52522 | 0,001 | 53211 | 0,203 | 53345 | -0,268 |
| 52334 | -0,062 | 52523 | -0,014 | 53212 | 0,147 | 53351 | -0,19 |
| 52335 | -0,146 | 52524 | -0,095 | 53213 | 0,132 | 53352 | -0,246 |
| 52341 | -0,015 | 52525 | -0,179 | 53214 | 0,051 | 53353 | -0,261 |
| 52342 | -0,071 | 52531 | 0,032 | 53215 | -0,033 | 53354 | -0,342 |
| 52343 | -0,086 | 52532 | -0,024 | 53221 | 0,105 | 53355 | -0,426 |
| 52344 | -0,167 | 52533 | -0,039 | 53222 | 0,048 | 53411 | 0,177 |
| 52345 | -0,251 | 52534 | -0,12 | 53223 | 0,034 | 53412 | 0,121 |
| 52351 | -0,173 | 52535 | -0,204 | 53224 | -0,047 | 53413 | 0,106 |
| 53414 | 0,025 | 53553 | -0,319 | 54242 | -0,108 | 54431 | 0,027 |
| 53415 | -0,059 | 53554 | -0,4 | 54243 | -0,123 | 54432 | -0,029 |
| 53421 | 0,078 | 53555 | -0,484 | 54244 | -0,204 | 54433 | -0,044 |
| 53422 | 0,022 | 54111 | 0,205 | 54245 | -0,288 | 54434 | -0,125 |
| 53423 | 0,007 | 54112 | 0,149 | 54251 | -0,21 | 54435 | -0,209 |
| 53424 | -0,074 | 54113 | 0,134 | 54252 | -0,266 | 54441 | -0,078 |
| 53425 | -0,158 | 54114 | 0,053 | 54253 | -0,281 | 54442 | -0,134 |
| 53431 | 0,054 | 54115 | -0,031 | 54254 | -0,362 | 54443 | -0,149 |
| 53432 | -0,002 | 54121 | 0,107 | 54255 | -0,446 | 54444 | -0,23 |
| 53433 | -0,017 | 54122 | 0,05 | 54311 | 0,169 | 54445 | -0,314 |
| 53434 | -0,098 | 54123 | 0,036 | 54312 | 0,113 | 54451 | -0,236 |
| 53435 | -0,182 | 54124 | -0,045 | 54313 | 0,098 | 54452 | -0,292 |
| 53441 | -0,051 | 54125 | -0,129 | 54314 | 0,017 | 54453 | -0,307 |
| 53442 | -0,107 | 54131 | 0,082 | 54315 | -0,067 | 54454 | -0,388 |
| 53443 | -0,122 | 54132 | 0,026 | 54321 | 0,071 | 54455 | -0,472 |
| 53444 | -0,203 | 54133 | 0,011 | 54322 | 0,014 | 54511 | 0,111 |

| | Statistical Analysis I fan 55/100/0K | | | | | | |
|---|---|---|---|---|---|---|---|
| Health state | Index Value | Health state | Index Value | Health state | Index Value | Health state | Index Value |
| 53445 | -0,287 | 54134 | -0,07 | 54323 | 0 | 54512 | 0,055 |
| 53451 | -0,209 | 54135 | -0,154 | 54324 | -0,081 | 54513 | 0,04 |
| 53452 | -0,265 | 54141 | -0,023 | 54325 | -0,165 | 54514 | -0,041 |
| 53453 | -0,28 | 54142 | -0,079 | 54331 | 0,046 | 54515 | -0,125 |
| 53454 | -0,361 | 54143 | -0,094 | 54332 | -0,01 | 54521 | 0,013 |
| 53455 | -0,445 | 54144 | -0,175 | 54333 | -0,025 | 54522 | -0,044 |
| 53511 | 0,138 | 54145 | -0,259 | 54334 | -0,106 | 54523 | -0,058 |
| 53512 | 0,082 | 54151 | -0,181 | 54335 | -0,19 | 54524 | -0,139 |
| 53513 | 0,067 | 54152 | -0,237 | 54341 | -0,059 | 54525 | -0,223 |
| 53514 | -0,014 | 54153 | -0,252 | 54342 | -0,115 | 54531 | -0,012 |
| 53515 | -0,098 | 54154 | -0,333 | 54343 | -0,13 | 54532 | -0,068 |
| 53521 | 0,04 | 54155 | -0,417 | 54344 | -0,211 | 54533 | -0,083 |
| 53522 | -0,017 | 54211 | 0,176 | 54345 | -0,295 | 54534 | -0,164 |
| 53523 | -0,032 | 54212 | 0,12 | 54351 | -0,217 | 54535 | -0,248 |
| 53524 | -0,113 | 54213 | 0,105 | 54352 | -0,273 | 54541 | -0,117 |
| 53525 | -0,197 | 54214 | 0,024 | 54353 | -0,288 | 54542 | -0,173 |
| 53531 | 0,015 | 54215 | -0,06 | 54354 | -0,369 | 54543 | -0,188 |
| 53532 | -0,041 | 54221 | 0,078 | 54355 | -0,453 | 54544 | -0,269 |
| 53533 | -0,056 | 54222 | 0,022 | 54411 | 0,15 | 54545 | -0,353 |
| 53534 | -0,137 | 54223 | 0,007 | 54412 | 0,094 | 54551 | -0,275 |
| 53535 | -0,221 | 54224 | -0,074 | 54413 | 0,079 | 54552 | -0,331 |
| 53541 | -0,09 | 54225 | -0,158 | 54414 | -0,002 | 54553 | -0,346 |
| 53542 | -0,146 | 54231 | 0,053 | 54415 | -0,086 | 54554 | -0,427 |
| 53543 | -0,161 | 54232 | -0,003 | 54421 | 0,052 | 54555 | -0,511 |
| 53544 | -0,242 | 54233 | -0,018 | 54422 | -0,005 | 55111 | 0,122 |
| 53545 | -0,326 | 54234 | -0,099 | 54423 | -0,019 | 55112 | 0,066 |
| 53551 | -0,248 | 54235 | -0,183 | 54424 | -0,1 | 55113 | 0,051 |
| 53552 | -0,304 | 54241 | -0,052 | 54425 | -0,184 | 55114 | -0,03 |
| 55115 | -0,114 | 55254 | -0,445 | 55443 | -0,232 | | |
| 55121 | 0,024 | 55255 | -0,529 | 55444 | -0,313 | | |
| 55122 | -0,033 | 55311 | 0,086 | 55445 | -0,397 | | |
| 55123 | -0,048 | 55312 | 0,03 | 55451 | -0,319 | | |
| 55124 | -0,129 | 55313 | 0,015 | 55452 | -0,375 | | |
| 55125 | -0,213 | 55314 | -0,066 | 55453 | -0,39 | | |
| 55131 | -0,001 | 55315 | -0,15 | 55454 | -0,471 | | |
| 55132 | -0,057 | 55321 | -0,013 | 55455 | -0,555 | | |
| 55133 | -0,072 | 55322 | -0,069 | 55511 | 0,028 | | |
| 55134 | -0,153 | 55323 | -0,084 | 55512 | -0,028 | | |
| 55135 | -0,237 | 55324 | -0,165 | 55513 | -0,043 | | |
| 55141 | -0,106 | 55325 | -0,249 | 55514 | -0,124 | | |
| 55142 | -0,162 | 55331 | -0,037 | 55515 | -0,208 | | |
| 55143 | -0,177 | 55332 | -0,093 | 55521 | -0,071 | | |
| 55144 | -0,258 | 55333 | -0,108 | 55522 | -0,127 | | |
| 55145 | -0,342 | 55334 | -0,189 | 55523 | -0,142 | | |
| 55151 | -0,264 | 55335 | -0,273 | 55524 | -0,223 | | |

| Health state | Index Value | Health state | Index Value | Health state | Index Value | Health state | Index Value |
|---|---|---|---|---|---|---|---|
| 55152 | -0,32 | 55341 | -0,142 | 55525 | -0,307 | 1100010 | 1111021 7 11110 |
| 55153 | -0,335 | 55342 | -0,198 | 55531 | -0,095 | | |
| 55154 | -0,416 | 55343 | -0,213 | 55532 | -0,151 | | |
| 55155 | -0,5 | 55344 | -0,294 | 55533 | -0,166 | | |
| 55211 | 0,093 | 55345 | -0,378 | 55534 | -0,247 | | |
| 55212 | 0,037 | 55351 | -0,3 | 55535 | -0,331 | | |
| 55213 | 0,022 | 55352 | -0,356 | 55541 | -0,2 | | |
| 55214 | -0,059 | 55353 | -0,371 | 55542 | -0,256 | | |
| 55215 | -0,143 | 55354 | -0,452 | 55543 | -0,271 | | |
| 55221 | -0,005 | 55355 | -0,536 | 55544 | -0,352 | | |
| 55222 | -0,062 | 55411 | 0,067 | 55545 | -0,436 | | |
| 55223 | -0,076 | 55412 | 0,011 | 55551 | -0,358 | | |
| 55224 | -0,157 | 55413 | -0,004 | 55552 | -0,414 | | |
| 55225 | -0,241 | 55414 | -0,085 | 55553 | -0,429 | | |
| 55231 | -0,03 | 55415 | -0,169 | 55554 | -0,51 | | |
| 55232 | -0,086 | 55421 | -0,032 | 55555 | -0,594 | | |
| 55233 | -0,101 | 55422 | -0,088 | | | | |
| 55234 | -0,182 | 55423 | -0,103 | | | | |
| 55235 | -0,266 | 55424 | -0,184 | | | | |
| 55241 | -0,135 | 55425 | -0,268 | | | | |
| 55242 | -0,191 | 55431 | -0,056 | | | | |
| 55243 | -0,206 | 55432 | -0,112 | | | | |
| 55244 | -0,287 | 55433 | -0,127 | | | | |
| 55245 | -0,371 | 55434 | -0,208 | | | | |
| 55251 | -0,293 | 55435 | -0,292 | | | | |
| 55252 | -0,349 | 55441 | -0,161 | | | | |
| 55253 | -0,364 | 55442 | -0,217 | | | | |